## GlaxoSmithKline group of companies

## TITLE PAGE

**Protocol Title:** A Phase III, Randomized, Multicenter, Parallel-Group, Double-Blind, Double-Dummy Study in Adolescent and Adult Female Participants Comparing the Efficacy and Safety of Gepotidacin to Nitrofurantoin in the Treatment of Uncomplicated Urinary Tract Infection (Acute Cystitis)

Protocol Number: 212390 / Amendment 3

Compound GSK2140944

**Number:** 

Study Phase: Phase III

**Short Title:** Phase III, Double-Blind, Parallel-Group, Comparator-Controlled, Efficacy and Safety Study of Gepotidacin in the Treatment of Uncomplicated Urinary Tract Infection (Acute Cystitis); Efficacy of Antibacterial Gepotidacin Evaluated (EAGLE-3)

# **Sponsor Name and Legal Registered Address:**

GlaxoSmithKline Research & Development Limited 980 Great West Road Brentford Middlesex, TW8 9GS UK

# **Sponsor Name and Legal Registered Address:**

GlaxoSmithKline 1250 South Collegeville Road PO Box 5089 Collegeville, PA 19426-0989 USA

# Medical monitor name and contact information can be found in the Study Reference Manual

### **Regulatory Agency Identifying Number:**

IND: 111885

EudraCT: 2020-000553-27

**Protocol Amendment Number: 3** 

**Approval Date:** 03-NOV-2021

Copyright 2021 the GlaxoSmithKline group of companies. All rights reserved. Unauthorized copying or use of this information is prohibited.

# **SPONSOR SIGNATORY:**

**Protocol Title:** A Phase III, Randomized, Multicenter, Parallel-Group, Double-Blind, Double-Dummy Study in Adolescent and Adult Female Participants Comparing the Efficacy and Safety of Gepotidacin to Nitrofurantoin in the Treatment of Uncomplicated Urinary Tract Infection (Acute Cystitis)

| Protocol Number: 212390 / Amendment 3 | | |
|---|---|---|
| Compound<br>Number: | GSK2140944 | |
| | Sc, MBBS (Hons), FRCP, FACE al Sciences (Infectious Diseases) | Date |

The signed page is a separate document.

**Medical Monitor Name and Contact Information** can be found in the Study Reference Manual.

# PROTOCOL AMENDMENT SUMMARY OF CHANGES TABLE

| DOCUMENT HISTORY | | |
|--------------------------|-------------|----------------|
| Document Date DNG Number | | |
| Amendment 3 | 03-NOV-2021 | TMF-13817737 |
| Amendment 2 | 14-APR-2021 | TMF-12037491 |
| Amendment 1 | 14-NOV-2019 | 2019N407320_01 |
| Original Protocol | 31-JUL-2019 | 2019N407320_00 |

### Amendment 3 03-NOV-2021

This global amendment is considered to be substantial.

Overall Rationale for the Amendment: This global amendment added details for an interim analysis to be conducted and managed by an Independent Data Monitoring Committee and sample size impact on the primary analysis population. The primary analysis method was updated from Cochran-Mantel-Haenszel to Miettinen and Nurminen. Other revisions include increasing the inclusion window for the onset of acute cystitis clinical signs and symptoms from  $\leq$ 72 hours to  $\leq$ 96 hours, minor revisions to 2 exclusion criteria were made, prescreening activities for consent and urine pregnancy testing were clarified, the potential for home healthcare visits was added, minor revisions were made to allow more site and participant flexibility at the Baseline Visit, and minor updates were made to the Schedule of Events table for the interactive response technology. The amendment also includes additional minor administrative and wording edits.

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| Synopsis | Added interim analysis and | To allow interim statistical |
| 4.2 Scientific<br>Rationale for Study<br>Design | Independent Data Monitoring Committee details, including updates to the number of evaluable participants needed and | evaluation for efficacy and futility |
| 6.3. Measures to Minimize Bias: Randomization and Blinding | sample size determination<br>revisions, as well as applicable<br>revisions to section numbers and<br>content (i.e. additions and | |
| 9.1 Statistical<br>Hypothesis | deletions) in the statistical section | |
| 9.2 Sample Size Determination | | |
| 9.4.1 General<br>Considerations | | |
| 9.4.2 Efficacy<br>Analysis | | |
| 9.5 Interim Analysis | | |
| 9.6 Data Monitoring<br>Committee or Other<br>Review Board | | |
| 10.3.5 Committee<br>Structure | | |
| Throughout | | |
| Synopsis | Revised the secondary | Consistency between primary and |
| 3 Objectives and Estimands/Endpoints | therapeutic response objective | secondary endpoint |
| Synopsis | Revised description of the number | Updated for clarification related to |
| 9.1 Statistical<br>Hypotheses | of participants in the primary analysis population based on interim analysis considerations | the interim analysis on the primary analysis population |
| 9.2 Sample Size<br>Determination | and clarified that the number of randomized participants may vary | |
| 9.5 Interim Analysis | based on evaluability rate and review of qualifying uropathogens | |
| 1.3 Schedule of<br>Activities | Divided the "Interactive response technology" row in to 2 separate rows specific for the screening and randomization modules | To align with how the interactive response is being used at study sites and to more closely follow the expected order of procedures |

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| 1.3 Schedule of | Clarified prescreening activities | Consistency with the Study |
| Activities | that may occur | Reference Manual |
| 8 Study Assessments and Procedures | | |
| 1.3 Schedule of Activities | Added text to allow potential home healthcare visits. Such visits will | To support study feasibility |
| 4.1 Overall Design | be limited to where applicable regulations and infrastructure | |
| 10.5.2 Study Procedures During the COVID-19 Pandemic | allow | |
| 2.3.1 Risk<br>Assessment | Minor text clarifications for clinical QTc effects and added relevant exposures for nonclinical embryofetal effects | Consistency with currently known safety data |
| 5.1 Inclusion Criteria<br>#2 | Revised the criterion to allow the onset of clinical signs and symptoms of acute cystitis within ≤96 hours prior to study entry | To support study enrollment |
| 5.2 Exclusion Criteria<br>#2 | Edited to include "uncontrolled" before high blood pressure | Text clarification |
| 5.2 Exclusion Criteria<br>#30 | Revised wording to support a "no" response, which is in line with this being an exclusion criterion | Text clarification |
| 8 Study Assessments and Procedures | Removed the requirement for participants to remain at the site for approximately 1 to 2 hours after dosing at the Baseline Visit; however, retained text indicating that posttreatment assessments still need to be completed | To support site flexibility for study conduct |
| 8 Study Assessments and Procedures | Removed topical antifungal restriction from the TOC Visit | After TOC assessments are complete, participants may be treated with either topical or systemic antifungals |

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| 8.1.2.1 Microbiological Outcome and Response 8.1.3.1. Clinical Signs and Symptom Scores, Clinical Outcomes, and Clinical | Removed footnote from tables with regard to comparing the date and time of other systemic antimicrobials received with the date and time of On-therapy Visit | Updated as "time" will not be used |
| Response | | |
| 9.1 Statistical<br>Hypothesis | Clarified null and alternative hypotheses for superiority testing | Clarification of the planned analysis |
| 9.4.2 Efficacy<br>Analysis | Revised the primary analysis to be performed using the Miettinen and Nurminen method instead of the Cochran-Mantel-Haenszel method | Consistency with the reporting and analysis plan |
| 10.3.1 Regulatory and Ethical Considerations | Clarified that, in countries where certain responsibilities reside with the sponsor instead of the investigator, GSK or its designee will be responsible for those activities | Clarification for study sites |
| Throughout | Minor editorial and document formatting revisions | Minor, therefore, have not been summarized |

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| ТІТ | TLE PAG | GE | 1 |
| SP | ONSOF | R SIGNATORY: | 2 |
| PR | отос | OL AMENDMENT SUMMARY OF CHANGES TABLE | 3 |
| 1. | PROT | OCOL SUMMARY | 10 |
| | 1.1. | Synopsis | |
| | 1.2. | Schema | |
| | 1.3. | Schedule of Activities (SoA) | |
| 2. | INTRO | ODUCTION | 19 |
| | 2.1. | Study Rationale | 19 |
| | 2.2. | Background | 20 |
| | 2.3. | Benefit/Risk Assessment | |
| | | 2.3.1. Risk Assessment | |
| | | 2.3.2. Benefit Assessment | |
| | | 2.3.3. Overall Benefit: Risk Conclusion | 29 |
| 3. | OBJE | CTIVES AND ESTIMANDS/ENDPOINTS | 30 |
| 4. | STUD | Y DESIGN | 36 |
| Τ. | 4.1. | Overall Design | |
| | 4.2. | Scientific Rationale for Study Design | |
| | 4.3. | Justification for Dose | 38 |
| | 4.4. | End-of-Study Definition | |
| 5. | STUD | Y POPULATION | 41 |
| | 5.1. | Inclusion Criteria | 41 |
| | 5.2. | Exclusion Criteria | |
| | 5.3. | Lifestyle Considerations | |
| | <b>-</b> 4 | 5.3.1. Meals and Dietary Restrictions | |
| | 5.4. | Screen Failures | 45 |
| 6. | | Y TREATMENT | |
| | 6.1. | Study Treatments Administered | |
| | 6.2. | Preparation/Handling/Storage/Accountability | |
| | 6.3.<br>6.4. | Measures to Minimize Bias: Randomization and Blinding | |
| | 6.5. | Study Treatment Compliance Concomitant Therapy | |
| | 0.5. | 6.5.1. Permitted Medications and Nondrug Therapies | |
| | | 6.5.2. Prohibited Medications and Nondrug Therapies | |
| | 6.6. | Dose Modification | |
| | 6.7. | Treatment after the End of the Study | |
| 7. | DISC | ONTINUATION OF STUDY TREATMENT AND PARTICIPANT | |
| | DISC | ONTINUATION/WITHDRAWAL | |
| | 7.1. | Discontinuation of Study Treatment | 52 |
| | | 7.1.1. Liver Chemistry Stopping Criteria | 52 |

| | | 7.1.2. QTc Stopping Criteria | 54 |
|---|---|---|---|
| | | 7.1.3. Rechallenge | 55 |
| | | 7.1.4. Gastrointestinal Evaluation Criteria | |
| | 7.2. | Participant Discontinuation/Withdrawal from the Study | |
| | 7.3. | Lost to Follow-Up | |
| 8. | STUD | Y ASSESSMENTS AND PROCEDURES | |
| | 8.1. | Efficacy Assessments | 59 |
| | | 8.1.1. Therapeutic Response Evaluation | 59 |
| | | 8.1.2. Bacteriology Samples | 59 |
| | | 8.1.3. Clinical Evaluation | 65 |
| | 8.2. | Safety Assessments | 69 |
| | | 8.2.1. Physical Examinations | |
| | | 8.2.2. Vital Signs | |
| | | 8.2.3. Electrocardiograms | |
| | | 8.2.4. Clinical Safety Laboratory Assessments | |
| | 8.3. | Adverse Events and Serious Adverse Events | |
| | 0.0. | 8.3.1. Time Period and Frequency for Collecting AE and SAE | |
| | | Information | 71 |
| | | 8.3.2. Method of Detecting AEs and SAEs | 72 |
| | | 8.3.3. Follow-up of AEs and SAEs | |
| | | 8.3.4. Regulatory Reporting Requirements for SAEs | |
| | | 8.3.5. Pregnancy | |
| | | 8.3.6. Cardiovascular and Death Events | 73 |
| | | 8.3.7. Adverse Events of Special Interest | |
| | 8.4. | Treatment of Overdose | |
| | 8.5. | Pharmacokinetics | |
| | 8.6. | Pharmacodynamics | |
| | 8.7. | Genetics | |
| | 8.8. | Biomarkers | |
| | 8.9. | Immunogenicity Assessments. | |
| | CCI | Illimunoqenicity Assessments. | 74 |
| 9. | | ISTICAL CONSIDERATIONS | |
| | 9.1. | | |
| | 9.2. | Sample Size Determination | |
| | | 9.2.1. Justification of Sample Size | |
| | | 9.2.2. Sample Size Sensitivity | |
| | 9.3. | Populations for Analyses | |
| | 9.4. | Statistical Analyses | |
| | | 9.4.1. General Considerations | 79 |
| | | 9.4.2. Efficacy Analyses | 80 |
| | | 9.4.3. Safety Analyses | 83 |
| | 9.5. | Interim Analysis | 84 |
| | 9.6. | Data Monitoring Committee or Other Review Board | |
| 40 | 01155 | ACRITING ROCKINGS TATION AND CREEKTION | |
| 10. | | ORTING DOCUMENTATION AND OPERATIONAL | |
| | | SIDERATIONS | 86 |
| | 10.1. | Appendix 1: Clostridium Difficile Testing Procedure and Algorithm | 86 |
| | 10.2. | 11 1 | |
| | | Information | |
| | | 10.2.1 Definitions: | 87 |

11.

| | 10.2.2. Contraception Guidance: | 88 |
|---|---|---|
| | 10.2.3. Collection of Pregnancy Information: | 89 |
| 10.3. | Appendix 3: Regulatory, Ethical, and Study Oversight | |
| | Considerations | |
| | 10.3.1. Regulatory and Ethical Considerations | |
| | 10.3.2. Financial Disclosure | |
| | 10.3.3. Informed Consent/Assent Process | |
| | 10.3.4. Data Protection | |
| | 10.3.5. Committees Structure | |
| | 10.3.6. Dissemination of Clinical Study Data | |
| | 10.3.7. Data Quality Assurance | 93 |
| | 10.3.8. Source Documents | |
| | 10.3.9. Study and Site Start and Closure | 94 |
| | 10.3.10. Publication Policy | 94 |
| 10.4. | Appendix 4: Algorithm for Determining Qualifying Uropathogens | 95 |
| 10.5. | Appendix 5: COVID-19 Protocol Information | 96 |
| | 10.5.1. Overall Rationale for this Appendix | 96 |
| | 10.5.2. Study Procedures During the COVID-19 Pandemic | 96 |
| 10.6. | Appendix 6: Clinical Signs and Symptoms Score for Acute Cystitis | 98 |
| CCI | | |
| 10.8. | Appendix 8: Clinical Laboratory Tests | 101 |
| 10.9. | Appendix 9: Additional Guidance on Permitted and Prohibited | |
| | Medications and Crediblemeds.org | 104 |
| 10.10. | Appendix 10: Liver Safety: Required Actions and Follow-up | |
| | Assessments | 107 |
| 10.11. | Appendix 11: Adverse Events: Definitions and Procedures for | |
| | Recording, Evaluating, Follow-up, and Reporting | 111 |
| | 10.11.1. Definition of Adverse Event | 111 |
| | 10.11.2. Definition of SAE | |
| | 10.11.3. Cardiovascular Adverse Events of Special Interest and | |
| | Cases of Clostridium Difficile | 113 |
| | 10.11.4. Recording and Follow-Up of AE and SAE | |
| | 10.11.5. Reporting of SAE to GSK/PPD | |
| 10 12 | Appendix 12: Genetics | |
| 10.12. | Appendix 13: Division of Microbiology and Infectious Diseases Adult | |
| 10.10. | Toxicity Tables for Adverse Event Assessment | 110 |
| 10 14 | Appendix 14: Abbreviations and Trademarks | |
| | Appendix 15: Protocol Amendment History | |
| 10.13. | Appendix 10. Flotocol Amendment History | 121 |
| REFE | RENCES | 134 |

# 1. PROTOCOL SUMMARY

# 1.1. Synopsis

**Protocol Title:** A Phase III, Randomized, Multicenter, Parallel-Group, Double-Blind, Double-Dummy Study in Adolescent and Adult Female Participants Comparing the Efficacy and Safety of Gepotidacin to Nitrofurantoin in the Treatment of Uncomplicated Urinary Tract Infection (Acute Cystitis)

**Short Title:** Phase III, Double-Blind, Parallel-Group, Comparator-Controlled, Efficacy and Safety Study of Gepotidacin in the Treatment of Uncomplicated Urinary Tract Infection (Acute Cystitis); Efficacy of Antibacterial Gepotidacin Evaluated (EAGLE-3)

### Rationale:

Urinary tract infections (UTIs; acute cystitis) are very common, with approximately 11% of women (greater than 18 years of age) reporting at least 1 episode of acute cystitis per year. In addition, one third of all female adolescents and women experience more than 1 episode of acute cystitis, requiring antimicrobial therapy, by the age of 24 years. The predominant uropathogen isolated in community-acquired UTIs is *Escherichia coli* (75% to 90%) followed by *Staphylococcus saprophyticus* (5% to 15%). Multidrug resistance, which is typically associated with nosocomial infections, has now emerged at the community level and has made treatment approaches for UTIs more difficult. Gepotidacin is a first-in-class, novel triazaacenaphthylene bacterial type II topoisomerase inhibitor. The microbiological spectrum of activity of gepotidacin includes *E. coli*, *S. saprophyticus*, and *Enterococcus faecalis*. This Phase III study aims to evaluate the therapeutic response (combined microbiological and clinical efficacy per participant) of oral gepotidacin compared to oral nitrofurantoin for acute cystitis in adolescent and adult female participants.

## **Objectives and Estimands/Endpoints:**

| Objectives | Endpoints |
|---|---|
| Primary | |
| To assess the combined clinical and microbiological efficacy of gepotidacin compared to nitrofurantoin, at the Test-of-Cure (TOC) Visit, in female participants with acute cystitis with qualifying bacterial uropathogen(s) at Baseline that all are susceptible to nitrofurantoin | Therapeutic response (combined per-participant microbiological and clinical response) at the TOC Visit |

TMF-13817737 212390

| Objectives | Endpoints |
|---|---|
| Secondary | |
| To assess the clinical efficacy of<br>gepotidacin compared to<br>nitrofurantoin, at the TOC and<br>Follow-up Visits, in female<br>participants with acute cystitis | Clinical outcome and response at the TOC and Follow-up Visits |
| To assess the clinical efficacy of gepotidacin compared to nitrofurantoin, at the TOC and Follow-up Visits, in female participants with acute cystitis with qualifying bacterial uropathogen(s) at Baseline that all are susceptible to nitrofurantoin | Clinical outcome and response at the TOC and Follow-up Visits |
| To assess the microbiological efficacy of gepotidacin compared to nitrofurantoin, at the TOC and Follow-up Visits, in female participants with acute cystitis with qualifying bacterial uropathogen(s) at Baseline that all are susceptible to nitrofurantoin | Microbiological outcome and response at the TOC and Follow-up Visits |
| To assess the combined clinical and microbiological efficacy of gepotidacin compared to nitrofurantoin, at the Follow-up Visit, in female participants with acute cystitis with qualifying bacterial uropathogen(s) at Baseline that all are susceptible to nitrofurantoin | Therapeutic response (combined per-participant microbiological and clinical response) at the Follow-up Visit |
| To assess the safety and tolerability of gepotidacin compared to nitrofurantoin in female participants with acute cystitis | Treatment-emergent adverse events and serious adverse events and change from baseline results for clinical laboratory tests, electrocardiograms, and vital sign measurements |

Note: Exploratory objectives are described in the main protocol text.

# **Primary Estimand**

The primary clinical question of interest is: What is the treatment effect on the therapeutic response after 5 days of treatment with gepotidacin 1500 mg twice daily compared to 5 days of treatment with nitrofurantoin 100 mg twice daily in participants with acute cystitis with qualifying bacterial uropathogen(s) at Baseline that all are susceptible to nitrofurantoin, regardless of treatment discontinuation for any reason. Receipt of systemic antimicrobials will impact the endpoint definition (see Section 8.1.2.1 and Section 8.1.3.1).

The primary estimand is described by the following attributes:

- Population: Female participants with acute cystitis with qualifying bacterial uropathogen(s) at Baseline that all are susceptible to nitrofurantoin.
- Treatment condition: Gepotidacin 1500 mg twice daily for 5 days versus nitrofurantoin 100 mg twice daily for 5 days, regardless of adherence.
- Variable: Therapeutic response (combined per-participant microbiological and clinical response) at the TOC Visit. Microbiological success is defined as eradication (i.e., reduction) of all qualifying bacterial uropathogens recovered at baseline to <10<sup>3</sup> colony-forming units/mL (CFU/mL) as observed on quantitative urine culture without the participant receiving other systemic antimicrobials. Clinical success is defined as resolution of signs and symptoms of acute cystitis present at Baseline (and no new signs and symptoms) without the participant receiving other systemic antimicrobials.
- Summary measure: Absolute difference in the therapeutic success rate in the gepotidacin and nitrofurantoin treatment groups.
- Intercurrent events (ICEs):
  - Study treatment discontinuation (due to any reason) treatment policy strategy (interest is in the treatment effect regardless of study treatment discontinuation).
  - Use of systemic antimicrobials composite strategy. This ICE is captured through the definitions of microbiological and clinical response (see Section 8.1.2.1 and Section 8.1.3.1) and will be counted as therapeutic failures.

### Rationale for Estimand:

Interest lies in the treatment effect regardless of whether the full course of 5 days of treatment was taken or not, which reflects how patients may be treated in clinical practice. Hence, a treatment policy strategy is appropriate for treatment withdrawal before completing 5 days of treatment. Use of other systemic antimicrobials may confound the bacterial culture results; thus, the microbiological response will be considered failure. For clinical data, the use of a systemic antimicrobial for acute cystitis is a sign of treatment failure and use of a systemic antimicrobial for another infection cannot be considered a success as it confounds the assessment of efficacy. Therefore, the definition of a successful therapeutic response precludes the use of other systemic antimicrobials.

# Secondary Estimands:

The secondary clinical questions of interest are: What is the treatment effect on each of the secondary efficacy endpoints after 5 days of treatment with gepotidacin 1500 mg twice daily compared to 5 days of treatment with nitrofurantoin 100 mg twice daily in participants with acute cystitis (clinical endpoints) and in participants with acute cystitis with qualifying bacterial uropathogen(s) at Baseline that all are susceptible to nitrofurantoin (therapeutic, clinical, and microbiological endpoints), regardless of treatment discontinuation for any reason. Receipt of systemic antimicrobials impacts the endpoint definition (see Section 8.1.2.1 and Section 8.1.3.1).

For each of the secondary endpoints the estimand will follow a similar approach to the estimand for the primary endpoint and will use the same strategies for the ICEs. The exception is the summary measure for the outcome endpoints. These endpoints are descriptively summarized; therefore, the summary measure will be the percentage in each clinical and microbiological outcome category in the gepotidacin and nitrofurantoin arms separately (as no direct comparison between treatment groups will be made) (see Section 8.1.2.1 and Section 8.1.3.1 for endpoint definitions).

The safety endpoint will use a treatment policy strategy of the ICE of withdrawal from treatment as the safety will be assessed at all postbaseline assessments irrespective of whether the participant completed the treatment.

See Table 1 for the components of estimand for the secondary endpoints.

# Overall Design:

- Study 212390 is a Phase III, randomized, multicenter, parallel-group, double-blind, double-dummy, comparator-controlled, noninferiority study in adolescent and adult female participants comparing the efficacy and safety of oral gepotidacin to oral nitrofurantoin in the treatment of uncomplicated UTI (acute cystitis).
- Participants will be stratified by age category and acute cystitis recurrence and will be randomly assigned in a 1:1 ratio to receive either oral gepotidacin or oral nitrofurantoin.
- Appropriate safety, efficacy, and microbiological assessments will be conducted at the Baseline (Day 1) Visit and repeated at the On-therapy (Day 2 to 4), TOC (Day 10 to 13), and Follow-up (Day 28±3) Visits.
- For the primary efficacy endpoint of therapeutic response (combined per-participant microbiological and clinical response), therapeutic success refers to participants who have been deemed both a microbiological success (reduction of all qualifying bacterial uropathogens [e.g., ≥10<sup>5</sup> colony-forming units/mL (CFU/mL)] recovered at Baseline to <10<sup>3</sup> CFU/mL as observed on quantitative urine culture without the participant receiving other systemic antimicrobials) and

a clinical success (resolution of signs and symptoms of acute cystitis present at Baseline [and no new signs and symptoms] without the participant receiving other systemic antimicrobials) at the TOC Visit in the Microbiological Intent-to-Treat Nitrofurantoin-Susceptible (micro-ITT NTF-S) Population, regardless of treatment discontinuation.

**Disclosure Statement**: This is a parallel-group treatment study with 2 arms that is participant, care provider, investigator, and outcomes assessor blinded.

# **Number of Participants:**

The study is planned to enroll approximately 2500 participants to fulfill the maximum target sample size of approximately 884 participants in the primary analysis micro-ITT NTF-S Population. The final number of randomized participants may vary based on the evaluability rate and review of qualifying uropathogens by an unblinded Statistical Data Analysis Center.

# **Treatment Groups and Duration:**

- Participants will receive 1 of the following treatments:
  - Gepotidacin: 1500 mg administered orally twice daily for 5 days (Note: Each dose should be taken after food consumption and with water to assist with tolerability.)
  - Nitrofurantoin: 100 mg administered orally twice daily for 5 days (Note: Each dose should be taken after food consumption and with water.)
- The duration of study participation is approximately 28 days with 4 planned study visits:
  - Baseline (Day 1) Visit
  - On-therapy (Day 2 to 4) Visit
  - TOC (Day 10 to 13) Visit
  - Follow-up (Day 28±3) Visit

**Data Monitoring or Other Committee:** Yes; this study will include an Independent Data Monitoring Committee for interim analysis purposes, a GlaxoSmithKline Safety Review Team will monitor blinded safety data, and a Microbiology Review Team will monitor blinded microbiological data instream.

# 1.2. Schema

Figure 1 Study Design Schematic



BID=twice daily; HPF=high-power field; TOC=Test-of-Cure; WBC=white blood cell.

- a. There will be central randomization with stratification by age category (<18 years, ≥18 to 50 years, or >50 years) and acute cystitis recurrence (nonrecurrent infection or recurrent infection, defined as a confirmed infection [not including the current infection in the calculation] with at least 1 prior episode within the past 3 months, at least 2 prior episodes within the past 6 months, or at least 3 prior episodes within the past 12 months before study entry).
- b. Study treatment will be administered under double-blind, double-dummy conditions. Each dose should be taken after food consumption and with water.

# 1.3. Schedule of Activities (SoA)

| Visit <sup>a</sup> | Bas | eline | On-Therapy <sup>b</sup> | TOC | Follow-up | Early<br>Withdrawal |
|---|---|---|---|---|---|---|
| Study Day | | 1 | | | | |
| Procedure | Predose | Postdose | 2 to 4 | 10 to 13 | 28±3 | NA |
| Written informed consent/assent | Х | | | | | |
| IRT – Screening module | Х | | | | | |
| Inclusion and exclusion criteria | Х | | | | | |
| Participant demography | Х | | | | | |
| Physical examination (including height and weight at Baseline only) | Х | | | Χc | | |
| Record acute cystitis signs and symptoms <sup>a</sup> | Х | | X | Х | Х | Х |
| CCI | | | | | | |
| Medical/surgical history | X | | | | | |
| Diagnosis of presumptive acute cystitisf | Х | | | | | |
| Bacteriology samples9 | Х | | χ'n | X | X | Х |
| Randomization | Х | | | | | |
| 12-lead ECGi | Х | | χi | | | |
| Vital sign measurementsi | X | | X | X | | |
| Hematology, chemistry, and urinalysis | Х | | X | X | | |
| Serology (hepatitis B and C and HIV) <sup>k</sup> | X | | | | | |
| Urine pregnancy test | Χı | | χı | X | | Х |
| Drug and alcohol screen | X | | | | | |
| OCI " | | | | | | |
| IRT – Randomization module | X | | | | | |
| Administer oral dose of study treatment <sup>n</sup> | | X | Χί,o | | | |
| Serious adverse events <sup>p</sup> | Χ | X | X | X | X | Х |
| Adverse events <sup>q</sup> | | X | X | X | X | X |
| Concomitant medication review | Х | X | X | X | X | Х |
| Study treatment compliancer | | | X | X | | |
| Schedule next visit | χ5 | | Χt | Xt | Xt | |
| Genetic sample <sup>u</sup> | X | | | | | |

ECG =electrocardiogram; HIV=human immunodeficiency virus; HPF=high-power field; IRT=interactive response technology; NA=not applicable; TOC=Test-of-Cure; UTI=urinary tract infection; WBC=white blood cell.

Note: To reduce participant on-site visits or if unforeseen issues impact clinic visits, and participants are unable to attend a site visit, home healthcare (home visits and telemedicine visits) may be used to conduct procedures as detailed in the Study Reference Manual. Home healthcare will only be utilized where applicable country and local regulations and infrastructure allow.

212390

- a. For all study visits, to minimize the amount of time that participants spend at the clinic, eConsent may be utilized and remote collection of study-related data may be obtained as described in the Study Reference Manual. Thus, some visit data may be collected through a combination of telemedicine and on-site visits. Collection of information via telemedicine will be performed only where local regulations permit. Prescreening activities may also be conducted, including a prescreening informed consent and urine testing, as detailed in Section 8 and the Study Reference Manual.
- b. For the On-therapy (Day 2 to 4) Visit: Participants will be instructed to return to the study site within 1 to 3 days postrandomization. Each treatment day will be assessed over 24 hours starting with the first dose of study treatment, as further detailed in the Study Reference Manual. For the TOC (Day 10 to 13) Visit: Participants will be instructed to return to the study site 5 to 8 days after completion of study treatment.
- At the TOC Visit, the physical examination may be symptom directed and is only required if indicated for a specific participant.
- d. Individual clinical signs and symptoms scores of acute cystitis will be recorded by a study physician or otherwise appropriately medically trained staff based on participant interview and using the scoring system in Appendix 6. The same scorer will be used at all assessment time points for each participant, on all occasions, whenever possible.

study physician or otherwise appropriately medically trained staff who performed the clinical scoring assessment.

- f. Based on confirmation of nitrite or pyuria (>15 WBC/HPF or the presence of 3+/large leukocyte esterase) from a pretreatment clean-catch midstream urine sample per local laboratory procedures.
- g. Participants will provide a clean-catch midstream urine sample at each visit for Gram stain, quantitative bacteriology culture, and in vitro antimicrobial susceptibility testing by a designated central laboratory(ies). Refer to the laboratory manual.
- A bacteriology urine sample will be collected at the On-therapy Visit, as further detailed in the Study Reference Manual.
- i. See Section 5.2 for ECG exclusion criterion for participants aged ≥12 to <18 years. For additional details see Section 7.1.2 and Section 8.2.3. Triplicate ECGs will be performed at Baseline. For the first approximately 1200 participants enrolled, On-therapy triplicate ECGs will also be obtained. The On-therapy ECGs will be collected at approximately 2 hours postdose (i.e., expected time of maximum concentration; ECG collection should ideally be within approximately 1.5 hours postdose to 4 hours postdose). After the first approximately 1200 participants have triplicate ECGs performed at On-therapy, the ECG collection at this visit is no longer a protocol requirement. Electrocardiograms will be reviewed locally by the investigator for safety purposes. Electrocardiograms will be centrally overread for the data analysis.</p>
- Take measurement of temperature, blood pressure, and pulse rate.
- k. If serology testing was performed within 3 months prior to the first dose of study treatment and the results were **positive**, testing at Baseline is **not required**. If testing was performed within 3 months and any result was **negative**, testing at Baseline is **required**.
- For women of childbearing potential, a negative high sensitivity urine pregnancy test is sufficient for eligibility. See Appendix 8 for Baseline urine test sensitivity requirements
  and Appendix 2 for associated contraception requirements. Pregnancy testing should be performed after Dose 4 and before Dose 8, as specified in Appendix 8.

n. Participants will receive oral study treatment twice daily for 5 days under double-blind, double-dummy conditions. The first oral dose will be administered at the study site during the Baseline Visit; participants will self-administer as outpatients thereafter, beginning with the second dose. Each dose should be taken after food consumption and with water. The date and time of each dose administered at the study site will be recorded in the source documents.

- o. At the On-therapy Visit, whenever it is possible, the participant will have the pregnancy test performed at the study site. If the visit coincides with the 8th dose, the participant will take their next dose of study treatment at the study site after negative pregnancy test results are confirmed. Note: The On-therapy Visit should be scheduled to support completion of the postdose ECG within the protocol-defined window. Also, in a woman of childbearing potential, the high sensitivity pregnancy test must be performed and show negative results at the latest before Dose 8 of study treatment is taken.
- p. Record serious adverse events from the time of consent/assent in order to fulfill international regulatory requirements.
- g. Record adverse events from the time of the first dose of study treatment.
- r. Determine study treatment compliance by performing pill count.
- s. Confirm return day/time for the On-therapy, TOC, and Follow-up Visits.
- t. Previsit reminder: Study site staff will contact the participant 24±4 hours before the scheduled On-therapy, TOC, and Follow-up Visits.
- u. Collect sample only if the participant has a signed consent/assent specific for this purpose. The Baseline Visit is the recommended time to collect the sample, but it can be collected at any time during the study.

# 2. INTRODUCTION

Gepotidacin (GSK2140944), a novel triazaacenaphthylene bacterial type II topoisomerase inhibitor, is being developed for the treatment of uncomplicated urinary tract infections (UTIs; acute cystitis). Gepotidacin has activity versus key pathogens, including drug-resistant strains associated with a range of conventional and biothreat infections. The microbiological spectrum of activity of gepotidacin includes *Escherichia coli*, the key causative pathogen of acute cystitis, *Staphylococcus saprophyticus*, and *Enterococcus faecalis*.

Gepotidacin selectively inhibits bacterial DNA replication by interacting in a unique way on the GyrA subunit of bacterial DNA gyrase and the ParC subunit of bacterial topoisomerase IV. This interaction appears to be highly specific to bacterial topoisomerases as evidenced by weak in vitro inhibition of human topoisomerase  $II\alpha$ , supporting the selective activity of gepotidacin against the bacterial target. The novel mode of action of this new class antibacterial affords in vitro activity against most target pathogens resistant to established antibacterials, including fluoroquinolones.

# 2.1. Study Rationale

This study is being conducted based on the need to identify new and effective oral antibiotic treatment options for acute cystitis, as such therapies are becoming limited due to the increase of multidrug-resistant (MDR) pathogens and extended-spectrum β-lactamase (ESBL)-producing Enterobacterales pathogens, which are impacting the efficacy of currently available oral antibacterial treatment options (see Section 2.2). Two Phase II studies have been conducted and the results demonstrated that gepotidacin was efficacious in the treatment of uncomplicated urogenital gonorrhea and acute bacterial skin and skin structure infections (ABSSSIs) (see Section 5.3.3 in the investigator's brochure [IB] for details). In addition, a Phase IIa pharmacokinetic (PK) study (206899) was conducted in 22 female participants with acute cystitis that also included exploratory clinical and microbiological efficacy objectives. All 22 participants were evaluable for PK and clinical efficacy analysis. Of the 22 participants, 19 participants (86%) and 18 participants (82%) achieved symptom resolution at the Test-of-Cure (TOC) and Follow-up Visits, respectively. Eight of 22 participants (36%) who received at least 1 dose of gepotidacin had a qualifying baseline uropathogen (5 with E. coli isolates, 1 with a S. saprophyticus isolate, 1 with a Klebsiella pneumoniae isolate, and 1 with a Citrobacter koseri isolate). Of these 8 participants, 7 participants (88%) and 6 participants (75%) had a microbiological response of microbiological success (<10<sup>3</sup> colony-forming units/mL [CFU/mL]) at the TOC and Follow-up Visits, respectively. Furthermore, of these 8 participants, 6 participants (75%) and 5 participants (63%) had a therapeutic response (combined per-participant microbiological and clinical response) of success at the TOC and Follow-up Visits, respectively. Refer to the IB for PK, safety, and additional efficacy results.

This study (212390) aims to evaluate the therapeutic response (combined microbiological and clinical efficacy per participant) of oral gepotidacin compared to oral nitrofurantoin for acute cystitis in adolescent and adult female participants.

#### 2.2. **Background**

Urinary tract infections are very common, with approximately 11% of women >18 years of age experiencing at least 1 episode of acute cystitis per year [Foxman, 2000]. Of these, half will experience more than 1 recurrent episode over their lifetime [Foxman, 2000]. The peak incidence of acute cystitis occurs in young, sexually active women ages 18 to 29 years [Fihn, 2003]. The predominant uropathogens isolated in community-acquired UTIs are E. coli (75% to 90%) followed by S. saprophyticus (5% to 15%) [Stamm, 1993; Talan, 2000; Foxman, 2010]. Klebsiella, Enterobacter, Proteus species, and enterococci are observed in only 5% to 10% of acute cystitis [Stamm, 1993; Talan, 2000; Foxman, 2010].

212390

Multidrug resistance, which is typically associated with nosocomial infections, has now emerged at the community level and has made treatment approaches for UTIs more difficult [Hooton, 2012; Flamm, 2014; Sanchez, 2016]. This has led to increasing patient morbidity, increasing costs due to reassessment and retreatment, higher rates of hospitalization, and increased use of broad-spectrum antibiotics [Foxman, 2002; Gupta, 2011a; Hooton, 2012]. Furthermore, ESBL-producing Enterobacteriaceae (now recognized as Enterobacterales), which includes E. coli, is recognized as a serious threat by the Centers for Disease Control and Prevention (CDC) [CDC, 2019] and drug-resistant Enterobacteriaceae is a critical priority pathogen for the World Health Organization (WHO) [WHO, 2017]. One reason for this serious threat level is the growing rise in the MDR E. coli sequence type (ST)-131 clone [Johnson, 2012; Nicolas-Chanoine, 2014]. Spread of this ST-131 clone has led to UTIs and blood stream infections caused by MDR E. coli worldwide [Peirano, 2010]. The availability of oral antimicrobials that are effective against ESBLs is limited and, for some outpatient infections, no oral options remain.

An in vitro evaluation of antimicrobial resistance of urinary E. coli isolates (n=12,253,679) among US outpatients between 2000 and 2010 was conducted using The Surveillance Network and found significant increases in the percentage of E. coli that were resistant to ciprofloxacin (3% to 17.1%) and trimethoprim-sulfamethoxazole (TMP-SXT) (17.9% to 24.2%), whereas there were minimal changes in the percentage of resistance to nitrofurantoin (0.8% to 1.6%) and ceftriaxone (0.2% to 2.3%) over time [Sanchez, 2012]. Another surveillance study, which looked at US susceptibility patterns and ESBL rates of E. coli from UTIs, showed an increase in ESBL rates from 7.8% to 18.3% (p<0.0001) from 2010 to 2014 [Lob, 2016]. The expansion of ESBL-producing E. coli, which are usually co-resistant to TMP-SXT and fluoroquinolones, is of urgent concern globally as well [Oteo, 2010]. Recent global surveillance data of E. coli showed high resistance rates to third-generation cephalosporins and fluoroquinolones in all 6 WHO regions [WHO, 2014]. An evaluation of the prevalence and susceptibility of acute cystitis pathogens in 9 European countries and Brazil from 2003 to 2006 showed that >10% of E. coli strains were MDR and 1.7% were ESBL producers [Schito, 2009]. A separate study in Brazil reported a prevalence of 7.6% ESBL-producing Enterobacterales among pathogens from community-acquired UTIs [Abreu, 2013]. In China, the prevalence of ESBLs in urinary E. coli in women ranged from 5% to 10.6% depending on the age group [Ho, 2007].

Based on these resistant pathogen trends, guidelines for acute cystitis now recommend first-line antibiotic treatment with nitrofurantoin, TMP-SXT, fosfomycin, or pivmecillinam, assuming the drug is available, and the patient does not have a concerning allergy history or tolerance issues [Gupta, 2011b]. Trimethoprim-sulfamethoxazole should not be used as a first-line treatment if the prevalence of resistance exceeds the 20% threshold or if TMP-SXT was used for treatment of a UTI in the previous 3 months. If any of these are concerns for a patient, then fluoroquinolones or β-lactams are recommended.

Gepotidacin is a first-in-class, novel triazaacenaphthylene antibacterial that has demonstrated in vitro activity against uropathogens including *E. coli* (see Section 4.2.1.2 of the IB for details) and provides high and sustained urine concentrations for the treatment of UTIs. With its unique ability to selectively inhibit bacterial DNA replication by a means not utilized by any currently approved human therapeutic agent, gepotidacin warrants further study as a potential opportunity to address an unmet medical need by providing a new and effective oral treatment option for acute cystitis.

A detailed description of the chemistry, pharmacology, efficacy, and safety of gepotidacin is provided in the IB. Details on the active comparator in this study, nitrofurantoin, may be found in the locally approved prescribing information.

## 2.3. Benefit/Risk Assessment

More detailed information about the known and expected benefits and risks and reasonably expected adverse events (AEs) of gepotidacin and nitrofurantoin may be found in the IB and the locally approved prescribing information, respectively.

# 2.3.1. Risk Assessment

| Potential Risk of Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Gepotidacin (GSK2140944) | | |
| Cardiovascular Effects Based on nonclinical data, cardiovascular effects were reversible increase in heart rate and blood pressure (dog and monkey); reversible 10 to 21 msec (4% to 9%) increase in QTc (monkey); and at the highest dose, a reversible 2 to 3 msec (6% to 8%) increase in QRS (monkey). Based on a thorough QTc clinical study, gepotidacin may cause mild, reversible heart rate effects and QT prolongation. | In a thorough QTc study, infusion of gepotidacin at doses of 1000 and 1800 mg over 2 hours caused a mild increased heart rate effect of approximately 6 to 10 bpm and QT prolongation measured as ΔΔQTcF of 12 to 22 msec. The QT prolongation evolved during the infusion and was quickly reversed over 2 hours after the end of the infusion (see Section 5.2.6 and Section 6 of the IB). In Phase I and II studies, concentration-dependent QT prolongation has been observed during clinical trials with gepotidacin; however, this increase has not translated into clinically significant QTc values or changes from baseline (change from baseline >60 msec or QTcF >500 msec) or cardiovascular AEs. In Phase I and II studies, gepotidacin did not have a clinically relevant effect on cardiac conduction (PR and QRS intervals). | See Section 5.2 for excluded cardiac conditions. Close monitoring of clinical parameters and AEs (Section 1.3) will be conducted, and treatment monitoring and evaluation criteria (Section 7.1.2) will be utilized to mitigate cardiovascular effects. Participants taking medications known to increase QT or potent CYP3A4 inhibitors will be excluded (see Section 6.5.2). See also the Renal and Hepatic sections within this table below. |

| Potential Risk of Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Gastrointestinal Effects Based on nonclinical data, gastrointestinal effects were mild ulceration of the nonglandular mucosa and minimal erosion and/or mural inflammation of the glandular mucosa in stomach (rat, oral study); moderate cecal ulceration and minimal colonic erosion (rat, IV study); and vomiting (dog). | See also the Acetylcholinesterase Inhibition section within this table below. Clostridium difficile-associated diarrhea has been observed in clinical trials with gepotidacin. | See Section 5.2 for excluded medical conditions. Close monitoring of clinical parameters and AEs (Section 1.3) will be conducted to mitigate and assess gastrointestinal effects. Suspected <i>C. difficile</i> infection will be managed according to a prespecified algorithm provided in Appendix 1. |
| Lower gastrointestinal effects (soft stools, flatulence, and diarrhea) are among the most common AEs reported in gepotidacin clinical studies. Nausea and vomiting AEs have also been commonly observed in gepotidacin clinical studies. | | |

212390

| Potential Risk of Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Acetylcholinesterase Inhibition In vitro testing showed gepotidacin to be a rapidly reversible inhibitor of acetylcholinesterase in the clinical plasma concentration range. Based on clinical data, caution should be used | Increased cholinergic effects can potentially be associated with more severe symptoms including atrioventricular block, seizure/convulsions, bronchospasm, and vasovagal syncope. No causal relationship between these events and the use of gepotidacin has been established during clinical trials to date. | Participants who have medical conditions or require medications that may be impacted by inhibition of acetylcholinesterase will be excluded from participation in this study. See Section 5.2 for excluded medical conditions and Section 6.5.2, Prohibited Medications and Nondrug Therapies, for prohibited medications. |
| in participants who have a condition requiring treatment with anticholinergic medications or who have certain medical conditions that may be exacerbated by the acetylcholinesterase inhibition activity of gepotidacin. | Adverse events consistent with acetylcholinesterase inhibition, including diarrhea, nausea, vomiting, gastrointestinal cramping and pain, dyspnea, bradycardia, lacrimation, salivation, and diaphoresis/sweating have been reported during clinical trials with gepotidacin. Mild and transient non-gastrointestinal AEs have been associated with Cmax levels higher than this dosing regimen. | Close monitoring of clinical parameters and AEs will be conducted to assess effects potentially related to acetylcholinesterase inhibition (Section 1.3). |
| Hepatic Effects In preclinical studies, increases in ALT, GLDH, alkaline phosphatase, and total bilirubin were observed in some rat studies of varying exposure. | Elevations in ALT have occurred in a few participants with pre-existing hepatitis C infection, but none were felt related to study treatment. The type and pattern of elevation in liver transaminases observed has not been suggestive of an adverse effect of gepotidacin and none were considered related to study treatment. A substantial increase in Cmax and AUC and decrease in clearance was observed in volunteer participants with severe hepatic impairment. | Participants with severe hepatic impairment are excluded from Phase III trials. See Section 5.2 for excluded medical conditions. Monitoring and stopping criteria liver events have been implemented. |

| Potential Risk of Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Renal Effects In preclinical trials, mild to moderate tubular degeneration was noted in the rat and proteinuria in the dog. Proteinuria was also observed in humans. | No clinical evidence of renal toxicity has been seen in clinical trials to date. A substantial increase in Cmax and AUC and decrease in clearance was observed in severe renal impairment/ESRD participants not on hemodialysis and in ESRD participants requiring hemodialysis (note: gepotidacin may have been administered at any time other than when receiving dialysis). | Participants with severe renal impairment/ESRD (including those who may require dialysis) are excluded from Phase III trials. See Section 5.2 for excluded medical conditions. Monitoring criteria have been implemented. |

| Potential Risk of Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Reproductive System Effects Preclinical studies demonstrated that gepotidacin was not genotoxic and no drug-related malformations were observed. Although positive in vitro findings for clastogenicity, consistent with a mechanism related to mammalian topoisomerase II inhibition were found, in vivo data from rat micronucleus and COMET assays suggest that gepotidacin does not pose a genotoxic hazard to humans. | There are no data on the use of gepotidacin in pregnant women. | Gepotidacin is contraindicated in pregnant or nursing mothers and women of childbearing potential who are not employing adequate contraceptive measures. See Appendix 2 for contraceptive measures and Appendix 8 for required pregnancy testing. |
| Gepotidacin effects on embryofetal development were limited to decreased fetal weights for male and female fetuses in rats and decreased fetal weights and increased fetal resorptions (fetal deaths) in mice, both at maternally toxic doses. These occurred at clinically relevant exposures (65 µg.h/mL in rat and 35 µg.h/mL in mouse). | | |

| Potential Risk of Clinical Significance | Mitigation Strategy | |
|---|---|---|
| Other Control of the | | |
| Nitrofurantoin | The most frequent AEs possibly or probably related to oral nitrofurantoin treatment are nausea (8%), headache (6%), and flatulence (1.5%). As with gepotidacin, there is also a need to monitor for <i>C. difficile</i> -associated diarrhea during nitrofurantoin treatment. | Close monitoring of clinical parameters and AEs (Section 1.3) will be conducted, and treatment monitoring and evaluation criteria (Section 7.1.1) will be utilized to mitigate hepatic effects. |
| | Nitrofurantoin is contraindicated for patients with anuria, oliguria, or significant impairment of renal | Because planned treatment in this study is only 5 days, the probability for adverse reactions associated with long-term use is low. |
| 42 wh un prody Rapa lor rech produced be more than the control of | function; pregnant patients at term (38 to 42 weeks' gestation), during labor and delivery, or when the onset of labor is imminent; neonates under 1 month of age; and patients with a previous history of cholestatic jaundice/hepatic dysfunction associated with nitrofurantoin. | The exclusion criteria for this study include contraindications to nitrofurantoin use and exclude participants at risk for nitrofurantoin adverse reactions, including acute porphyria as an example of a rare genetic risk (see Section 5.2). |
| | Rare adverse reactions that generally occur in patients receiving treatment for 6 months or longer are acute, subacute, or chronic pulmonary reactions, with potential insidious development of chronic pulmonary reactions (diffuse interstitial pneumonitis or pulmonary fibrosis, or both). | Participants with a history of sensitivity to nitrofurantoin, or components thereof, will not be allowed to enroll in the study (Section 5.2). Participant's medical history will be carefully evaluated for history of hypersensitivity. |
| | Peripheral neuropathy has occurred, which may be enhanced for patients with anemia, diabetes mellitus, electrolyte imbalance, vitamin B deficiency, and debilitating disease. | Participants must agree not to use antacid preparations containing magnesium trisilicate or uricosuric drugs during study treatment (see Section 5.2). |
| | Nitrofurantoin has induced the occurrence of hemolytic anemia of the primaquine-sensitivity | |

| Potential Risk of Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| | type, which appear to be linked to a glucose-6-phosphate dehydrogenase deficiency in the red blood cells of the affected patients. | Suspected <i>C. difficile</i> infection will be managed according to a prespecified algorithm provided in Appendix 1. |
| | Hepatic reactions, including hepatitis, cholestatic jaundice, chronic active hepatitis, and hepatic necrosis, occur rarely. | Precautions related to nitrofurantoin are summarized in detail in the Study Reference Manual. |
| | Concomitant administration of nitrofurantoin with antacids containing magnesium trisilicate reduces both the rate and extent of absorption, and uricosuric drugs, such as probenecid and sulfinpyrazone, can inhibit renal tubular secretion of nitrofurantoin. | |
| | Refer to locally approved nitrofurantoin prescribing information for specific details relating to nitrofurantoin. | |

bpm=beats per minute; AE=adverse event; ALT=alanine aminotransferase; AUC=area under the drug concentration-time curve; Cmax=maximum concentration; CYP3A4=cytochrome P450 enzyme 3A4; ESRD=end-stage renal disease; GLDH=glutamate dehydrogenase; IB=investigator's brochure; IV=intravenous; \( \Delta \text{QTCF} = \text{placebo-corrected change from baseline in corrected QT interval using the Fridericia formula; QTc=corrected QT interval; QTcF=interval corrected for heart rate according to Fridericia's formula. TMF-13817737 212390

#### 2.3.2. **Benefit Assessment**

Acute cystitis is among the most common indications for which antimicrobials are prescribed for otherwise healthy women [Gupta, 2011b]. The increase in antimicrobial resistance among pathogens causing community-acquired UTIs over the past 2 decades has made treatment approaches for UTIs more difficult. Gepotidacin is active in vitro and in vivo against the key causative pathogen in acute cystitis, E. coli, including most isolates resistant to other antibacterial treatments. Given gepotidacin's spectrum of activity against E. coli, S. saprophyticus, and E. faecalis, as well as human safety data and the PK profile, it is anticipated that gepotidacin will benefit participants with acute cystitis.

The active comparator in this study is nitrofurantoin, a marketed antibiotic for the treatment acute uncomplicated UTIs (acute cystitis) caused by susceptible strains of E. coli or S. saprophyticus (refer to locally approved nitrofurantoin prescribing information). Participants randomly assigned to this treatment group are also expected to experience treatment benefits. It is expected that gepotidacin will have a similar efficacy profile to nitrofurantoin.

Overall, all participants in this study will not only receive routine medical monitoring appropriate for acute cystitis, but they will also receive heightened monitoring to minimize safety risks when participating in a clinical study.

#### 2.3.3. **Overall Benefit: Risk Conclusion**

Antimicrobial resistance among uropathogens causing acute cystitis has increased in the past decades [Gupta, 2011b; Sanchez, 2016]. However, even in the face of increasing drug resistance to existing agents, few new antibiotics with novel mechanisms of action are being developed. Gepotidacin selectively inhibits bacterial DNA replication by a means not utilized by any currently approved human therapeutic agent. Based on the known preclinical data for gepotidacin against E. coli, S. saprophyticus, and E. faecalis, the Phase II results showing the efficacious treatment of uncomplicated urogenital gonorrhea and ABSSSIs, Phase IIa results indicating efficacy in acute cystitis, and the cumulative safety results from Phase I and Phase II studies with oral gepotidacin treatment, this study will test whether gepotidacin is noninferior to 1 of the current recommended treatments and thus represents a potential new treatment option for acute cystitis.

None of the potential or identified risks seen to date in participants dosed with gepotidacin preclude further clinical development. Mitigation strategies have been implemented to promptly identify and appropriately address risks in order to protect participant safety and to better characterize the safety profile of the study treatments (Section 2.3.1). Furthermore, a GlaxoSmithKline (GSK) Safety Review Team (SRT) will monitor blinded safety data instream (see Appendix 3). Careful safety monitoring should also identify any emerging safety issues for gepotidacin and contribute to the benefit-risk profile of nitrofurantoin.

The investigator may also, at his or her discretion, discontinue the participant from study treatment at any time and initiate appropriate alternative therapy.

TMF-13817737 212390

Taking into account the measures taken to minimize risk to participants participating in this study, the potential risks identified in association with gepotidacin and nitrofurantoin are justified by the anticipated benefits that may be afforded to participants with acute cystitis.

#### **OBJECTIVES AND ESTIMANDS/ENDPOINTS** 3.

| Objectives | Endpoints |
|---|---|
| To assess the combined clinical and microbiological efficacy of gepotidacin compared to nitrofurantoin, at the TOC Visit, in female participants with acute cystitis with qualifying bacterial uropathogen(s) at Baseline that all are susceptible to nitrofurantoin | Therapeutic response (combined per-participant microbiological and clinical response) at the TOC Visit |
| Secondary | |
| To assess the clinical efficacy of<br>gepotidacin compared to nitrofurantoin, at<br>the TOC and Follow-up Visits, in female<br>participants with acute cystitis | Clinical outcome and response at the TOC and Follow-up Visits |
| To assess the clinical efficacy of<br>gepotidacin compared to nitrofurantoin, at<br>the TOC and Follow-up Visits, in female<br>participants with acute cystitis with<br>qualifying bacterial uropathogen(s) at<br>Baseline that all are susceptible to<br>nitrofurantoin | Clinical outcome and response at the TOC and Follow-up Visits |
| To assess the microbiological efficacy of gepotidacin compared to nitrofurantoin, at the TOC and Follow-up Visits, in female participants with acute cystitis with qualifying bacterial uropathogen(s) at Baseline that all are susceptible to nitrofurantoin | Microbiological outcome and response at<br>the TOC and Follow-up Visits |
| To assess the combined clinical and microbiological efficacy of gepotidacin compared to nitrofurantoin, at the Follow-up Visit, in female participants with acute cystitis with qualifying bacterial uropathogen(s) at Baseline that all are susceptible to nitrofurantoin | Therapeutic response (combined per-participant microbiological and clinical response) at the Follow-up Visit |

| Objectives | Endpoints |
|---|---|
| Secondary continued | |
| <ul> <li>To assess the safety and tolerability of<br/>gepotidacin compared to nitrofurantoin in<br/>female participants with acute cystitis</li> </ul> | Treatment-emergent AEs and serious<br>AEs (SAEs) and change from baseline<br>results for clinical laboratory tests,<br>electrocardiograms (ECGs), and vital sign<br>measurements |
| CCI | |

| Objectives | Endpoints |
|------------|-----------|
| CCI | |

# Primary Estimand

The primary clinical question of interest is: What is the treatment effect on the therapeutic response after 5 days of treatment with gepotidacin 1500 mg twice daily compared to 5 days of treatment with nitrofurantoin 100 mg twice daily in participants with acute cystitis with qualifying bacterial uropathogen(s) at Baseline that all are susceptible to nitrofurantoin, regardless of treatment discontinuation for any reason. Receipt of systemic antimicrobials will impact the endpoint definition (see Section 8.1.2.1 and Section 8.1.3.1).

The primary estimand is described by the following attributes:

- Population: Female participants with acute cystitis with qualifying bacterial uropathogen(s) at Baseline that all are susceptible to nitrofurantoin.
- Treatment condition: Gepotidacin 1500 mg twice daily for 5 days versus nitrofurantoin 100 mg twice daily for 5 days, regardless of adherence.
- Variable: Therapeutic response (combined per-participant microbiological and clinical response) at the TOC Visit. Microbiological success is defined as eradication (i.e., reduction) of all qualifying bacterial uropathogens recovered at baseline to <10<sup>3</sup> colony-forming units/mL (CFU/mL) as observed on quantitative urine culture without the participant receiving other systemic antimicrobials. Clinical success is defined as resolution of signs and symptoms of acute cystitis present at Baseline (and no new signs and symptoms) without the participant receiving other systemic antimicrobials.
- Summary measure: Absolute difference in the therapeutic success rate in the gepotidacin and nitrofurantoin treatment groups.
- Intercurrent events (ICEs):
  - Study treatment discontinuation (due to any reason) treatment policy strategy (interest is in the treatment effect regardless of study treatment discontinuation).
  - Use of systemic antimicrobials composite strategy. This ICE is captured through the definitions of microbiological and clinical response (see Section 8.1.2.1 and Section 8.1.3.1) and will be counted as therapeutic failures.

### Rationale for Estimand:

Interest lies in the treatment effect regardless of whether the full course of 5 days of treatment was taken or not, which reflects how patients may be treated in clinical practice. Hence, a treatment policy strategy is appropriate for treatment withdrawal before completing 5 days of treatment. Use of other systemic antimicrobials may

confound the bacterial culture results; thus, the microbiological response will be considered failure. For clinical data, the use of a systemic antimicrobial for acute cystitis is a sign of treatment failure and use of a systemic antimicrobial for another infection cannot be considered a success as it confounds the assessment of efficacy. Therefore, the definition of a successful therapeutic response precludes the use of other systemic antimicrobials.

212390

## Secondary Estimands:

The secondary clinical questions of interest are: What is the treatment effect on each of the secondary efficacy endpoints after 5 days of treatment with gepotidacin 1500 mg twice daily compared to 5 days of treatment with nitrofurantoin 100 mg twice daily in participants with acute cystitis (clinical endpoints) and in participants with acute cystitis with qualifying bacterial uropathogen(s) at Baseline that all are susceptible to nitrofurantoin (therapeutic, clinical, and microbiological endpoints), regardless of treatment discontinuation for any reason. Receipt of systemic antimicrobials impacts the endpoint definition (see Section 8.1.2.1 and Section 8.1.3.1).

For each of the secondary endpoints the estimand will follow a similar approach to the estimand for the primary endpoint and will use the same strategies for the ICEs. The exception is the summary measure for the outcome endpoints. These endpoints are descriptively summarized; therefore, the summary measure will be the percentage in each clinical and microbiological outcome category in the gepotidacin and nitrofurantoin arms separately (as no direct comparison between treatment groups will be made) (see Section 8.1.2.1 and Section 8.1.3.1 for endpoint definitions).

The safety endpoint will use a treatment policy strategy of the ICE of withdrawal from treatment as the safety will be assessed at all postbaseline assessments irrespective of whether the participant completed the treatment.

Components of estimand for all secondary endpoints are listed in Table 1.

Table 1 Estimand for the Secondary Endpoints

| Secondary<br>Endpoint | Population | Treatment Condition | Variable | Summary Measure | Intercurrent Event |
|---|---|---|---|---|---|
| Clinical response at<br>the TOC and<br>Follow-up Visits | Female participants with acute cystitis | Gepotidacin 1500 mg<br>BID for 5 days versus<br>nitrofurantoin 100 mg<br>BID for 5 days,<br>regardless of<br>adherence | See Table 10 and Table 11 | Absolute difference in the clinical success rate in the gepotidacin and nitrofurantoin treatment groups | Study treatment discontinuation (due to any reason) – treatment policy Use of systemic antimicrobials – composite strategy |
| Clinical outcome at<br>the TOC and<br>Follow-up Visits | Female participants with acute cystitis | Gepotidacin 1500 mg<br>BID for 5 days versus<br>nitrofurantoin 100 mg<br>BID for 5 days,<br>regardless of<br>adherence | See Table 10 and Table 11 | Percentage of participants in each outcome category in the gepotidacin and nitrofurantoin arms separately | Study treatment discontinuation (due to any reason) – treatment policy Use of systemic antimicrobials – composite strategy |
| Clinical response at<br>the TOC and<br>Follow-up Visits | Female participants with acute cystitis with qualifying bacterial uropathogen(s) at Baseline that all are susceptible to nitrofurantoin | Gepotidacin 1500 mg<br>BID for 5 days versus<br>nitrofurantoin 100 mg<br>BID for 5 days,<br>regardless of<br>adherence | See Table 5 | Absolute difference in the clinical success rate in the gepotidacin and nitrofurantoin treatment groups | Study treatment discontinuation (due to any reason) – treatment policy Use of systemic antimicrobials – composite strategy |
| Clinical outcome at<br>the TOC and<br>Follow-up Visits | Female participants with acute cystitis with qualifying bacterial uropathogen(s) at baseline that all are susceptible to nitrofurantoin | Gepotidacin 1500 mg<br>BID for 5 days versus<br>nitrofurantoin 100 mg<br>BID for 5 days,<br>regardless of<br>adherence | See Table 5 | Percentage of participants in each outcome category in the gepotidacin and nitrofurantoin arms separately | Study treatment discontinuation (due to any reason) – treatment policy Use of systemic antimicrobials – composite strategy |

| Secondary<br>Endpoint | Population | Treatment Condition | Variable | Summary Measure | Intercurrent Event |
|---|---|---|---|---|---|
| Microbiological response at the TOC and Follow-up Visits | Female participants with acute cystitis with qualifying bacterial uropathogen(s) at Baseline that all are susceptible to nitrofurantoin | Gepotidacin 1500 mg<br>BID for 5 days versus<br>nitrofurantoin 100 mg<br>BID for 5 days,<br>regardless of<br>adherence | See Table 5 | Absolute difference in the microbiological success rate in the gepotidacin and nitrofurantoin treatment groups | Study treatment discontinuation<br>(due to any reason) – treatment<br>policy<br>Use of systemic antimicrobials –<br>composite strategy |
| Microbiological outcome at the Follow-up Visit | Female participants with acute cystitis with qualifying bacterial uropathogen(s) at Baseline that all are susceptible to nitrofurantoin | Gepotidacin 1500 mg<br>BID for 5 days versus<br>nitrofurantoin 100 mg<br>BID for 5 days,<br>regardless of<br>adherence | See Table 5 | Percentage of participants in each outcome category in the gepotidacin and nitrofurantoin arms separately | Study treatment discontinuation<br>(due to any reason) – treatment<br>policy<br>Use of systemic antimicrobials –<br>composite strategy |
| Therapeutic response at the Follow-up Visit | Female participants with acute cystitis with qualifying bacterial uropathogen(s) at Baseline that all are susceptible to nitrofurantoin | Gepotidacin 1500 mg<br>BID for 5 days versus<br>nitrofurantoin 100 mg<br>BID for 5 days,<br>regardless of<br>adherence | See Table 5 and Table 11 | Absolute difference in the therapeutic success rate in the gepotidacin and nitrofurantoin treatment groups | Study treatment discontinuation<br>(due to any reason) – treatment<br>policy<br>Use of systemic antimicrobials –<br>composite strategy |
| Safety | Female participants with acute cystitis infection | Gepotidacin 1500 mg<br>BID for 5 days versus<br>nitrofurantoin 100 mg<br>BID for 5 days,<br>regardless of<br>adherence | TEAEs, SAEs, as well as change from baseline results for clinical laboratory tests, ECGs, and vital sign measurements | Summary statistics (appropriate for each type of endpoint) in the gepotidacin and nitrofurantoin arms separately | Study treatment discontinuation (due to any reason) – treatment policy |

BID=twice daily; EGG=electrocardiogram; SAE=serious adverse event; TEAE=treatment-emergent adverse event; TOC=Test-of-Cure.

TMF-13817737 212390

#### 4. STUDY DESIGN

#### 4.1. Overall Design

- Study 212390 is a Phase III, randomized, multicenter, parallel-group, double-blind, double-dummy, comparator-controlled, noninferiority study in adolescent and adult female participants comparing the efficacy and safety of oral gepotidacin to oral nitrofurantoin in the treatment of uncomplicated UTI (acute cystitis).
- Participants will be stratified by age category (<18 years, ≥18 to 50 years, or >50 years) and acute cystitis recurrence (nonrecurrent infection or recurrent infection, defined as a confirmed infection [not including the current infection in the calculation] with at least 1 prior episode within the past 3 months, at least 2 prior episodes within the past 6 months, or at least 3 prior episodes within the past 12 months before study entry) and will be randomly assigned in a 1:1 ratio to receive 1 of the following study treatments:
  - Gepotidacin: 1500 mg administered orally twice daily (BID) for 5 days (Note: Each dose should be taken after food consumption and with water to assist with tolerability.)
  - Nitrofurantoin: 100 mg administered orally BID for 5 days (Note: Each dose should be taken after food consumption and with water.)
- Appropriate safety, efficacy, and microbiological assessments will be conducted at the Baseline (Day 1) Visit and repeated at the On-therapy (Day 2 to 4), TOC (Day 10 to 13), and Follow-up (Day 28±3) Visits.

Each treatment day will be assessed over 24 hours starting with the first dose of study treatment, as further detailed in the Study Reference Manual (SRM).

- For the primary efficacy endpoint of the apeutic response (combined per-participant microbiological and clinical response), therapeutic success refers to participants who have been deemed both a microbiological success (reduction of all qualifying bacterial uropathogens [e.g., ≥10<sup>5</sup> CFU/mL; defined in Appendix 4] recovered at Baseline to <10<sup>3</sup> CFU/mL as observed on quantitative urine culture without the participant receiving other systemic antimicrobials) and a clinical success (resolution of signs and symptoms of acute cystitis present at Baseline [and no new signs and symptoms] without the participant receiving other systemic antimicrobials) at the TOC Visit in the Microbiological Intent-to-Treat Nitrofurantoin-Susceptible (micro-ITT NTF-S) Population, regardless of treatment discontinuation. The TOC Visit is 10 to 13 days after randomization, which is also 5 to 8 days after completion of study treatment.
- Participants may return to the study site at any time due to AEs or if they are experiencing new or continuing signs and symptoms of acute cystitis. Participants will be assessed and treated per the investigator's judgement. If a participant is switched to a different antibiotic before or during the TOC Visit, all TOC procedures should be completed before the other antibiotic is started.
- Participants with a concomitant fungal infection can only be treated with topical antifungals per local standard of care.
- Participants will return to the study site on Day 28  $(\pm 3)$  for a Follow-up Visit. Participants experiencing signs and symptoms suggestive of infection recurrence or relapse will be assessed and treated per the investigator's judgement.
- The duration of study participation is approximately 28 days with 4 planned study visits (see Section 8 for study visit details):
  - Baseline (Day 1) Visit
  - On-therapy (Day 2 to 4) Visit
  - TOC (Day 10 to 13) Visit
  - Follow-up (Day 28±3) Visit

A study design schematic is depicted in Figure 1. The Schedule of Activities (SoA) is provided is Section 1.3.

Refer to Appendix 5 for details regarding allowed revisions to study conduct and/or monitoring due to coronavirus disease (COVID-19). For all study visits, to minimize the amount of time that participants spend at the clinic, eConsent may be utilized and remote collection of study-related data may be obtained as described in the SRM. Thus, some visit data may be collected through a combination of telemedicine and on-site visits. Collection of information via telemedicine will be performed only where local regulations permit.

Of note, to reduce participant on-site visits or if unforeseen issues impact clinic visits, and participants are unable to attend a site visit, home healthcare (home visits and telemedicine visits) may be used to conduct procedures as detailed in the Study Reference Manual. Home healthcare will only be utilized where applicable country and local regulations and infrastructure allow.

### 4.2. Scientific Rationale for Study Design

The study design is based on the Food and Drug Administration (FDA) guidance for industry for developing drug treatments for uncomplicated and complicated UTIs [DHHS, 2019; DHHS, 2018], the European Medicines Agency (EMA) addendum to the guideline on the evaluation of medicinal products indicated for treatment of bacterial infections [EMA, 2013], and feedback from the FDA and EMA. The primary efficacy endpoint will be the therapeutic response (combined per-participant microbiological and clinical response) at the TOC Visit (i.e., 10 to 13 days after randomization, which is also 5 to 8 days after completion of study treatment) in participants who have a qualifying bacterial uropathogen at Baseline. Although the guidances differ in their criteria for defining qualifying uropathogens, this study has been designed with the qualifying uropathogen criteria defined in Appendix 4 and microbiological success defined as reduction of all qualifying bacterial uropathogens recovered at Baseline to <10<sup>3</sup> CFU/mL as observed on quantitative urine culture without the participant receiving other systemic antimicrobials. Clinical success at the TOC Visit is defined as the resolution of signs and symptoms of acute cystitis present at Baseline (and no new signs and symptoms) without

the participant receiving other systemic antimicrobials. Therapeutic success refers to participants who have been deemed both a microbiological success and a clinical success (i.e., responders).

212390

Nitrofurantoin has been selected as the active comparator in this study. Nitrofurantoin is an approved treatment that is indicated for the treatment of acute uncomplicated UTI (acute cystitis) caused by susceptible strains of *E. coli* or *S. saprophyticus* (refer to locally approved prescribing information). It is globally available in most regions and is a recommended oral first-line treatment for acute cystitis per current US, UK, and European Association of Urology guidelines [Gupta, 2011b; NICE, 2019; EAU, 2019]. Both gepotidacin and nitrofurantoin will be administered BID for a treatment duration of 5 days. As described in Section 4.3, the dose of each study treatment and the 5-day duration were selected to provide efficacious treatment for acute cystitis and is in alignment with current clinical practice. Having the same dose regimen will also support double-blind dose administration. A noninferiority margin of 10% has been selected for this study [DHHS, 2019].

Both adult and adolescent (≥12 to <18 years of age) eligible female participants will be enrolled in this double-blinded study. The study is restricted to female participants per FDA guidance [DHHS, 2019]. Adolescent participants will only be enrolled at study sites where investigators have experience in this population and if allowed per the study site's institutional ethics committees and local country/national regulatory guidelines and enrollment will be contingent upon such approvals. Adolescent assent forms and adult consent forms will be developed with oversight from local governing institutional review boards (IRBs)/independent ethics committees (IECs) (see Appendix 3). There is no upper age limit for study participants; however, participants are excluded if they reside in a nursing home or dependent care type-facility, or if they have any comorbidities associated with complicated UTI. Thus, any participants >75 years of age will only be eligible for the study if they are residing independently.

In order to maximize the efficiency of this study while minimizing discomfort and inconvenience to participants consenting to this protocol, a GSK SRT will monitor blinded safety data instream, while a Microbiology Review Team will monitor blinded uropathogen identification and susceptibility data instream, including the enrollment rate of participants with a qualifying bacterial uropathogen at Baseline and the resistance profile of uropathogens. For details on these review teams, refer to Appendix 3. In addition, an Independent Data Monitoring Committee (IDMC) will manage the interim analysis (IA) as described in Section 9.5.

## 4.3. Justification for Dose

The oral gepotidacin dose in this study is 1500 mg BID (total daily dose of 3000 mg) for 5 days. A 5-day dosing duration is in alignment with current treatment guidelines for efficacious antibacterial treatment of uncomplicated acute cystitis in women, which typically ranges from 3 to 7 days [Gupta, 2011b; NICE, 2019; EAU, 2019]. The safety and tolerability at this oral dose and duration have been evaluated in Phase I studies and in Phase II studies (BTZ116704 and 206899) (see Section 5 of the IB for details).

Furthermore, high urine concentrations of gepotidacin are expected in this study based on a healthy volunteer Phase I study (BTZ117351) and a Phase IIa study in participants with acute cystitis (206899). In BTZ117351, approximately 287 mg of unchanged gepotidacin was excreted in urine after a single oral 1500-mg (2  $\times$  750-mg tablets) dose of gepotidacin (minimum urine area under drug concentration-time curve over 12 hours [AUC12h]=807  $\mu g.h/mL$ ). In the Phase IIa study, 206899, in participants with uncomplicated UTIs, approximately 460 mg of unchanged gepotidacin was excreted in urine over the steady-state dosing interval of 12 hours after repeat BID oral dosing of 1500 mg (2  $\times$  750-mg tablets) gepotidacin (minimum steady-state urine AUC12h=2256  $\mu g.h/mL$ ).

The gepotidacin dose and duration for this study were selected based on in vitro and in vivo studies including experimental animal pyelonephritis studies that simulated human PK exposures of gepotidacin to determine the efficacy of gepotidacin against isolates of *E. coli*, including MDR strains (see Section 4.2 of the IB for further details). Based on GSK assessment of the limitations of the current acute cystitis efficacy model in rodents, the pyelonephritis model is considered to allow evaluation of antibacterial efficacy in a more robust UTI.

Additionally, an in vitro study to determine the PK/pharmacodynamic (PD) characteristics of gepotidacin against  $E.\ coli$  (dose-fractionation and dose-ranging studies) indicate that AUC/MIC is the primary PK/PD index predictive of gepotidacin efficacy against  $E.\ coli$ . The magnitude of the ratio of free-drug AUC to MIC over 24 hours (fAUC/MIC) required to achieve net bacterial stasis as well as 1- and 2-log reductions in bacterial burden from Baseline across multiple  $E.\ coli$  isolates with gepotidacin MIC values ranging from 1 to 4  $\mu$ g/mL, were 34.5, 41.3, and 49.7, respectively.

A set of duplicate 10-day hollow fiber infection model studies was also completed using  $E.\ coli$  isolate NCTC 13441 to determine the fAUC/MIC exposure of gepotidacin required to prevent the amplification of a resistant subpopulation. An inverted-U shaped function described the relationship between drug resistance amplification and fAUC, with fAUC values  $\geq 549$  preventing resistance amplification to gepotidacin for  $E.\ coli$  in the hollow fiber infection model for 10 days. This equates to an fAUC/MIC value  $\geq 275$  when applying the gepotidacin broth microdilution MIC of 2  $\mu g/mL$  for  $E.\ coli$  13441, as determined in this study.

When taking the fAUC/MIC target of 275 for resistance suppression into consideration with the concentrations of gepotidacin in human urine measured in BTZ117351 (minimum urine AUC12h=807 µg.h/mL; thus, minimum urine AUC over 24 hours [AUC24h]=1614 µg.h/mL) and applying an MIC value of 4 µg/mL, the minimum human urine AUC/MIC achieved for the 1500 mg oral BID dose exceeds the fAUC/MIC resistance suppression target of 275 by approximately 1.5-fold and 100% target attainment for a urine AUC/MIC target of 275 would be expected for participants with  $E.\ coli$  isolates with gepotidacin MICs  $\leq$ 4 µg/mL following 1500 mg BID oral dosing.

When applying the higher concentrations of gepotidacin in human urine measured in the Phase IIa study (206899; minimum urine AUC12h=2256  $\mu$ g.h/mL; thus,

AUC24h=4512 µg.h/mL) and applying a MIC value of 4 µg/mL, the minimum human urine AUC/MIC achieved for the 1500 mg oral BID dose further exceeds the fAUC/MIC resistance suppression target of 275 by approximately 4-fold and 100% target attainment for a urine AUC/MIC target of 275 would also be expected for participants with E. coli isolates with gepotidacin MICs  $\leq$ 4 µg/mL following 1500 mg BID oral dosing.

212390

Additionally, in the Phase IIa study (206899), for 4 participants with available urine AUC24h steady-state PK parameters and qualifying Enterobacterales uropathogens who were microbiological successes at TOC, the plasma fAUC24h/MIC values ranged from 7 to 90.5 and urine AUC24h/MIC ratios ranged from 1292 to 121,698. The participant with the lowest plasma fAUC/MIC (7.0) and urine AUC/MIC (1292) had a K. pneumoniae uropathogen with a gepotidacin MIC of 4  $\mu$ g/mL. No participants had an outcome of microbiological persistence at TOC.

In conclusion, minimum urine levels of gepotidacin are anticipated to be in excess of the fAUC/MIC target necessary for both efficacy and resistance suppression for *E. coli* as determined from the in vitro PK/PD models. Given that the bladder is the primary site of infection in cystitis, the use of gepotidacin urine PK data, coupled with the robust in vivo efficacy demonstrated in the Phase IIa uncomplicated UTI study and human simulated PK pyelonephritis model, is appropriate for selecting the gepotidacin 1500 mg BID oral dose for 5 days for study in the treatment of participants with acute cystitis.

In addition, a PK evaluation (Study 209611) in healthy adult and adolescent participants has been completed (see Section 5 of the IB for further details). Overall, plasma Cmax values were 27% higher in adolescents; however, the range of Cmax values were similar, and AUC(0-∞) values were similar for adults and adolescents following a 1500-mg single gepotidacin dose. Following the first of two 3000 mg gepotidacin doses 6 hours apart, Cmax values were 29% higher in adolescents; however, the ranges of Cmax values were similar, and following the second dose for adults and adolescents Cmax values were similar. The AUC(0-τ) was approximately 35% higher in adolescents following both doses compared to adults. The total amount of gepotidacin excreted in urine was similar in adult and adolescent participants following a 1500-mg single gepotidacin dose. Following two 3000 mg gepotidacin doses given 6 hours apart, the total amount excreted was approximately 35% higher in adolescents compared to adults. The maximum dose of gepotidacin evaluated in adolescents was 3000 mg given as 2 doses 6 hours apart. Across the age groups, the safety-risk profile was similar.

The oral nitrofurantoin dose in this study is 100 mg BID (total daily dose of 200 mg) for 5 days. This oral dose and duration of nitrofurantoin is within the prescribed labeling recommendations, which is 100 mg BID for up to 7 days for adults and pediatric patients over 12 years of age (refer to locally approved prescribing information). The labeled 7-day dosing duration of nitrofurantoin was based on clinical registration studies from several decades ago. More recently, a 5-day dosing duration of nitrofurantoin was shown to be efficacious for the treatment of uncomplicated acute cystitis in women [Gupta, 2007] and a treatment duration of <7 days for nitrofurantoin is in alignment with current treatment guidelines [Gupta, 2011b; NICE, 2019; EAU, 2019].

## 4.4. End-of-Study Definition

A participant is considered to have completed study treatment if she has taken all doses of the randomly assigned study treatment and completed the TOC Visit. A participant is considered to have completed the study if she has completed all study visits including the Follow-up Visit.

The end of the study is defined as the date of the last visit of the last participant in the study.

## 5. STUDY POPULATION

Prospective approval of protocol deviations to recruitment and enrollment criteria, also known as protocol waivers or exemptions, is not permitted.

## 5.1. Inclusion Criteria

Otherwise healthy participants are eligible to be included in the study only if all of the following criteria apply:

## Age

1. The participant is  $\ge 12$  years of age at the time of signing the informed consent/assent and has a body weight  $\ge 40$  kg.

**Note**: Although participants as young as 12 years may enroll in the study, study sites must follow their institutional ethics committee and local country/national regulatory guidelines and enrollment will be contingent upon such approvals regarding the allowed lower age limit for clinical study participants.

## Type of Participant and Disease Characteristics

- 2. The participant has 2 or more of the following clinical signs and symptoms of acute cystitis with onset <96 hours prior to study entry: dysuria, frequency, urgency, or lower abdominal pain (see Appendix 6).
- 3. The participant has nitrite or pyuria (>15 WBC/HPF or the presence of 3+/large leukocyte esterase) from a pretreatment clean-catch midstream urine sample based on local laboratory procedures.

## Sex

4. The participant is female.

Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

• A female participant is eligible to participate if she is a woman of childbearing potential (WOCBP) who is not pregnant as confirmed by a high sensitivity urine pregnancy test at Baseline (Day 1) regardless of current or prior contraception use or abstinence, is not breastfeeding, or is not a WOCBP.

**Note:** Pregnancy testing requirements, contraceptive guidance, and WOCBP definitions are provided in Appendix 2 and requirements for pregnancy testing during and after study treatment are located in Appendix 8.

- Additional requirements for pregnancy testing during and after study treatment are located in Appendix 8.
- The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.

### **Informed Consent**

5. The participant is capable of giving signed informed consent/assent as described in Appendix 3 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF)/assent form and in this protocol.

## 5.2. Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

### **Medical Conditions**

- 1. The participant resides in a nursing home or dependent care type-facility.
- 2. The participant has a body mass index ≥40.0 kg/m² or a body mass index ≥35.0 kg/m² and is experiencing obesity-related health conditions such as uncontrolled high blood pressure or uncontrolled diabetes.
- 3. The participant has a history of sensitivity to the study treatments, or components thereof, or a history of a drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates her participation.
- 4. The participant is immunocompromised or has altered immune defenses that may predispose the participant to a higher risk of treatment failure and/or complications (e.g., uncontrolled diabetes, renal transplant recipients, participants with clinically significant persistent granulocytopenia [absolute neutrophil count <1000/μL], and participants receiving immunosuppressive therapy, including corticosteroid therapy [>40 mg/day prednisolone or equivalent for >1 week, ≥20 mg/day prednisolone or equivalent for >2 weeks, or prednisolone or equivalent ≥10 mg/day for >6 weeks]). Participants with a known CD4 count of <200 cells/mm³ should not be enrolled.
- 5. The participant has any of the following:
  - Medical condition that requires medication that may be impacted by inhibition of acetylcholinesterase, such as:
    - Poorly controlled asthma or chronic obstructive pulmonary disease at Baseline and, in the opinion of the investigator, not stable on current therapy
    - Acute severe pain, uncontrolled with conventional medical management
    - Active peptic ulcer disease

- Parkinson disease
- Myasthenia gravis
- A history of seizure disorder requiring medications for control (this does not include a history of childhood febrile seizures)

212390

OR

- Known acute porphyria
- Any surgical or medical condition (active or chronic) that may interfere with drug absorption, distribution, metabolism, or excretion of the study treatment (e.g., ileostomy or malabsorption syndrome)
- The participant has a known glucose-6-phosphate dehydrogenase deficiency.
- The participant, in the judgment of the investigator, would not be able or willing to comply with the protocol or complete study follow-up.
- The participant has a serious underlying disease that could be imminently lifethreatening, or the participant is unlikely to survive for the duration of the study period.

## Urinary Tract Infection/Renal/Urogenital Exclusions

- The participant has acute cystitis that is known or suspected to be due to fungal, parasitic, or viral pathogens; or known or suspected to be due to *Pseudomonas* aeruginosa or Enterobacterales (other than E. coli) as the contributing pathogen.
- 10. The participant has symptoms known or suspected to be caused by another disease process, such as asymptomatic bacteriuria, overactive bladder, chronic incontinence, or chronic interstitial cystitis, that may interfere with the clinical efficacy assessments or preclude complete resolution of acute cystitis symptoms.
- 11. The participant has an anatomical or physiological anomaly that predisposes the participant to UTIs or may be a source of persistent bacterial colonization, including calculi, obstruction or stricture of the urinary tract, primary renal disease (e.g., polycystic renal disease), or neurogenic bladder, or the participant has a history of anatomical or functional abnormalities of the urinary tract (e.g., chronic vesico-ureteral reflux, detrusor insufficiency).
- 12. The participant has an indwelling catheter, nephrostomy, ureter stent, or other foreign material in the urinary tract.
- 13. The participant who, in the opinion of the investigator, has an otherwise complicated UTI, an active upper UTI (e.g., pyelonephritis, urosepsis), signs and symptom onset  $\geq$ 96 hours before study entry, or a temperature  $\geq$ 101.4°F ( $\geq$ 38°C), flank pain, chills, or any other manifestations suggestive of upper UTI.
- 14. The participant has known anuria, oliguria, or significant impairment of renal function (creatinine clearance <60 mL/min or clinically significant elevated serum creatinine as determined by the investigator).
- 15. The participant presents with vaginal discharge at Baseline (e.g., suspected sexually transmitted disease).

## **Cardiac Exclusions**

- 16. The participant has congenital long QT syndrome or known prolongation of the corrected QT (QTc) interval.
- 17. The participant has uncompensated heart failure.
- 18. The participant has severe left ventricular hypertrophy.
- 19. The participant has a family history of QT prolongation or sudden death.
- 20. The participant has a recent history of vasovagal syncope or episodes of symptomatic bradycardia or brady arrhythmia within the last 12 months.
- 21. The participant is taking QT-prolonging drugs or drugs known to increase the risk of torsades de pointes (TdP) per the www.crediblemeds.org. "Known Risk of TdP" category at the time of her Baseline Visit, which cannot be safely discontinued from the Baseline Visit to the TOC Visit; or the participant is taking a strong cytochrome P450 enzyme 3A4 (CYP3A4) inhibitor.

## **Cardiac ECG Exclusions**

- 22. For any participant ≥12 to <18 years of age, the participant has an abnormal ECG reading at Baseline or during the study treatment.
- 23. The participant has a QTc >450 msec or a QTc >480 msec for participants with bundle-branch block.

### Note:

- The QTc is the QT interval corrected for heart rate according to either Bazett's formula (QTcB), or Fridericia's (QTcF) formula, and/or another method. It is either machine read or manually overread.
- The specific formula used to determine eligibility and discontinuation for an individual participant should be determined prior to initiation of the study. In other words, several different formulas cannot be used to calculate the QTc for an individual participant and then the lowest QTc value used to include or discontinue the participant from the trial.
- 24. The participant has a documented or recent history of uncorrected hypokalemia within the past 3 months.

## **Hepatic Exclusions**

- 25. The participant has a known alanine aminotransferase (ALT) value >2 × upper limit of normal (ULN).
- 26. The participant has a known bilirubin value  $>1.5 \times ULN$  (isolated bilirubin  $>1.5 \times ULN$  is acceptable if bilirubin is fractionated and direct bilirubin <35%).
- 27. The participant has cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice.

**Note**: Stable noncirrhotic chronic liver disease (including Gilbert's syndrome, asymptomatic gallstones, and chronic stable hepatitis B or C [e.g., presence of hepatitis B surface antigen or positive hepatitis C antibody test result]) is acceptable if the participant otherwise meets entry criteria.

28. The participant has a previous history of cholestatic jaundice/hepatic dysfunction associated with nitrofurantoin.

## **Prior Antibiotic/Antifungal Use Exclusion**

29. The participant has received treatment with other systemic antimicrobials or systemic antifungals within 1 week before study entry.

### **Concomitant Medication Use Exclusion**

30. The participant plans to use any of the prohibited medications or nondrug therapies from the Baseline Visit through the TOC Visit as detailed in Section 6.5.2.

## Prior/Concurrent Clinical Study Experience

- 31. The participant has been previously enrolled in this study or has previously been treated with gepotidacin.
- 32. The participant has participated in a clinical trial and has received an investigational product within 30 days or 5 half-lives, whichever is longer.

## 5.3. Lifestyle Considerations

Participants will be requested to abstain from sexual activity from the Baseline Visit through the TOC Visit to prevent possible re-infection.

## 5.3.1. Meals and Dietary Restrictions

Study treatment should be taken after food consumption (a meal or a snack) and with water (see Section 6.1).

## 5.4. Screen Failures

Screen failures are defined as participants who consent to participate in the clinical study but are not subsequently randomized. A minimal set of screen failure information is required to ensure transparent reporting of screen failure participants to meet the Consolidated Standards of Reporting Trials (CONSORT) publishing requirements and to respond to queries from regulatory authorities. Minimal information includes demography, screen failure details, eligibility criteria, any protocol deviations and any SAEs.

Participants who are screen failures are allowed to be rescreened for the same infection episode or a subsequent infection episode and participate in the study if they meet all of the inclusion and exclusion criteria.

TMF-13817737 212390

#### 6. STUDY TREATMENT

Study treatment is defined as any investigational treatment(s), marketed product(s), placebo, or medical device(s) intended to be administered to a study participant according to the study protocol.

### 6.1. **Study Treatments Administered**

All doses of study treatment should always be taken after food consumption and with water. Participants will receive oral study treatment (gepotidacin [2 tablets] + nitrofurantoin matching placebo [1 capsule] or nitrofurantoin [1 capsule] + gepotidacin matching placebo [2 tablets]) BID (approximately every 12 hours) for 5 days.

- The first oral dose will be administered at the study site during the Baseline Visit; participants will self-administer subsequent doses as outpatients thereafter.
- At the On-therapy Visit, whenever it is possible, the participant will have the pregnancy test performed at the study site. If the visit coincides with the 8th dose, the participant will take their next dose of study treatment at the study site after negative pregnancy test results are confirmed.
- Before the On-therapy Visit, if the requirement for the single pregnancy test to be done between dose 4 and dose 8 cannot be done at the study site due to availability of open clinic hours and the investigator considers the participant reliable to accurately perform the study-provided pregnancy test at home will be instructed to do so. If the pregnancy test is negative, those participants will be instructed to take their next dose of study treatment at home via text or by study site staff before going to the study site for their On-therapy Visit.

**Note:** The On-therapy Visit should be scheduled to support completion of the postdose ECG within the protocol-defined window. Also, in WOCBP, the high sensitivity pregnancy test must be performed and show negative results at the latest before Dose 8 of study treatment is taken.

| Study<br>Treatment<br>Name: | Gepotidacin | Placebo<br>(Matched to<br>Nitrofurantoin) | Nitrofurantoin | Placebo<br>(Matched to<br>Gepotidacin) |
|---|---|---|---|---|
| Туре: | Drug | Drug | Drug | Drug |
| Dose<br>Formulation: | Tablets containing gepotidacin and inactive formulation excipients | Over-encapsulated unit-dose nitrofurantoin placebo-to-match capsule | Over-encapsulated capsules containing nitrofurantoin (25 mg nitrofurantoin macrocrystals and 75 mg nitrofurantoin monohydrate) and inactive formulation excipients | Unit-dose<br>gepotidacin<br>placebo-to-match<br>tablet |
| Unit-Dose<br>Strengths/<br>Dosage Levels: | 2 x 750-mg tablets | Not applicable | 1 x 100-mg capsule | Not applicable |
| Route of Administration: | Oral | Oral | Oral | Oral |
| Dosing<br>Instructions: | Administer twice daily for 5 days: | Administer twice daily for 5 days: | Administer twice daily for 5 days: | Administer twice daily for 5 days: |
| | 1500 mg – 2 tablets | 1 capsule | 100 mg – 1 capsule | 2 tablets |
| | (3000 mg total daily dose) Each dose should be taken after food consumption and with water. | Each dose should be taken after food consumption and with water. | (200 mg total daily dose) Each dose should be taken after food consumption and with water. | Each dose should be taken after food consumption and with water. |
| Packaging and Labeling: | Gepotidacin tablets<br>will be provided in<br>bottles. Each bottle<br>will be labeled as<br>required per country<br>requirement. | Placebo-to-match nitrofurantoin capsules will be over-encapsulated and provided in bottles. Each bottle will be labeled as required per country requirement. | Nitrofurantoin capsules will be over-encapsulated and provided in bottles. Each bottle will be labeled as required per country requirement. | Placebo-to-match<br>gepotidacin tablets<br>will be provided in<br>bottles. Each bottle<br>will be labeled as<br>required per country<br>requirement. |
| Manufacturer: | Patheon Canada<br>(part of Thermo<br>Fisher Scientific) | Almac, LTD<br>(Over-encapsulation<br>by Almac, LTD) | Alvogen<br>(Over-encapsulation<br>by Almac, LTD) | Patheon Canada<br>(part of Thermo<br>Fisher Scientific) |

## 6.2. Preparation/Handling/Storage/Accountability

- 1. The investigator or designee must confirm appropriate temperature conditions have been maintained during transit for all study treatment received and any discrepancies are reported and resolved before use of the study treatment.
- 2. Only participants enrolled in the study may receive study treatment and only authorized site staff may supply or administer study treatment. All study treatments must be stored in a secure, environmentally controlled, and monitored (manual or automated) area in accordance with the labeled storage conditions with access limited to the investigator and authorized site staff.
- 3. The investigator, institution, or the head of the medical institution (where applicable) is responsible for study treatment accountability, reconciliation, and record maintenance (i.e., receipt, reconciliation, and final disposition records).
- 4. Further guidance and information for the final disposition of unused study treatment are provided in the SRM.

Under normal conditions of handling and administration, study treatment is not expected to pose significant safety risks to site staff.

A Material Safety Data Sheet or equivalent document describing occupational hazards and recommended handling precautions either will be provided to the investigator, where this is required by local laws, or is available upon request from GSK.

## 6.3. Measures to Minimize Bias: Randomization and Blinding

Participants will be stratified by age category (<18 years, ≥18 to 50 years, or >50 years) and acute cystitis recurrence (nonrecurrent infection or recurrent infection, defined as a confirmed infection [not including the current infection in the calculation] with at least 1 prior episode within the past 3 months, at least 2 prior episodes within the past 6 months, or at least 3 prior episodes within the past 12 months before study entry). Participants will be centrally randomized in a 1:1 ratio to either gepotidacin + matching nitrofurantoin placebo or nitrofurantoin + matching gepotidacin placebo. All participants will be centrally randomized using interactive response technology (IRT). Before the study is initiated, information and directions for the IRT will be provided to each study site.

Study treatment will be dispensed at the study visits summarized in Section 1.3.

Returned study treatment should not be re-dispensed to other participants.

This is a double-blind, double-dummy study. The study treatment taken during the study will be double-blind. Neither the participant nor study personnel (i.e., investigators, GSK, PPD [full service partner]) will know which study treatment a participant is receiving. In order to maintain study treatment blinding, participants will receive, in addition to their randomized active treatment (gepotidacin or nitrofurantoin), a matching placebo form of the active treatment to which they were not assigned. The matching placebos will look identical to the active form.

The IRT will be programmed with blind-breaking instructions. In case of an emergency, the investigator has the sole responsibility for determining if unblinding of a participant's treatment assignment is warranted. Participant safety must always be the first consideration in making such a determination. If the investigator decides that unblinding is warranted, the investigator should make every effort to contact GSK/PPD prior to unblinding a participant's treatment assignment unless this could delay emergency treatment of the participant. If a participant's treatment assignment is unblinded GSK/PPD must be notified within 24 hours after breaking the blind. The date and reason that the blind was broken must be recorded in the source documentation and electronic case report form (eCRF), as applicable.

A participant may continue in the study if that participant's treatment is unblinded provided that there are no safety concerns for the participant per the investigator's judgement.

The GSK SRT, which will monitor safety data instream, will remain blinded to participant treatment assignment throughout the study (see Appendix 3). A Microbiology Review Team will monitor blinded pathogen identification and susceptibility data instream as well as the number of participants eligible for the micro-ITT Population. Blinded monitoring of pathogens will be conducted, to determine whether end-of-study targets are likely to be achieved. Provision will be made for a limited degree of unblinding of a minority of participant sample data should this be viewed as appropriate for planning closure of trial enrollment. Procedures will be described in a separate microbiology sample monitoring plan, and no impact on trial integrity is expected.

The IDMC and Statistical Data Analysis Center (SDAC) will be unblinded for the IA (Section 9.5). The IDMC details will be described in a separate charter and analysis plan. The GSK and PPD study teams that are operating the study and conducting the final analysis will remain blinded.

GSK's Global Clinical Safety and Pharmacovigilance staff may unblind the treatment assignment for any participant with an SAE. If the SAE requires that an expedited regulatory report be sent to one or more regulatory agencies, a copy of the report, identifying the participant's treatment assignment, may be sent to investigators in accordance with local regulations and/or GSK policy.

## 6.4. Study Treatment Compliance

- When participants are dosed at the study site during the Baseline and On-therapy Visits, they will take their study treatment when directed by the investigator or designee, under medical supervision. The date and time of each dose administered at the study site will be recorded in the source documents. The dose of study treatment and study participant identification will be confirmed at the time of dosing by a member of the study site staff other than the person administering the study treatment.
- When participants self-administer study treatment as outpatients, compliance with gepotidacin, nitrofurantoin placebo, nitrofurantoin, and gepotidacin placebo will be assessed through querying the participant during the study site visits and documented in the source documents and eCRF. A record of the number of gepotidacin and

gepotidacin placebo tablets and nitrofurantoin and nitrofurantoin placebo capsules dispensed to and returned by each participant must be maintained and reconciled with study treatment and compliance records. Study treatment start and stop dates, including dates for study treatment delays, will also be recorded in the eCRF.

## 6.5. Concomitant Therapy

Any medication or vaccine (including over-the-counter or prescription medicines, vitamins, and/or herbal supplements) that the participant is receiving within 30 days prior to the Baseline Visit or receives during the study must be recorded in the eCRF. In addition, any antibiotic use within 6 months prior to the Baseline Visit or during the study must be recorded in the eCRF. The concomitant therapy name must be recorded in the eCRF along with the following:

- Reason for use
- Dates of administration including start and end dates
- Dosage information including dose and frequency

The medical monitor should be contacted if there are any questions regarding concomitant or prior therapy.

## 6.5.1. Permitted Medications and Nondrug Therapies

The use of H<sub>1</sub> antihistaminics not associated with QT prolongation is allowed (e.g., loratadine, cetirizine, ebastine, and fexofenadine). The use of topical, nonsystemic antibacterials (e.g., topical clindamycin, neomycin, or polymyxin) and topical, nonsystemic antifungals (e.g., topical clotrimazole, tolnaftate, or ketoconazole) is allowed throughout the study. Please also refer to Appendix 9.

Acetaminophen or paracetamol use is permitted throughout the study as it does not mask symptoms of the disease under study. A list of permitted medications commonly used for nausea, vomiting, pain, and diarrhea per investigator discretion is provided in Appendix 9. As described in Appendix 9, low-dose acetylsalicylic acid (≤100 mg/day) is permitted for the prevention of cardiovascular (CV) disease events.

A further detailed list of medications will be provided in the SRM.

## 6.5.2. Prohibited Medications and Nondrug Therapies

At the time of enrollment and/or during the study from the Baseline Visit through the TOC Visit, the participant is prohibited from use of the following medications and nondrug therapies:

- An investigational product within 30 days or 5 half-lives, whichever is longer, of the Baseline Visit.
- Treatment with other systemic antimicrobials (e.g., oral ciprofloxacin, amoxicillin/clavulanate, cephalexin, or doxycycline) or systemic antifungals (e.g., oral fluconazole, itraconazole, or terbinafine) within 1 week before study entry.

Treatment with systemic fluconazole or other systemic antifungals per local standard of care is only allowed after all TOC Visit procedures have been completed.

- Immunosuppressive therapy, including corticosteroid therapy (>40 mg/day prednisolone or equivalent for >1 week, ≥20 mg/day prednisolone or equivalent for >2 weeks, or prednisolone or equivalent ≥10 mg/day for >6 weeks).
- QT-prolonging drugs or drugs with known TdP risk, per the www.crediblemeds.org "Known Risk of TdP" category, at the time of their Baseline Visit, which cannot be safely discontinued from the Baseline Visit to the TOC Visit. Details regarding website access are provided in the SRM; additional guidance is provided in Appendix 9. Of note, ondansetron is not allowed from the Baseline Visit to the TOC Visit due to its known TdP risk. Alternative antiemetics that are permitted per investigator discretion are listed in Appendix 9.

**Note**: Crediblemeds.org categorizes drugs into 4 categories. The only category for exclusion in this study is the "Known Risk of TdP" category; participants taking drugs that meet criteria of other categories are NOT excluded from participation.

- Strong CYP3A4 inhibitors (a list of strong CYP3A4 inhibitors is provided in the SRM).
- St John's wort or other strong CYP3A4 inducers are not permitted from 14 days before study entry through the TOC Visit (a list is provided in the SRM).
- Prescription, nonprescription, or supplements that may impact UTI clinical or microbiological efficacy outcomes including, but not limited to, *Uva ursi*,
   D-mannose, cranberry tablets, phenazopyridine, nonsteroidal anti-inflammatory drugs including ibuprofen and cyclooxygenase-2 inhibitors, and uricosuric drugs (e.g., probenecid and sulfinpyrazone). As described in Appendix 9, acetylsalicylic acid (doses >100 mg/day) is not permitted.

In addition, antacid preparations containing magnesium trisilicate are prohibited from the start of study treatment at the Baseline Visit throughout the completion of the dosing period (i.e., until all 10 doses of study treatment have been received).

Due to the gepotidacin's property of acetylcholinesterase inhibition, the concomitant use of succinylcholine or other nondepolarizing paralytic agents is also prohibited. Caution should be used in participants who have a condition requiring medication that may exacerbate the inhibition of acetylcholinesterase, or neuromuscular blocking agents.

## 6.6. Dose Modification

The study design does not allow for dose modifications.

## 6.7. Treatment after the End of the Study

Participants will not receive any additional treatment from GSK after they discontinue or complete the study (i.e., after the Follow-up Visit). Participants experiencing signs and symptoms suggestive of infection recurrence or relapse at the Follow-up Visit will be assessed and treated per the investigator's judgement.

# 7. DISCONTINUATION OF STUDY TREATMENT AND PARTICIPANT DISCONTINUATION/WITHDRAWAL

## 7.1. Discontinuation of Study Treatment

In rare instances, it may be necessary for a participant to permanently discontinue (definitive discontinuation) study treatment. If study treatment is definitively discontinued, the participant will remain in the study to be evaluated for safety and efficacy. See the SoA (Section 1.3) for data to be collected at the time of discontinuation of study treatment and follow-up and for any further evaluations that need to be completed.

Participants may voluntarily discontinue study treatment at any time. The investigator may also, at his or her discretion, discontinue the participant from study treatment at any time and initiate appropriate alternative therapy.

Reasons for study treatment discontinuation may include the following:

- Adverse event
- Protocol deviation
- Termination of the study by GSK
- Investigator discretion
- Lack of efficacy

**Note**: Pathogen identification or in vitro resistance of recovered uropathogens is not a reason for study treatment discontinuation.

The reason for study treatment discontinuation will be recorded in the eCRF. Participants who discontinue study treatment for the reasons above will not be considered withdrawn from the study and should attend all subsequent study visits (see Section 1.3).

## 7.1.1. Liver Chemistry Stopping Criteria

Liver chemistry stopping, and increased monitoring criteria have been designed to assure participant safety and evaluate liver event etiology.

Discontinuation of study treatment for abnormal liver tests is required when:

- a participant meets one of the conditions outlined in Algorithm A or Algorithm B.
- when in the presence of abnormal liver chemistries not meeting protocol-specified stopping rules, the investigator believes study treatment discontinuation is in the best interest of the participant.

# Algorithm A: Phase III Liver Chemistry Stopping and Increased Monitoring Algorithm



Abbreviations: ALT = alanine transaminase; INR = international normalized ratio; SAE = serious adverse event; ULN = upper limit of normal.

Refer to Appendix 10 for required Liver Safety Actions and Follow-up Assessments.

Algorithm B: Phase III Liver Chemistry Increased Monitoring Algorithm with Continued Therapy for ALT  $\geq$ 3 × ULN but <8 × ULN



Abbreviations: ALT = alanine transaminase; bili = bilirubin; INR = international normalized ratio; SAE = serious adverse event; ULN = upper limit of normal.

Refer to Appendix 10 for required Liver Safety Actions and Follow-up Assessments.

## 7.1.2. QTc Stopping Criteria

A participant who meets the bulleted criteria based on the average of triplicate ECG readings will be withdrawn from study treatment:

- QTc >500 msec OR <u>Uncorrected</u> QT >600 msec
- Change from baseline of QTc >60 msec

For patients with underlying bundle branch block, follow the discontinuation criteria listed below:

| Baseline QTc with Bundle<br>Branch-Block | Discontinuation QTc with<br>Bundle-Branch Block |
|---|---|
| <450 msec | >500 msec |
| 450 to 480 msec | ≥530 msec |

- The *same* QT correction formula *must* be used for *each individual participant* to determine eligibility for and discontinuation from the study. This formula may not be changed or substituted once the participant has been enrolled. (Note: Ideally, all ECGs for a participant should be performed with the same ECG machine.)
  - For example, if a participant is eligible for the protocol based on QTcB, then QTcB must be used for discontinuation of this individual participant as well.
  - Once the QT correction formula has been chosen for a participant's eligibility, the *same formula* must continue to be used for that participant *for all QTc data being collected for data analysis*. Safety ECGs and other nonprotocol-specified ECGs are an exception.
- The QTc should be based on the average of triplicate ECG readings obtained over a brief (e.g., 5- to 10-minute) recording period.

## 7.1.3. Rechallenge

## 7.1.3.1. Study Treatment Restart or Rechallenge After Liver Stopping Criteria Met

Study treatment restart or rechallenge after liver chemistry stopping criteria are met by any participant in this study is not allowed.

### 7.1.4. Gastrointestinal Evaluation Criteria

If a participant meets the criteria in Appendix 1, *Clostridium difficile* toxin testing should be conducted and the specific eCRF page completed. *C. difficile* infection or colitis is considered an AE of special interest (Section 8.3.7).

## 7.2. Participant Discontinuation/Withdrawal from the Study

- A participant may withdraw from the study at any time at her own request or may be withdrawn at any time at the discretion of the investigator for safety, behavioral, compliance, or administrative reasons.
- Reasons for study withdrawal include:
  - Participant lost to follow-up
  - Participant withdrew consent
  - Termination of the study by GSK
  - Investigator discretion
- If the participant withdraws consent for disclosure of future information, the sponsor may retain and continue to use any data collected before such a withdrawal of consent.
- If a participant withdraws from the study, she may request destruction of any samples taken and not tested, and the investigator must document this in the site study records.

• At the time of discontinuing from the study, if possible, an early withdrawal visit should be conducted, as shown in the SoA (Section 1.3). See the SoA for data to be collected at the time of study discontinuation and follow-up and for any further evaluations that need to be completed.

The reason for participant withdrawal will be recorded in the eCRF. Participants who are withdrawn from the study should return to the study site and have the microbiological and clinical outcomes assessed at the time of withdrawal (see the SoA in Section 1.3), if data permit, and return all unused study treatment. Data from these participants will be considered evaluable up to the point at which they are withdrawn, using the same criteria for evaluability as for participants who complete the study.

## 7.3. Lost to Follow-Up

A participant will be considered lost to follow-up if she repeatedly fails to return for scheduled visits and is unable to be contacted by the study site.

The following actions must be taken if a participant fails to return to the study site for a required study visit:

- The study site must attempt to contact the participant and reschedule the missed visit as soon as possible and counsel the participant on the importance of maintaining the assigned visit schedule and ascertain whether or not the participant wishes to and/or should continue in the study.
- Before a participant is deemed lost to follow-up, the investigator or designee must make every effort to regain contact with the participant (where possible, 3 telephone calls and, if necessary, a certified letter to the participant's last known mailing address or local equivalent methods). These contact attempts should be documented in the participant's medical record.
- Should the participant continue to be unreachable, she will be considered to have withdrawn from the study with a primary reason of lost to follow-up.

Discontinuation of specific sites or of the study as a whole are handled as part of Appendix 3.

## 8. STUDY ASSESSMENTS AND PROCEDURES

- Study procedures and their timing are summarized in the SoA (Section 1.3).
- Protocol waivers or exemptions are not allowed.
- Immediate safety concerns should be discussed with the sponsor immediately upon occurrence or awareness to determine if the participant should continue or discontinue study treatment.
- Adherence to the study design requirements, including those specified in the SoA, is essential and required for study conduct.
- All baseline screening evaluations must be completed and reviewed to confirm that potential participants meet all eligibility criteria. The investigator will maintain a

screening log to record details of all participants screened and to confirm eligibility or record reasons for screening failure, as applicable.

212390

- Procedures conducted as part of the participant's routine clinical management (e.g., blood count) and obtained before signing of ICF may be utilized for screening or baseline purposes provided the procedure met the protocol-specified criteria and was performed within the time frame defined in the SoA.
- Prescreening activities may be conducted, including a prescreening informed consent
  and urine testing, as further detailed in the SRM. The required baseline urine
  specimen may be collected as part of an optional prescreening process, if not already
  part of standard of care, and is further detailed in the SRM. This specimen can be
  used for the required baseline procedures of the diagnosis of presumptive acute
  cystitis and pregnancy testing.
- The maximum amount of blood collected from each participant over the duration of the study, including any extra assessments that may be required, will not exceed 200 mL.
- Repeat or unscheduled samples may be taken for safety reasons or for technical issues with the samples.
- Participants may return to the study site at any time due to AEs or if they are
  experiencing new or continuing signs and symptoms of acute cystitis. Participants
  will be assessed and treated per the investigator's judgement. If a participant is
  switched to a different antibiotic before or during the TOC Visit, all TOC procedures
  should be completed before the other antibiotic is started.
- Each treatment day will be assessed over 24 hours starting with the first dose of study treatment, as further detailed in the SRM.

The study will comprise the following 4 planned study visits:

Note: For all study visits, to minimize the amount of time that participants spend at the clinic, eConsent may be utilized and remote collection of study-related data may be obtained as described in the SRM. Thus, some visit data may be collected through a combination of telemedicine and on-site visits. Collection of information via telemedicine will be performed only where local regulations permit.

- Baseline (Day 1) Visit: The Baseline Visit will be performed before dosing on Day 1. Assessments will be performed as shown in in the SoA (Section 1.3), including the following:
  - Pretreatment baseline specimens for microbiological testing will be collected, as described in Section 8.1.1. Clinical signs and symptoms of acute cystitis will be recorded, as described in Section 8.1.3.1 and Appendix 6.
  - Following completion of all pretreatment assessments, eligible participants will be randomly assigned to a study treatment, as described in Section 6.3.
  - The first dose of randomly assigned oral study treatment will be administered at the study site. After dose administration, Day 1 posttreatment assessments will be performed, as shown in Section 1.3. Any AEs or clinically significant

changes should be followed accordingly. Subsequent to administration of the first dose at the study site, participants will self-administer doses as outpatients thereafter, beginning with the second dose. (Note: Each dose should be taken after food consumption and with water.)

- The On-therapy, TOC, and Follow-up Visits should be scheduled before the
  participant leaves the study site on Day 1 (as per the Schedule of Activities
  Table in Section 1.3); the planned return day/time should be at the convenience
  of the participant and also the availability of the study site staff.
- On-therapy (Day 2 to 4) Visit: Participants will be instructed to return to the study site 1 to 3 days following study treatment administration at Baseline in order to complete the On-therapy Visit. Assessments will be performed as shown in the SoA (Section 1.3), including the following:
  - The On-therapy Visit will be preceded by a documented reminder contact from the study site to the participant 24 ± 4 hours before the scheduled appointment time per the method (e.g., text message, telephone call, e-mail) confirmed with the study site staff prior to departing the study site on Day 1.
  - At the On-therapy Visit, whenever it is possible, the participant will have the
    pregnancy test performed at the study site. If the visit coincides with the 8<sup>th</sup>
    dose, the participant will take their next dose of study treatment at the study site
    after negative pregnancy test results are confirmed.
  - Before the On-therapy Visit, if the requirement for the single pregnancy test to
    be done between dose 4 and dose 8 cannot be done at the study site due to
    availability of open clinic hours and the investigator considers the participant
    reliable to accurately perform the study-provided pregnancy test at home will be
    instructed to do so. If the pregnancy test is negative, those participants will be
    instructed to take their next dose of study treatment at home via text or by study
    site staff before going to the study site for their On-therapy Visit.

Note: The On-therapy Visit should be scheduled to support completion of the postdose ECG within the protocol-defined window. Also, in WOCBP, the high sensitivity pregnancy test must be performed and show negative results at the latest *before* Dose 8 of study treatment is taken.

- Specimens for microbiological testing will be collected, as described in Section 8.1. Clinical signs and symptoms of acute cystitis will be recorded, as described in Section 8.1.3.1 and Appendix 6.
- Pregnancy testing, as required, after Dose 4 and before Dose 8. Refer to Appendix 8 for details.
- Participants will remain at the study site until approximately 2 to 4 hours postdose. A triplicate ECG will be performed at approximately 2 hours postdose, as detailed in Section 1.3.
- TOC (Day 10 to 13) Visit: Participants will be instructed to return to the study site
   5 to 8 days after completion of study treatment in order to complete the TOC Visit.

Assessments will be performed as shown in the SoA (Section 1.3), including the following:

212390

- The TOC Visit will be preceded by a documented reminder contact from the study site to the participant 24 ± 4 hours before the scheduled appointment time per the method (e.g., text message, telephone call, e-mail) confirmed with the study site staff prior to departing the study site on Day 1.
- Specimens for microbiological testing will be collected, as described in Section 8.1. Clinical signs and symptoms of acute cystitis will be recorded, as described in Section 8.1.3.1 and Appendix 6.
- Follow-up (Day 28±3) Visit. Participants will be instructed to return to the study site 28 (±3) days postrandomization in order to complete the Follow-up Visit.
   Assessments will be performed as shown in Section 1.3, including the following:
  - The Follow-up Visit will be preceded by a documented reminder contact from the study site to the participant 24 ±4 hours before the scheduled appointment time per the method (e.g., text message, telephone call, e-mail) confirmed with the study site staff prior to departing the study site on Day 1.
  - Specimens for microbiological testing will be collected, as described in Section 8.1. Clinical signs and symptoms of acute cystitis will be recorded, as described in Section 8.1.3.1 and Appendix 6.
  - Participants experiencing signs and symptoms suggestive of infection recurrence or relapse will be assessed and treated per the investigator's judgement.

## 8.1. Efficacy Assessments

## 8.1.1. Therapeutic Response Evaluation

Therapeutic response (success/failure) is a measure of the overall efficacy response. A therapeutic success refers to participants who have been deemed both a "microbiological success" (see Section 8.1.2.1) and a "clinical success" (see Section 8.1.3.1). All other combinations (other than clinical success + microbiological success) will be deemed failures for therapeutic response.

Therapeutic response will be determined by statistical programming for the TOC and Follow-up Visits.

Therapeutic response at TOC is the primary efficacy endpoint.

## 8.1.2. Bacteriology Samples

At the Baseline Visit, a pretreatment, clean-catch midstream urine sample must be obtained from all randomized participants for Gram stain, quantitative bacteriological culture, and in vitro antimicrobial susceptibility testing at a designated central

laboratory(ies). For inclusion in the micro-ITT Population, a baseline qualifying bacterial uropathogen is required as defined in Appendix 4; for inclusion in the micro-ITT NTF-S Population, the baseline qualifying uropathogen must also be susceptible to nitrofurantoin. At the On-therapy, TOC, and Follow-up Visits, a clean-catch midstream urine sample will be obtained and sent to a designated central laboratory(ies) for Gram stain, quantitative bacteriological culture, and in vitro antimicrobial susceptibility testing. Identification and susceptibility testing of isolates recovered from urine specimens at all visits will also be conducted at a designated central laboratory(ies). Additional tests, as needed, to further characterize recovered isolates will also be performed by a designated central laboratory(ies). Instructions for sample collection, processing, and shipment are provided in the SRM and the laboratory manual. The study site should follow the Microbiology Procedures section of the laboratory manual to minimize potential contamination of the specimens.

## 8.1.2.1. Microbiological Outcome and Response

Only those participants who have a qualifying bacterial uropathogen (defined in Appendix 4) identified at Baseline will be evaluated for microbiological outcome and response by baseline qualifying uropathogen for the primary efficacy endpoint. The microbiological outcome and response to study treatment will be determined programatically for each participant/uropathogen prior to breaking of the study blind.

The microbiological outcome by baseline qualifying uropathogen is determined by comparing the baseline culture results to the culture results at each subsequent visit (see Table 2, Table 3, and Table 4 for baseline qualifying uropathogen outcomes). The corresponding microbiological response (success or failure) "by uropathogen" is then assigned, as shown in Table 3 and Table 4. Participant-level microbiological response is a measure of the combined "by uropathogen" response(s). Participant-level microbiological success refers to participants who have been deemed a "microbiological success" for all of their "by uropathogen" microbiological responses. All other combinations (other than all "microbiological successes") are deemed failures for participant-level microbiological response. The participant-level microbiological outcome and response definitions are provided in Table 5.

Microbiological outcome criteria for new qualifying uropathogens (i.e., uropathogens not identified at Baseline) are defined by visit in

Table 6, Table 7, and Table 8.

Table 2 Microbiological Outcome by Baseline Qualifying Uropathogen at the On-Therapy Visit

| Defining Criteria | Outcome |
|------------------------------------------------|-----------------------------|
| A quantitative urine culture taken at the | Microbiological eradication |
| On-therapy Visit shows that the qualifying | |
| bacterial uropathogen recovered at Baseline is | |
| reduced to <103 CFU/mL, without the | |
| participant receiving other systemic | |
| antimicrobials before the On-therapy Visit | |
| A quantitative urine culture taken at the | Microbiological persistence |
| On-therapy Visit shows that the qualifying | |
| bacterial uropathogen recovered at Baseline | |
| grows ≥10³ CFU/mL, without the participant | |
| receiving other systemic antimicrobials before | |
| the On-therapy Visit | |
| 1) The On-therapy urine culture result is | Unable to determine |
| missing, or | |
| 2) The participant received other systemic | |
| antimicrobials before the On-therapy Visit | |

CFU=colony-forming units.

Table 3 Microbiological Outcome and Response by Baseline Qualifying Uropathogen at the Test-of-Cure Visit

| Defining Criteria | Outcome | Response |
|---|---|---|
| Participants considered microbiological failures microbiological failures at the Follow-up Visit. | at the TOC Visit will also | be considered |
| A quantitative urine culture taken at the TOC | Microbiological | Microbiological |
| Visit shows reduction of the qualifying | eradication | success |
| bacterial uropathogen recovered at Baseline | | |
| to <10 <sup>3</sup> CFU/mL, without the participant | | |
| receiving other systemic antimicrobials | | |
| before the TOC Visit | Migrabialagical | Microbiological failure |
| A quantitative urine culture taken at the TOC Visit shows that the qualifying bacterial | Microbiological persistence | Microbiological failure |
| uropathogen recovered at Baseline, and | persistence | |
| which was also shown to persist or unable to | | |
| determine at the On-therapy Visit, grows | | |
| ≥10 <sup>3</sup> CFU/mL, without the participant | | |
| receiving other systemic antimicrobials | | |
| before the TOC Visit | | |
| A quantitative urine culture taken at the TOC | Microbiological | Microbiological failure |
| Visit shows that the qualifying bacterial | recurrence | |
| uropathogen recovered at Baseline, and | | |
| which was also shown to be eradicated at | | |
| the On-therapy Visit, grows ≥10³ CFU/mL, | | |
| without the participant receiving other systemic antimicrobials before the TOC Visit | | |
| The TOC urine culture result is missing, | Unable to determine | Microbiological failure |
| or | Chable to determine | Wildiobiological fallate |
| 2) The participant received other systemic | | |
| antimicrobials before the TOC Visit | | |

CFU=colony-forming units; TOC=Test-of-Cure.

Table 4 Microbiological Outcome and Response by Baseline Qualifying Uropathogen at the Follow-Up Visit

| Participants considered microbiological failures at the TOC Visit will also be considered microbiological failures at the Follow-up Visit. A quantitative urine culture taken at the Follow-up Visit shows reduction of the qualifying bacterial uropathogen recovered at Baseline to <10³ CFU/mL, following microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows that the qualifying bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, following microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows that the qualifying bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the TOC Visit, without the participant receiving other systemic antimicrobiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobiological eradication at the TOC Visit, without the participant receiving other systemic and so did not achieve an outcome of microbiological eradication at the TOC Visit, without the participant receiving other systemic and the TOC Visit, without the participant receiving other systemic and the TOC Visit, without the participant receiving other systemic and the TOC Visit, without the participant receiving other systemic and the TOC Visit, without the participant receiving other systemic and the TOC Visit, without the partici | Defining Criteria | Outcome | Response |
|---|---|---|---|
| A quantitative urine culture taken at the Follow-up Visit shows reduction of the qualifying bacterial uropathogen recovered at Baseline to <10³ CFU/mL, following microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows that the qualifying bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, following microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows that the qualifying bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit Delayed microbiological failure bacterial uropathogen recovered at Baseline to <10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the | | the TOC Visit will also be | |
| Follow-up Visit shows reduction of the qualifying bacterial uropathogen recovered at Baseline to <10³ CFU/mL, following microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the participant receiving other systemic anoutcome of microbiological eradication at the TOC Visit, without the participant receiving other systemic anoutcome of microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit shows that the qualifying bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, and also did not achieve an outcome of microbiological eradication of the qualifying bacterial uropathogen recovered at Baseline to <10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the | microbiological failures at the Follow-up Visit. | | |
| bacterial uropathogen recovered at Baseline to <10³ CFU/mL, following microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows that the qualifying bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, following microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows that the qualifying bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows reduction of the qualifying bacterial uropathogen recovered at Baseline to <10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the | A quantitative urine culture taken at the | Sustained | Microbiological |
| <10³ CFU/mL, following microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows that the qualifying bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, following microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows that the qualifying bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows reduction of the qualifying bacterial uropathogen recovered at Baseline to <10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the | Follow-up Visit shows reduction of the qualifying | microbiological | success |
| eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows that the qualifying bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, following microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows that the qualifying bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows reduction of the qualifying bacterial uropathogen recovered at Baseline to <10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the | bacterial uropathogen recovered at Baseline to | eradication | |
| participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows that the qualifying bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, following microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows that the qualifying bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows reduction of the qualifying bacterial uropathogen recovered at Baseline to <10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the | | | |
| antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows that the qualifying bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, following microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows that the qualifying bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows reduction of the qualifying bacterial uropathogen recovered at Baseline to <10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the outcome of microbiological eradication at the outcome of microbiological eradication at the | · | | |
| A quantitative urine culture taken at the Follow-up Visit shows that the qualifying bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, following microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows that the qualifying bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows reduction of the qualifying bacterial uropathogen recovered at Baseline to <10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the | 1 ' ' | | |
| Follow-up Visit shows that the qualifying bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, following microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows that the qualifying bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows reduction of the qualifying bacterial uropathogen recovered at Baseline to <10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the | • | | |
| bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, following microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows that the qualifying bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows reduction of the qualifying bacterial uropathogen recovered at Baseline to <10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the | · | Microbiological | _ |
| grows ≥10³ CFU/mL, following microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows that the qualifying bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows reduction of the qualifying bacterial uropathogen recovered at Baseline to <10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the | | recurrence | failure |
| eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows that the qualifying bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows reduction of the qualifying bacterial uropathogen recovered at Baseline to <10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the | . • | | |
| participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows that the qualifying bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows reduction of the qualifying bacterial uropathogen recovered at Baseline to <10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the | , | | |
| A quantitative urine culture taken at the Follow-up Visit shows that the qualifying bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows reduction of the qualifying bacterial uropathogen recovered at Baseline to <10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the | , | | |
| A quantitative urine culture taken at the Follow-up Visit shows that the qualifying bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows reduction of the qualifying bacterial uropathogen recovered at Baseline to <10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the | 1 ' ' | | |
| Follow-up Visit shows that the qualifying bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows reduction of the qualifying bacterial uropathogen recovered at Baseline to <10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the | • | | |
| bacterial uropathogen recovered at Baseline grows ≥10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows reduction of the qualifying bacterial uropathogen recovered at Baseline to <10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the | | _ | _ |
| grows ≥10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows reduction of the qualifying bacterial uropathogen recovered at Baseline to <10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the | | persistence | failure |
| an outcome of microbiological eradication at the TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows reduction of the qualifying bacterial uropathogen recovered at Baseline to <10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the | . • | | |
| TOC Visit, without the participant receiving other systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows reduction of the qualifying bacterial uropathogen recovered at Baseline to <10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the | , | | |
| systemic antimicrobials before the Follow-up Visit A quantitative urine culture taken at the Follow-up Visit shows reduction of the qualifying bacterial uropathogen recovered at Baseline to <10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the Microbiological microbiological eradication at the | _ | | |
| Visit A quantitative urine culture taken at the Follow-up Visit shows reduction of the qualifying bacterial uropathogen recovered at Baseline to <10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the Microbiological failure eradication | , , | | |
| A quantitative urine culture taken at the Follow-up Visit shows reduction of the qualifying bacterial uropathogen recovered at Baseline to <10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the Delayed microbiological failure eradication | 1 7 | | |
| Follow-up Visit shows reduction of the qualifying bacterial uropathogen recovered at Baseline to <10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the | | D.I. I | NA: 1:1 : 1 |
| bacterial uropathogen recovered at Baseline to <a href="https://www.ncbi.nlm">to</a> eradication <a href="https://www.ncbi.nlm">to</a> eradication outcome of microbiological eradication at the | • | | |
| <10³ CFU/mL, and also did not achieve an outcome of microbiological eradication at the | | | lallure |
| outcome of microbiological eradication at the | , , | eradication | |
| | l · | | |
| systemic antimicrobials before the Follow-up | | | |
| Visit | 1 - 7 | | |
| The Follow-up urine culture result is Unable to determine | | Unable to determine | Microbiological |
| missing, or failure | , , | Shabio to dotominio | |
| 2) The participant received other systemic | ) · | | ianaio |
| antimicrobials before the Follow-up Visit | 1 | | |

CFU=colony-forming units; TOC=Test-of-Cure.

212390

Table 5 Participant-Level Microbiological Outcome and Response Definitions per Study Visit

| Defining Criteria at the On-Therapy Visit | Outcome | Response |
|---|---|---|
| All qualifying baseline uropathogens have a microbiological | Microbiological | NA |
| outcome of eradication at On-therapy | eradication | |
| At least one qualifying baseline uropathogen has an | Microbiological | NA |
| outcome of persistence at On-therapy | persistence | |
| All qualifying baseline uropathogen outcomes are unable to | Unable to determine | NA |
| determine at On-therapy | | |
| Defining Criteria at the TOC Visit | Outcome | Response |
| All qualifying baseline uropathogens have a microbiological | Microbiological | Microbiological |
| outcome of eradication at TOC | eradication | success |
| At least one qualifying baseline uropathogen has an | Microbiological | Microbiological |
| outcome of persistence at TOC | persistence | failure |
| At least one qualifying baseline uropathogen has an | Microbiological | Microbiological |
| outcome of recurrence and none have an outcome of | recurrence | failure |
| persistence at TOC | | |
| All qualifying baseline uropathogen outcomes are unable to | Unable to determine | Microbiological |
| determine at TOC | | failure |
| | 1 | 1 |
| Defining Criteria at the Follow-up Visit | Outcome | Response |
| All qualifying baseline uropathogens have a microbiological | Sustained | Microbiological |
| outcome of sustained eradication at Follow-up | microbiological | success |
| | eradication | |
| At least one qualifying baseline uropathogen has an | Microbiological | Microbiological |
| outcome of recurrence and none have an outcome of | recurrence | failure |
| persistence at Follow-up | | |
| At least one qualifying baseline uropathogen has an | Microbiological | Microbiological |
| outcome of persistence at Follow-up | persistence | failure |
| At least one qualifying baseline uropathogen has an | Delayed | Microbiological |
| outcome of delayed eradication and none have an outcome | microbiological | failure |
| of persistence or recurrence at Follow-up | eradication | |
| All qualifying baseline uropathogen outcomes are unable to | Unable to determine | Microbiological |
| determine at Follow-up | | failure |

NA=Not applicable; TOC=Test-of-Cure.

Table 6 Microbiological Outcome by New Qualifying Uropathogen at the On-Therapy Visit

| Defining Criteria | Outcome |
|----------------------------------------------|-----------------|
| A new qualifying bacterial uropathogen, not | New uropathogen |
| identified at Baseline, is documented by | |
| quantitative urine culture at the On-therapy | |
| Visit | |

212390

Table 7 Microbiological Outcome by New Qualifying Uropathogen at the **Test-of-Cure Visit** 

| Defining Criteria | Outcome |
|---|---|
| A new qualifying bacterial uropathogen, not identified at Baseline, is documented by quantitative urine culture at the Test-of-Cure Visit in a participant who did not achieve a | New infection |
| clinical outcome of clinical resolution at the Test-of-Cure Visit | |
| A new qualifying bacterial uropathogen, not identified at Baseline, is documented by quantitative urine culture at the Test-of-Cure Visit in a participant who did achieve a clinical outcome of clinical resolution at the Test-of-Cure Visit | Colonization |

Table 8 Microbiological Outcome by New Qualifying Uropathogen at the **Follow-up Visit** 

| Defining Criteria | Outcome |
|---------------------------------------------------|---------------|
| A new qualifying bacterial uropathogen, not | New infection |
| identified at Baseline, is documented by | |
| quantitative urine culture at the Follow-up Visit | |
| in a participant who did not achieve a clinical | |
| resolution at the Follow-up Visit | |
| A new qualifying bacterial uropathogen, not | Colonization |
| identified at Baseline, is documented by | |
| quantitative urine culture at the Follow-up Visit | |
| in a participant who did achieve a clinical | |
| resolution at the Follow-up Visit | |

#### 8.1.3. Clinical Evaluation

### 8.1.3.1. Clinical Signs and Symptom Scores, Clinical Outcomes, and Clinical Response

Clinical signs and symptoms of acute cystitis will be recorded based on participant interview per the SoA (Section 1.3) using the scoring system and instructions in Appendix 6. At Baseline, the participant must present with at least 2 signs and symptoms and have a total cumulative symptom score ≥2. At TOC, success is defined as normal presentation of signs and symptoms with a total cumulative symptom score of zero and no new signs and symptoms of the infection under study.

A study physician or otherwise appropriately medically trained staff will determine the individual clinical signs and symptoms scores for acute cystitis (Appendix 6) at the On-therapy, TOC, and Follow-up Visits. The same scorer will be used at all assessment time points for each participant, on all occasions, whenever possible. The score will be used to programmatically determine the clinical outcome at the On-therapy Visit (Table 9) and the clinical outcome and response (success or failure) at the TOC Visit (Table 10) and the Follow-up Visit (Table 11).

Table 9 Clinical Outcome at the On-Therapy Visit

| Defining Criteria | Outcome <sup>a</sup> |
|---|---|
| Resolution of signs and symptoms of acute cystitis present at Baseline (and no new signs and symptoms), without the participant receiving other systemic antimicrobials before the On-therapy Visit | Clinical resolution |
| Improvement in total symptom scores from Baseline, but not complete resolution, without the participant receiving other systemic antimicrobials before the On-therapy Visit | Clinical improvement |
| Worsening or no change in total symptom scores from Baseline or the participant received other systemic antimicrobials for the current infection prior to or on the date of the On-therapy Visit | Clinical worsening |
| The Baseline score is missing, or The On-therapy assessment is missing, or The participant received other systemic antimicrobials not for the current infection prior to the assessment (unless clinical worsening outcome criteria were met) | Unable to determine |

a. A study physician or otherwise appropriately medically trained staff will determine the individual clinical signs and symptoms scores for acute cystitis (Appendix 6), which will then be used to programmatically determine the clinical outcome. The same scorer will be used at all assessment time points for each participant, on all occasions, whenever possible.

Table 10 Clinical Outcome and Response at the Test-of-Cure Visit

| Defining Criteria | Outcome <sup>a</sup> | Response |
|---|---|---|
| Resolution of signs and symptoms of acute cystitis present at Baseline (and no new signs or symptoms), without the participant receiving other systemic antimicrobials before the TOC Visit | Clinical resolution | Clinical success |
| Improvement in total symptom scores from Baseline, but not complete resolution, without the participant receiving other systemic antimicrobials before the TOC Visit | Clinical improvement | Clinical failure |
| Worsening or no change in total symptom scores from Baseline or the participant received other systemic antimicrobials for the current infection before or on the date of the TOC Visit | Clinical worsening | Clinical failure |
| The Baseline score is missing, or The TOC assessment is missing, or The participant received other systemic antimicrobials not for the current infection prior to the assessment (unless clinical worsening criteria were met) TOC Test of Cure | Unable to determine | Clinical failure |

TOC = Test-of-Cure

a. A study physician or otherwise appropriately medically trained staff will determine the individual clinical signs and symptoms scores for acute cystitis (Appendix 6), which will then be used to programmatically determine the clinical outcome. The same scorer will be used at all assessment time points for each participant, on all occasions, whenever possible.

Table 11 Clinical Outcome and Response at the Follow-up Visit

| Defining Criteria | Outcome <sup>a</sup> | Response |
|---|---|---|
| Resolution of signs and symptoms of | Sustained clinical resolution | Clinical success |
| acute cystitis demonstrated at the TOC | | |
| Visit persist at the Follow-up Visit (and no | | |
| new signs and symptoms), without the | | |
| participant receiving other systemic | | |
| antimicrobials before the Follow-up Visit | | |
| Resolution of signs and symptoms of | Delayed clinical resolution | Clinical failure |
| acute cystitis present at Baseline (and no | | |
| new signs or symptoms), after clinical | | |
| failure at TOC, without the participant | | |
| receiving other systemic antimicrobials | | |
| before the Follow-up Visit | | |
| Improvement in total symptom scores | Clinical improvement | Clinical failure |
| from Baseline, but not complete | | |
| resolution, without the participant | | |
| receiving other systemic antimicrobials | | |
| before the Follow-up Visit | | |
| Worsening or no change in total symptom | Clinical worsening | Clinical failure |
| scores at Follow-up compared to Baseline | | |
| after clinical failure at TOC, or the | | |
| participant received other systemic | | |
| antimicrobials for the current infection | | |
| before or on the date of the Follow-up | | |
| Visit | | |
| Signs and symptoms of acute cystitis | Clinical recurrence | Clinical failure |
| reoccur at the Follow-up Visit after clinical | | |
| success at TOC | | 0" ' 16" |
| 1) The Baseline score is missing, or | Unable to determine | Clinical failure |
| 2) The Follow-up assessment is missing, | | |
| Or | | |
| 3) The participant received other | | |
| systemic antimicrobials not for the | | |
| current infection prior to the | | |
| assessment (unless the clinical | | |
| worsening or recurrence outcome | | |
| criteria were met) | | |

TOC = Test-of-Cure

a. A study physician or otherwise appropriately medically trained staff will determine the individual clinical signs and symptoms scores for acute cystitis (Appendix 6), which will then be used to programmatically determine the clinical outcome. The same scorer will be used at all assessment time points for each participant, on all occasions, whenever possible.



## 8.2. Safety Assessments

Planned time points for all safety assessments are provided in the SoA (Section 1.3).

## 8.2.1. Physical Examinations

- A physical examination will be performed at the time points indicated in the SoA (Section 1.3).
  - At Baseline, the examination will include assessments of the respiratory, CV, abdominal, gastrointestinal, neurological, and urogenital systems. Height and weight will only be measured and recorded at the Baseline Visit (before dosing).
  - At the TOC Visit, the physical examination may be symptom directed and is only required if indicated for a specific participant.
- Investigators should pay special attention to clinical signs related to previous serious illnesses.
- Clinically significant changes from baseline or clinically significant new clinical signs will be reported as AEs.

## 8.2.2. Vital Signs

- Vital signs will be measured at the time points indicated in the SoA (Section 1.3).
- Vital signs will be measured in a semi-supine position after 5 minutes rest and will include temperature, systolic and diastolic blood pressure, and pulse rate.

- Vital sign measurements should be obtained before any blood draws scheduled on the same assessment day.
- Clinically significant changes from baseline will be reported as AEs.

### 8.2.3. **Electrocardiograms**

- Electrocardiograms will be performed at the time points indicated in the SoA (Section 1.3).
- Triplicate 12-lead ECGs (over an approximate 5- to 10-minute period) will be performed using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals. Refer to Section 7.1.2 for QTc withdrawal criteria and additional QTc readings that may be necessary.
- Ideally, ECGs will be obtained before any vital sign measurements or blood draws scheduled on the same assessment day; however, sites may perform procedures in an order per their standard of care, as long as participants return to a resting state prior to the start of the ECG collections.
- Triplicate ECGs will be performed at Baseline.
- For the first approximately 1200 participants enrolled, On-therapy Visit triplicate ECGs will also be obtained. The On-therapy ECGs will be collected approximately 2 hours postdose (i.e., expected time of maximum concentration; ECG collection should ideally be within approximately 1.5 hours postdose to 4 hours postdose). After the first approximately 1200 participants have triplicate ECGs performed at On-therapy, the ECG collection at this visit is no longer a protocol requirement.
- If any additional ECGs are performed during the study (if deemed necessary by the investigator), those may be collected as a single ECG; however, if that initial single reading shows QTc prolongation, then triplicate ECGs should also be performed (see Section 7.1.2).
- If clinically significant changes occur during the study, they will be reported as AEs.
- Electrocardiograms will be reviewed locally by the investigator for safety purposes. Electrocardiograms will be centrally overread for the data analysis.

### 8.2.4. Clinical Safety Laboratory Assessments

- Refer to Appendix 8 for the list of clinical laboratory tests to be performed and to the SoA (Section 1.3) for the timing and frequency.
- The investigator must review the laboratory report, document this review, and record any clinically relevant changes occurring during the study in the AE section of the eCRF. The laboratory reports must be filed with the source documents. Clinically significant abnormal laboratory findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.

- All laboratory tests with values considered clinically significantly abnormal during participation in the study should be repeated until the values return to normal or baseline or are no longer considered significantly abnormal by the investigator or medical monitor.
- If such values do not return to normal/baseline within a period of time judged reasonable by the investigator, the etiology should be identified and the sponsor notified.
- All protocol-required laboratory assessments, as defined in Appendix 8 must be conducted in accordance with the laboratory manual and the SoA.

## 8.3. Adverse Events and Serious Adverse Events

The definitions of an AE or SAE can be found in Appendix 11.

Adverse events will be reported by the participant (or, when appropriate, by a caregiver, surrogate, or the participant's legally authorized representative).

The investigator and any qualified designees are responsible for detecting, documenting, and reporting events that meet the definition of an AE or SAE and remain responsible for following up AEs that are serious, considered related to the study treatment or the study, or that caused the participant to discontinue the study treatment or from the study (see Section 7).

## 8.3.1. Time Period and Frequency for Collecting AE and SAE Information

- All SAEs will be collected from the signing of the informed consent form until the Follow-up Visit at the time points specified in the SoA (Section 1.3).
- All AEs will be collected from the start of treatment until the Follow-up Visit at the time points specified in the SoA (Section 1.3).
- Medical occurrences that begin before the start of study treatment but after obtaining informed consent will be recorded on the Medical History/Current Medical Conditions section of the eCRF and not the AE section.
- All SAEs will be recorded and reported to the sponsor or designee immediately and under no circumstance should this exceed 24 hours, as indicated in Appendix 11. The investigator will submit any updated SAE data to the sponsor within 24 hours of it being available.
- Investigators are not obligated to actively seek AEs or SAEs after the conclusion of the study participation. However, if the investigator learns of any SAE, including a death, at any time after a participant has been discharged from the study, and he/she considers the event to be reasonably related to the study treatment or study participation, the investigator must promptly notify the sponsor.

## 8.3.2. Method of Detecting AEs and SAEs

- The method of recording, evaluating, and assessing causality of AEs and SAEs and the procedures for completing and transmitting SAE reports are provided in Appendix 11.
- Care will be taken not to introduce bias when detecting AEs and/or SAEs.
   Open-ended and nonleading verbal questioning of the participant is the preferred method to inquire about AE occurrence.

## 8.3.3. Follow-up of AEs and SAEs

After the initial AE/SAE report, the investigator is required to proactively follow each participant at subsequent visits/contacts. All SAEs, and nonserious AEs of special interest (as defined in Section 8.3.7), will be followed until the event is resolved, stabilized, otherwise explained, or the participant is lost to follow-up (as defined in Section 7.3). Further information on follow-up procedures is given in Appendix 11.

## 8.3.4. Regulatory Reporting Requirements for SAEs

- Prompt notification by the investigator to the sponsor of a SAE is essential so that legal obligations and ethical responsibilities towards the safety of participants and the safety of a study treatment under clinical investigation are met.
- The sponsor has a legal responsibility to notify both the local regulatory authority and other regulatory agencies about the safety of a study treatment under clinical investigation. The sponsor will comply with country-specific regulatory requirements relating to safety reporting to the regulatory authority, IRB/IEC, and investigators.
- For all studies except those utilizing medical devices, investigator safety reports
  must be prepared for suspected unexpected serious adverse reactions according
  to local regulatory requirements and sponsor policy and forwarded to
  investigators as necessary.
- An investigator who receives an investigator safety report describing a SAE or other specific safety information (e.g., summary or listing of SAEs) from the sponsor will review and then file it along with the IB and will notify the IRB/IEC, if appropriate according to local requirements.

## 8.3.5. Pregnancy

- Details of all pregnancies in female participants will be collected after the start of study treatment and through the Follow-up Visit.
- If a pregnancy is reported, the investigator should inform GSK within 24 hours of learning of the pregnancy and should follow the procedures outlined in Appendix 2.
- Abnormal pregnancy outcomes (e.g., spontaneous abortion, fetal death, stillbirth, congenital anomalies, ectopic pregnancy) are considered SAEs.
#### 8.3.6. Cardiovascular and Death Events

For any CV events detailed in Appendix 11 and all deaths, whether or not they are considered SAEs, specific CV and Death sections of the eCRF will be required to be completed. These sections include questions regarding CV (including sudden cardiac death) and non-CV death.

The CV eCRFs are presented as queries in response to reporting of certain CV Medical Dictionary for Regulatory Activities (MedDRA) terms. The CV information should be recorded in the specific CV section of the eCRF within 1 week of receipt of a CV Event data query prompting its completion.

The Death eCRF is provided immediately after the occurrence or outcome of death is reported. Initial and follow-up reports regarding death must be completed within 1 week of when the death is reported.

### 8.3.7. Adverse Events of Special Interest

Predefined AEs of special interest for this study are CV events, gastrointestinal events, *C. difficile* infection or colitis events, and AEs related to acetylcholinesterase inhibition (see Section 2.3.1), which will be identified by a prespecified list of coded terms or determined by algorithm, as described in the reporting and analysis plan (RAP). Additional details are provided in Appendix 11.

#### 8.4. Treatment of Overdose

There is no specific antidote for overdose with a bacterial topoisomerase inhibitor. In the event of a suspected overdose, it is recommended that the appropriate supportive clinical care should be instituted, as dictated by the participant's clinical status.

Occasional incidents of acute overdosage of nitrofurantoin have not resulted in any specific symptoms other than vomiting (refer to locally approved prescribing information). Induction of emesis is recommended. There is no specific antidote, but a high fluid intake should be maintained to promote urinary excretion of the drug.

In the event of an overdose, the investigator should:

- 1. Contact the medical monitor immediately.
- 2. Closely monitor the participant for AEs/SAEs and laboratory abnormalities until study treatment can no longer be detected systemically (at least 72 hours).
- 3. Obtain a plasma sample for PK analysis within 24 hours from the date of the last dose of study treatment if requested by the medical monitor (determined on a case-by-case basis).
- 4. Document the quantity of the excess dose as well as the duration of the overdosing in the case report form (CRF).

Decisions regarding dose interruptions or modifications will be made by the investigator in consultation with the medical monitor based on the clinical evaluation of the participant.

#### 8.5. Pharmacokinetics

Pharmacokinetics are not evaluated in this study.

## 8.6. Pharmacodynamics

Pharmacodynamics are not evaluated in this study.

#### 8.7. Genetics

A 6-mL blood sample for DNA isolation will be collected from participants who have consented to participate in the genetics analysis component of the study. Participation is optional. Participants who do not wish to participate in the genetic research may still participate in the study.

In the event of DNA extraction failure, a replacement genetic blood sample may be requested from the participant. Signed informed consent will be required to obtain a replacement sample unless it was included in the original consent.

Details on processes for collection and shipment and destruction of these samples can be found in Appendix 12.

#### 8.8. Biomarkers

Biomarkers are not evaluated in this study.

## 8.9. Immunogenicity Assessments

This section is not applicable.



#### 9. STATISTICAL CONSIDERATIONS

Full details of all data handling conventions and statistical analyses conducted for this study will be provided in the RAP.

## 9.1. Statistical Hypotheses

The study is designed to demonstrate that gepotidacin administered orally is noninferior compared to nitrofurantoin administered orally on the primary efficacy endpoint of therapeutic response (combined per-participant microbiological and clinical response) at the TOC Visit in participants with a qualifying bacterial uropathogen at Baseline that is susceptible to nitrofurantoin. Microbiological success is defined as eradication (i.e., reduction of all qualifying bacterial uropathogens recovered at Baseline to <10<sup>3</sup> CFU/mL as observed on quantitative urine culture) without the participant receiving other systemic antimicrobials. Clinical success is defined as resolution of signs and symptoms of acute cystitis present at Baseline (and no new signs and symptoms) without the participant receiving other systemic antimicrobials.

The following are null and alternative hypotheses for the primary analysis of the therapeutic success rates at the prespecified noninferiority margin of -10.0%:

H<sub>0</sub>: therapeutic success rate of gepotidacin 1500 mg BID – therapeutic success rate of nitrofurantoin 100 mg BID ≤-10.0%

 $H_1$ : therapeutic success rate of gepotidacin 1500 mg BID – therapeutic success rate of nitrofurantoin 100 mg BID >-10.0%

The use of a -10% noninferiority margin in the primary efficacy estimand is in accordance with current FDA guidance [DHHS, 2019; EMA, 2013].

If noninferiority is declared between gepotidacin and nitrofurantoin, superiority will be tested with the following null and alternative hypotheses:

H<sub>0</sub>: therapeutic success rate of gepotidacin 1500 mg BID – therapeutic success rate of nitrofurantoin 100 mg BID ≤0%

H<sub>1</sub>: therapeutic success rate of gepotidacin 1500 mg BID – therapeutic success rate of nitrofurantoin 100 mg BID >0%

An IA is planned as described in Section 9.5. The study will utilize a group sequential design with 1 IA using Lan-DeMets spending function [Lan, 1983]. The timing of the IA is planned to occur when approximately 60% of the maximum planned participants in the micro-ITT NTF-S Population (N≈884) have achieved the TOC Visit. The stopping boundary for assessing efficacy will use the Pocock stopping rule for efficacy and the O'Brien-Flemming stopping rule for futility. At the time of the IA, the IDMC will perform an unblinded review to confirm that there are sufficient microbiological data for regulatory submission before proceeding to the IA for efficacy and futility. If in any case the microbiological data are not sufficient, the IDMC will instead conduct a futility-only IA. If futility is not declared, the sample size needed for the final analysis will be approximately 768 participants in the micro-ITT NTF-S Population. This will be based on the O'Brien-Flemming stopping boundary for futility. Details on the timing and design selection process are described in Section 9.5.

## 9.2. Sample Size Determination

#### 9.2.1. Justification of Sample Size

Participants will be randomized to gepotidacin and nitrofurantoin in a 1:1 ratio. Assuming a 76% therapeutic success rate for both nitrofurantoin and gepotidacin, a sample size of approximately 884 participants in the micro-ITT NTF-S Population is required, for a design with 1 IA allowing for stopping the study based on efficacy or futility, to provide approximately 90% power to demonstrate noninferiority in the therapeutic response rate of gepotidacin to nitrofurantoin with a 0.025 one-sided alpha level and a -10.0% noninferiority margin. The minimal response rate difference that would meet the statistical criterion for noninferiority is provided in Table 12.

Table 12 Minimal Response Rate Difference for Efficacy and Futility Interim Analysis

| Design | Information<br>Fraction | Micro-ITT NTF-S<br>Sample Size | Minimal Response Rate Difference<br>for Noninferiority |
|---|---|---|---|
| Analysis for Efficiency and Eutility | 60% | 530 | -2.2% |
| Analysis for Efficacy and Futility | 100% | 884 | -3.6% |

Micro-ITT NTF-S=Microbiological Intent-to-Treat Nitrofurantoin-Susceptible.

In case a futility-only IA is conducted, under the same assumption for response rate, significance level, and noninferiority margin, a sample size of 768 participants in the micro-ITT NTF-S Population will provide approximately 88% power to demonstrate noninferiority. The minimal response rate difference that would meet the statistical criterion for noninferiority is -4.0% for the final analysis.

The study is planned to enroll approximately 2500 participants to ensure a sufficient number of participants in the primary analysis population (i.e., micro-ITT NTF-S Population). If the study proceeds to an efficacy and futility IA, the maximum target sample size (assuming there is a decision to continue the study at the IA) for the primary analysis population will be around 884 participants. If the study proceeds to the futility-only IA, the maximum target sample size (assuming a decision to continue the study at the IA) for the primary analysis population will be approximately 768 participants. The final number of randomized participants may vary based on the evaluability rate and review of qualifying uropathogens by an unblinded SDAC.

**Note**: "Enrolled" means that a participant's or their legally acceptable representative's agreement to participate in the clinical study following completion of the informed consent process. Potential participants who are screened for the purpose of determining eligibility for the study, but do not participate in the study, are not considered enrolled, unless otherwise specified in the protocol.

## 9.2.2. Sample Size Sensitivity

Sensitivity of the sample size has been explored considering various therapeutic success rates. Table 13 and Table 14 show the minimum power under various assumptions of

"true" therapeutic success rates of gepotidacin and nitrofurantoin under 2 different IA designs, when the IA is conducted at approximately 60% information fraction of the design allowing for efficacy and futility stop at the IA. For all of these cases, the 1-sided type I error is 2.5%, the noninferiority margin is -10%.

Table 13 Power of the Study Under Various Assumptions of the True Therapeutic Success Rates for Efficacy and Futility Group Sequential Design

| Therapeutic<br>Success Rate of<br>Nitrofurantoin | Therapeutic<br>Success Rate<br>of Gepotidacin | Total Number of<br>Participants in<br>the Primary<br>Analysis | Number of<br>Participants in the<br>Primary Analysis in<br>the Interim Analysis | Power |
|---|---|---|---|---|
| 76% | 76% | 884 | 530 | 90% |
| 72% | 72% | 884 | 530 | 87% |
| 68% | 68% | 884 | 530 | 84% |
| 64% | 64% | 884 | 530 | 81% |
| 60% | 60% | 884 | 530 | 79% |

Table 14 Power of the Study Under Various Assumptions of the True Therapeutic Success Rates for Futility Only Group Sequential Design

| Therapeutic<br>Success Rate of<br>Nitrofurantoin | Therapeutic<br>Success Rate of<br>Gepotidacin | Total Number of<br>Participants in<br>the Primary<br>Analysis | Number of<br>Participants in the<br>Primary Analysis in<br>the Interim Analysis | Power |
|---|---|---|---|---|
| 76% | 76% | 768 | 530 | 88% |
| 72% | 72% | 768 | 530 | 85% |
| 68% | 68% | 768 | 530 | 81% |
| 64% | 64% | 768 | 530 | 79% |
| 60% | 60% | 768 | 530 | 77% |

## 9.3. Populations for Analyses

For purposes of analysis, the following populations are defined:

| Population | Description |
|---|---|
| Intent-to-Treat (ITT) Population | All participants randomly assigned to study treatment. Participants will be analyzed according to their randomized study treatment. |

| Population | Description |
|---|---|
| Microbiological ITT (micro-ITT) Population | All participants randomly assigned to study treatment who receive at least 1 dose of study treatment and have a qualifying baseline uropathogen (defined in Appendix 4), from a quantitative bacteriological culture of a pretreatment clean-catch midstream urine specimen. Participants will be analyzed according to their randomized study treatment. |
| Micro-ITT NTF-S<br>Population | All participants in the micro-ITT Population whose baseline qualifying bacterial uropathogens all are susceptible to nitrofurantoin (NTF-S). Participants with missing MIC susceptibility results for any qualifying uropathogens will not be included in the NTF-S subpopulation. Participants will be analyzed according to their randomized study treatment. This is the primary analysis population. |
| Micro-ITT NTF-NS Population | All participants in the micro-ITT Population who have any qualifying baseline bacterial uropathogens that are not susceptible to nitrofurantoin (NTF-NS), defined as resistant to nitrofurantoin, intermediate to nitrofurantoin, or have no interpretation to nitrofurantoin. Participants with missing MIC susceptibility results for all qualifying uropathogens will not be included in the NTF-NS subpopulation. Participants will be analyzed according to their randomized study treatment. |
| Microbiologically Evaluable (ME) Population | Participants who meet the definition of the micro-ITT Population, follow important components of the study (as specified in the RAP) and have an interpretable quantitative urine culture at the specified visit. Note: Visit-specific ME populations will be defined in the RAP. |
| ME NTF-S Population | All participants in the ME visit-specific population whose baseline qualifying bacterial uropathogens all are susceptible to nitrofurantoin (NTF-S). Note: Visit-specific ME NTF-S populations will be defined in the RAP. |
| ME NTF-NS Population | All participants in the ME visit-specific population who have any baseline qualifying bacterial uropathogens that are not susceptible to nitrofurantoin (NTF-NS). Note: Visit-specific ME NTF-NS populations will be defined in the RAP. |
| Clinically Evaluable (CE)<br>Population | All participants in the ITT Population who follow important components of the study as specified in the RAP. Note: Visit-specific CE populations will be defined in the RAP. |

| Population | Description |
|---|---|
| Safety Population | All randomized participants who receive at least 1 dose of study treatment. Participants will be analyzed according to their actual treatment received. |

## 9.4. Statistical Analyses

The RAP will be finalized prior to unblinding and will include a more technical and detailed description of the statistical analyses described in this section. This section is a summary of the planned statistical analyses of the most important endpoints including primary, secondary, and exploratory endpoints.

#### 9.4.1. General Considerations

Treatment effect to be estimated for primary and secondary estimands are clinical outcome/response, microbiological outcome/response, and therapeutic response at the designated visits in female participants with acute cystitis (clinical outcome/response) and female participants with acute cystitis with qualifying bacterial uropathogen(s) at Baseline that all are susceptible to nitrofurantoin (clinical outcome/response, microbiological outcome/response, and therapeutic response). Intercurrent events include receiving other systemic antimicrobials and treatment discontinuation; a combination of composite strategy and treatment policy strategy will be implemented to account for the 2 ICEs, respectively. The ICE event strategies determine that (1) treatment effects will be estimated regardless of study treatment discontinuation when the analysis population is the ITT Population or its derivatives; and (2) the definition of a successful response or a positive outcome (clinical resolution and microbiological eradication) precludes the use of other systemic antimicrobials.

Any supplemental analyses will be detailed in the RAP. Any additional analyses or outputs needed as a result of COVID-19 on the study will be detailed in the RAP.

## 9.4.2. Efficacy Analyses

| Estimands/Endpoints | Statistical Analysis Methods |
|---|---|
| Primary | The primary analysis of the primary efficacy endpoint will be performed using the micro-ITT NTF-S Population. |
| | • The primary treatment effect to be estimated (estimand) is therapeutic response (combined per-participant microbiological and clinical response) at the TOC Visit in female participants with acute cystitis with a qualifying bacterial uropathogen(s) at Baseline that all are susceptible to nitrofurantoin. Microbiological success at the TOC Visit is defined as reduction of all qualifying bacterial uropathogens recovered at Baseline to <10³ CFU/mL as observed on quantitative urine culture without the participant receiving other systemic antimicrobials; clinical success is defined as resolution of signs and symptoms of acute cystitis present at Baseline (and no new signs and symptoms) without the participant receiving other systemic antimicrobials. Therapeutic success refers to participants who have been deemed both a microbiological success and a clinical success (i.e., responders). The primary treatment effect will be estimated regardless of treatment discontinuation, as per the treatment policy strategy. The ICE of use of other systemic antimicrobial therapy is captured through the definitions of microbiological and clinical response and will be counted as failures (composite strategy). If a participant experiences both ICEs of study treatment discontinuation and use of systemic antimicrobials, then a composite strategy (assigning therapeutic response as a failure) will be used from the point that the relevant systemic antimicrobial was taken. Further details on the primary estimand are provided in Section 3. |
| | The population-level effect will be estimated by the difference in percentage response and its 95% CI. For this analysis, participants who do not return for the TOC Visit or have missing data at the TOC Visit will be treated as failures. |
| | The number and percentage of participants with therapeutic success will be summarized, along with the 95% CI, at the TOC Visit by treatment group. |

| Estimands/Endpoints | Statistical Analysis Methods |
|---|---|
| • | • The testing procedure at the IA and the final analysis involves comparing the noninferiority test statistics with the stopping boundary. Test statistics of the therapeutic success rate difference between the 2 treatment groups for noninferiority (-10% margin) will be calculated using the Miettinen and Nurminen method stratified by age category (<18 years, ≥18 to 50 years, or >50 years) and acute cystitis recurrence (nonrecurrent infection or recurrent infection) [Miettinen, 1985] and compared to the stopping boundaries. If noninferiority is established, test statistics of the success rate difference between the 2 treatment groups for superiority will be calculated using the same method to compare with the stopping boundary for superiority. Details on the testing procedure and stopping boundaries are provided in the IDMC analysis plan. |
| | <ul> <li>In the event that a participant is mis-stratified at randomization, the<br/>actual stratum will be used instead of the randomized stratum in<br/>the primary analysis.</li> </ul> |
| | <ul> <li>Sensitivity analysis on the primary endpoint will be done with<br/>details provided in the RAP. In addition, a tipping point analysis<br/>may be performed for the primary estimand, if warranted by the<br/>degree of missing data.</li> </ul> |
| | <ul> <li>Subgroup analysis and supplemental analysis on additional<br/>populations for the primary endpoint may be performed with<br/>details provided in the RAP.</li> </ul> |
| | Handling of protocol deviations will be described in the RAP. |

| Estimands/Endpoints | Statistical Analysis Methods |
|---|---|
| Secondary | Secondary efficacy endpoints for clinical outcome and response will be summarized using the ITT Population and micro-ITT NTF-S Population. Secondary efficacy endpoints for microbiological outcome and response, as well as therapeutic response, will be summarized using the micro-ITT NTF-S Population. |
| | <ul> <li>There will be no multiplicity adjustment for the testing of the<br/>secondary endpoints. No formal hypothesis testing will be<br/>performed.</li> </ul> |
| | The clinical outcome and response (number and percentage of participants with resolution of signs and symptoms) will be summarized by treatment group at the TOC and Follow-up Visits. The ICE of use of other systemic antimicrobials is captured through the defining criteria of clinical outcome and response (Section 8.1.3.1). |
| | The microbiological outcome and response (number and percentage of participants with microbiological success) will be summarized by treatment group at the TOC and Follow-up Visits. The ICE of use of other systemic antimicrobials is captured through the defining criteria of microbiological outcome and response (Section 8.1.2.1). |
| | Therapeutic response (combined per-participant microbiological<br>and clinical response) will be summarized by treatment group at<br>the Follow-up Visit. |
| | Sensitivity analysis on the secondary endpoints, if warranted, will be described in the RAP. |
| | Subgroup analysis by qualifying baseline uropathogen will be done for microbiological outcome and response at relevant visits. Additional subgroup analyses and supplemental analysis on additional populations may be carried out. Details of these analyses will be provided in the RAP. |

212390



#### 9.4.3. Safety Analyses

All safety analyses will be performed on the Safety Population. The severity of AEs and SAEs will be determined by the investigator according to the US National Institute of Allergy and Infectious Diseases Division of Microbiology and Infectious Diseases (DMID) criteria for adult toxicity assessment [DMID, 2007a], with the exception of serum creatinine adolescent laboratory data, which will be assessed using pediatric toxicity criteria [DMID, 2007b] (Appendix 13). All reported AEs will be coded using MedDRA and summarized by system organ class and preferred terms.

| Estimands/Endpoints | Statistical Analysis Methods |
|---|---|
| Secondary | <ul> <li>The safety endpoint will use a treatment policy strategy for the ICE<br/>of withdrawal from treatment, as safety will be assessed at all<br/>postbaseline assessments irrespective of whether the participant<br/>completed the treatment.</li> </ul> |

| Estimands/Endpoints | Statistical Analysis Methods |
|---|---|
| | The number and percentage of treatment-emergent AEs, study treatment-related AEs, deaths, SAEs, and AEs leading to study treatment or study withdrawal will be provided. |
| | Treatment-emergent AEs will be summarized by severity. |
| | <ul> <li>Change from baseline over time in laboratory parameters, ECGs,<br/>and vital signs will be summarized with descriptive statistics.</li> <li>Note: Electrocardiograms will be centrally overread for the data<br/>analysis.</li> </ul> |
| | The frequency of laboratory abnormality events along with the shift from baseline to the worst-case postbaseline value will be provided. Abnormal liver chemistry results will be determined using increases above the upper limit of normal. Change from baseline values will be summarized with descriptive statistics. |
| | The severity of specified AEs and laboratory abnormalities will be graded according to the modified DMID toxicity grading system (Appendix 13). Data will be tabulated and reported by absolute grade for Grades 3 and higher and shift tables, as appropriate. |
| | <ul> <li>Adverse events of special interest will include CV, gastrointestinal,<br/>and C. difficile infection or colitis events. In addition, AEs<br/>associated with acetylcholinesterase inhibition are also considered<br/>special interest. As described in the RAP, manual and<br/>programmatic reviews of AEs/preferred terms will be used to<br/>assess these events.</li> </ul> |

## 9.5. Interim Analysis

One IA is planned to assess either both efficacy and futility or just futility by the IDMC. The IDMC will meet when approximately 60% of participants in the micro-ITT NTF-S Population have achieved the TOC Visit to evaluate the primary endpoint, identify potential treatment benefit, and make recommendations for continuing or stopping the study, as per the IDMC charter. The IDMC members will include at least 3 independent experts, including an infectious disease specialist, a chairperson with experience chairing IDMC meetings, and a statistician. Details regarding the IDMC process will be described in the IDMC charter.

The SDAC will conduct and provide all unblinded analyses to the IDMC before the meeting is held. Details on the content and structure of the data output will be described in a separate IDMC analysis plan. The GSK and PPD study teams that are operating the study and conducting the final analysis will remain blinded. The IDMC and SDAC will maintain unblinded data in a secure area to ensure the integrity of the data until the study is completed. Details on protecting blind and data integrity will be described in a blinding plan.

At the time the IA is conducted, the IDMC will review unblinded data to confirm that sufficient microbiological data exist for the unblinded gepotidacin treatment arm before deciding how to proceed.

If the IDMC confirms there is sufficient microbiology data in the gepotidacin arm, an IA with stopping rules for both efficacy and futility will be performed. The nominal significance levels for the interim and final analyses will be determined by the Lan-DeMets spending functions approach [Lan, 1983]. This will be based on the Pocock stopping boundary for efficacy and the O'Brien-Flemming stopping boundary for futility. The futility bounds of this study are nonbinding and are considered guidance rather than strict bounds.

During the course of the IA, the accrual of the study will continue. If efficacy success is reached at the IA and the study is stopped early, data collected between the IA data cut and IA decision are considered overrun. Overrun data will be pooled with the IA data to repeat the primary efficacy analysis as sensitivity analysis.

During the course of the IA, the accrual of the study will continue. If efficacy success (i.e., noninferiority) is reached at the IA and the study is stopped early, the IA will be the primary analysis and data collected between the IA data cut and the time when the study is stopped will be considered overrun. Overrun data will be pooled with the IA data to repeat the primary efficacy analysis as sensitivity analysis. If efficacy success is not reached at the IA, the study will continue to the maximum target sample size for the micro-ITT NTF-S Population of approximately 884 participants.

Details on timing, microbiological data criteria, design selection, and stopping boundaries for the IA are described in the IDMC charter.

A GSK SRT will review the blinded safety data of this study at regular intervals. Details regarding the SRT process will be available in relevant SRT documents. The SRT will inform the IDMC if any safety signals are identified.

## 9.6. Data Monitoring Committee or Other Review Board

This study will have an IDMC as described in Section 9.5. In addition, there will be a GSK SRT and Microbiology Review Team. For details on these review teams, refer to Appendix 3.

# 10. SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS

## 10.1. Appendix 1: *Clostridium Difficile* Testing Procedure and Algorithm

Signs/Symptoms indicate possible GI disturbance and Subject has ≥3 non-formed stool specimens in a 24 hour period or a significant change from baseline Collect specimen in a sterile container (no preservative) Transport to local lab at 2-8°C\* Local lab performs testing or sends to a reference lab (if according to their procedures\*\*) Freeze remaining portion of sample and save for further testing (if necessary) GDH Assay Toxin A/B assay (EIA) or Cytotoxin Neutralization (can be conducted in parallel with GDH assay) (lab performs as 1°/ stand alone test) positive= positive= negative= positive negative= negative Negative for Positive for Negative for Positive for Toxigenic Toxigenic Toxigenic Toxigenic C. difficile C. difficile C. difficile C. difficile Toxin A/B assay (EIA) or Cytotoxin Neutralization NAAT assay or Toxigenic Culture For any specimens determined to be positive for positive= Not Available negative positive= negative = toxigenic Positive for Positive for Negative for C. difficile Toxigenic Toxigenic Toxigenic Maintain storage of C. difficile C. difficile C. difficile remaining frozen specimen Contact CRA and refer to SRM NAAT assay or Toxigenic Culture Instructions will be provided to send frozen specimen to a reference lab for C. difficile culture and for molecular negative= positive= typing Positive for Negative for Toxigenic Toxigenic

C. difficile

C. difficile

Note: This algorithm is subject to investigator discretion when the clinical presentation and time course of diarrhea (e.g., during or within 12 hours immediately after dosing) do not fit the Clostridium difficile-associated diarrhea definition; consideration should be given to diarrhea occurring in this early time frame to be suggestive of a cholinergic effect.

<sup>\*</sup>If processing and testing cannot be performed within 24 hours, the specimen should be frozen immediately after collection.

<sup>\*\*</sup>If specimen is sent to a reference laboratory, the procedures to be ordered should follow the same algorithm above.

GDH = glutamate dehydrogenase; NAAT = nucleic acid amplification test

CRA = clinical research associate (PPD site monitor); SRM = Study Reference Manual

# 10.2. Appendix 2: Contraceptive Guidance and Collection of Pregnancy Information

#### 10.2.1. Definitions:

### Woman of Childbearing Potential (WOCBP)

A woman is considered fertile following menarche and until becoming postmenopausal unless permanently sterile (see below).

If fertility is unclear (e.g., amenorrhea in adolescents or athletes) and a menstrual cycle cannot be confirmed before first dose of study treatment, additional evaluation should be considered.

#### Women in the following categories are not considered WOCBP

- 1. Premenarchal
- 2. Premenopausal female with 1 of the following:
  - Documented hysterectomy
  - Documented bilateral salpingectomy
  - Documented bilateral oophorectomy

For individuals with permanent infertility due to an alternate medical cause other than the above, (e.g., mullerian agenesis, androgen insensitivity), investigator discretion should be applied to determining study entry.

**Note:** Documentation can come from the site personnel's: review of the participant's medical records, medical examination, or medical history interview.

- 3. Postmenopausal female
  - A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
    - A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy (HRT). However, in the absence of 12 months of amenorrhea, confirmation with more than one FSH measurement is required.
  - Females on HRT and whose menopausal status is in doubt will be required to
    use 1 of the non-estrogen hormonal highly effective contraception methods if
    they wish to continue their HRT during the study. Otherwise, they must
    discontinue HRT to allow confirmation of postmenopausal status before
    study enrollment.
  - Refer to Appendix 8 for pregnancy testing requirements.

## 10.2.2. Contraception Guidance:

Refer to Appendix 8 regarding pregnancy testing for female participants at Baseline (Day 1) and associated pretreatment contraception and abstinence requirements. Female participants who enter the study using contraception must continue to do so throughout the study.

As described in Section 5.3, participants will be requested to abstain from sexual activity from the Baseline Visit through the TOC Visit to prevent possible re-infection.

#### CONTRACEPTIVES<sup>a</sup> ALLOWED DURING THE STUDY INCLUDE:

- Highly Effective Methods<sup>b</sup> That Have Low User Dependency Failure rate of <1% per year when used consistently and correctly
- Implantable progestogen-only hormone contraception associated with inhibition of ovulation<sup>c</sup>
- Intrauterine device (IUD)
- Intrauterine hormone-releasing system (IUS)<sup>c</sup>
- Bilateral tubal occlusion
- Vasectomized partner
  - Note: Vasectomized partner is a highly effective contraceptive method provided that
    the partner is the sole sexual partner of the woman of childbearing potential and the
    absence of sperm has been confirmed. If not, an additional highly effective method of
    contraception should be used. Spermatogenesis cycle is approximately 90 days.
- **Highly Effective Methods**<sup>b</sup> **That Are User Dependent** *Failure rate of <1% per year when used consistently and correctly*
- Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation<sup>c</sup>
  - oral
  - intravaginal
  - transdermal
  - injectable
- Progestogen-only hormone contraception associated with inhibition of ovulation<sup>c</sup>
  - oral
  - injectable
- Sexual abstinence
  - Note: Sexual abstinence is considered a highly effective method only if defined as
    refraining from heterosexual intercourse during the entire period of risk associated with
    the study treatment. The reliability of sexual abstinence needs to be evaluated in
    relation to the duration of the study and the preferred and usual lifestyle of the
    participant.
- a. Contraceptive use by men or women should be consistent with local regulations regarding the use of contraceptive methods for those participating in clinical studies.

- b. Failure rate of <1% per year when used consistently and correctly. Typical use failure rates differ from those when used consistently and correctly.
- c. Male condoms must be used in addition to hormonal contraception. If locally required, in accordance with Clinical Trial Facilitation Group (CTFG) guidelines, acceptable contraceptive methods are limited to those which inhibit ovulation as the primary mode of action.

Note: Periodic abstinence (calendar, sympto-thermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhoea method (LAM) are not acceptable methods of contraception. Male condom and female condom should not be used together (due to risk of failure with friction).

## 10.2.3. Collection of Pregnancy Information:

### Female participants who become pregnant

- Investigator will collect pregnancy information on any female participant, who becomes pregnant while participating in this study.
- The initial information will be recorded on the appropriate form and submitted to GlaxoSmithKline (GSK)/PPD within 24 hours of learning of a participant's pregnancy.
- Participant will be followed to determine the outcome of the pregnancy. The investigator will collect follow-up information on participant and neonate, which will be forwarded to GSK. Generally, follow-up will not be required for longer than 6 to 8 weeks beyond the estimated delivery date.
- Any termination of pregnancy will be reported, regardless of fetal status (presence or absence of anomalies) or indication for procedure.
- While pregnancy itself is not considered to be an adverse event (AE) or serious AE
  (SAE), any pregnancy complication or elective termination of a pregnancy for
  medical reasons will be reported as an AE or SAE.
- A spontaneous abortion (occurring at <22 weeks gestational age) or still birth (occurring at >22 weeks gestational age) is always considered to be an SAE and will be reported as such.
- Any SAE occurring as a result of a poststudy pregnancy that is considered reasonably related to the study treatment by the investigator, will be reported to GSK/PPD as described in Appendix 11. While the investigator is not obligated to actively seek this information in former study participants, he or she may learn of an SAE through spontaneous reporting.

Any female participant who becomes pregnant while participating will discontinue study treatment.

## 10.3. Appendix 3: Regulatory, Ethical, and Study Oversight Considerations

## 10.3.1. Regulatory and Ethical Considerations

- This study will be conducted in accordance with the protocol and with:
  - Consensus ethical principles derived from international guidelines including the Declaration of Helsinki and Council for International Organizations of Medical Sciences (CIOMS) International Ethical Guidelines
  - Applicable International Council on Harmonisation (ICH) Good Clinical Practice (GCP) Guidelines
  - Applicable laws and regulations
- The protocol, protocol amendments, informed consent form (ICF)/assent form/eConsent (if applicable), investigator's brochure, and other relevant documents (e.g., advertisements) must be submitted to an institutional review board/independent ethics committee (IRB/IEC) by the investigator and reviewed and approved by the IRB/IEC before the study is initiated.\*
- Any amendments to the protocol will require IEC/IRB approval before implementation of changes made to the study design, except for changes necessary to eliminate an immediate hazard to study participants.
- The investigator will be responsible for the following:
  - Providing written summaries of the status of the study to the IRB/IEC annually or more frequently in accordance with the requirements, policies, and procedures established by the IRB/EC\*
  - Notifying the IRB/IEC of serious adverse events (SAEs) or other significant safety findings as required by IRB/IEC procedures\*
  - Providing oversight of the conduct of the study at the site and adherence to requirements of 21 Code of Federal Regulations (CFR), ICH guidelines, the IRB/IEC, European regulation 536/2014 for clinical studies (if applicable), and all other applicable local regulations

\*Note: In countries where the responsibility to perform these submissions and notifications resides with the sponsor rather than the investigator, GSK or their designee PPD (as described in the applicable powers of attorney) will take these responsibilities.

#### 10.3.2. Financial Disclosure

Investigators and subinvestigators will provide the sponsor with sufficient, accurate financial information as requested to allow the sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate regulatory authorities. Investigators are responsible for providing information on financial interests during the course of the study and for 1 year after completion of the study.

#### 10.3.3. Informed Consent/Assent Process

- The investigator or his/her representative will explain the nature of the study to the participant or her legally authorized representative and answer all questions regarding the study.
- Participants must be informed that their participation is voluntary. Participants
  or their legally authorized representative will be required to sign a statement of
  informed consent and/or eConsent (if applicable) that meets the requirements of
  21 CFR 50, local regulations, ICH guidelines, Health Insurance Portability and
  Accountability Act (HIPAA) requirements, where applicable, and the IRB/IEC
  or study site.
- The medical record must include a statement that written informed consent and/or eConsent (if applicable) was obtained before the participant was enrolled in the study and the date informed consent was obtained. The authorized person obtaining the informed consent must also sign the ICF.
- Participants must be re-consented to the most current version of the ICF(s)/eConsent during their participation in the study.
- A copy of the ICF(s)/eConsent must be provided to the participant or the participant's legally authorized representative.
- Adolescent participants should be asked for their written assent or eConsent (if applicable) to participate in the study.
- As applicable, the IRB/IEC will be consulted before assent form development for guidance around age-appropriate groupings and any specific IRB/IEC requirements or local laws for conducting and documenting assent.

Participants who are rescreened are required to sign a new ICF or provide eConsent (if applicable).

GSK (alone or working with others) may use participant's coded study data and samples and other information to carry out this study; understand the results of this study; learn more about gepotidacin or about the study disease; publish the results of these research efforts; work with government agencies or insurers to have gepotidacin approved for medical use or approved for payment coverage.

#### 10.3.4. Data Protection

- Participants will be assigned a unique identifier by the sponsor. Any participant records or datasets that are transferred to the sponsor will contain the identifier only; participant names or any information which would make the participant identifiable will not be transferred.
- The participant must be informed that her personal study-related data will be used by the sponsor in accordance with local data protection law. The level of disclosure must also be explained to the participant who will be required to give consent for their data to be used as described in the informed consent.

 The participant must be informed that her medical records may be examined by Clinical Quality Assurance auditors or other authorized personnel appointed by the sponsor, by appropriate IRB/IEC members, and by inspectors from regulatory authorities.

#### 10.3.5. Committees Structure

To protect the safety interests of participants, a GlaxoSmithKline (GSK) Safety Review Team will review blinded safety data instream on a regular basis throughout study conduct. Data reviewers will include but are not limited to the following participants: medical monitor, safety team lead, statistician, clinical team lead, and data quality lead.

A Microbiology Review Team will monitor blinded uropathogen identification and susceptibility data instream, including the enrollment rate of participants with a qualifying bacterial uropathogen at Baseline and the resistance profile of uropathogens.

Procedures will be described in a separate microbiology sample monitoring plan.

An Independent Data Monitoring Committee will manage the interim analysis, with details provided in a separate charter and analysis plan.

Written documentation regarding key decisions made by the review teams/committee will be promptly distributed to participating investigators and IRB/IECs.

#### 10.3.6. Dissemination of Clinical Study Data

- Where required by applicable regulatory requirements, an investigator signatory will be identified for the approval of the clinical study report. The investigator will be provided reasonable access to statistical tables, figures, and relevant reports and will have the opportunity to review the complete study results at a GSK site or other mutually agreeable location.
- GSK will also provide the investigator with the full summary of the study results. The investigator is encouraged to share the summary results with the study participants, as appropriate.
- GSK will provide the investigator with the randomization codes for their site only after completion of the full statistical analysis.
- The procedures and timing for public disclosure of the protocol and results summary and for development of a manuscript for publication for this study will be in accordance with GSK policy.
- GSK intends to make anonymized participant-level data from this trial available
  to external researchers for scientific analyses or to conduct further research that
  can help advance medical science or improve patient care. This helps ensure the
  data provided by trial participants are used to maximum effect in the creation of
  knowledge and understanding.

TMF-13817737 212390

#### 10.3.7. **Data Quality Assurance**

- All participant data relating to the study will be recorded on printed CRFs or electronic CRFs (eCRFs) unless transmitted to the sponsor or designee electronically (e.g., laboratory data). The investigator is responsible for verifying that data entries are accurate and correct by physically or electronically signing the eCRF.
- The investigator must maintain accurate documentation (source data) that supports the information entered in the eCRF.
- The investigator must permit study-related monitoring, audits, IRB/IEC review, and regulatory agency inspections and provide direct access to source data documents.
- Monitoring details describing strategy (e.g., risk-based initiatives in operations and quality such as Risk Management and Mitigation Strategies and Analytical Risk-Based Monitoring), methods, responsibilities and requirements, including handling of noncompliance issues and monitoring techniques (central, remote, or on-site monitoring) are provided in the Monitoring Plan. In addition, refer to Appendix 5 for details regarding allowed revisions to study conduct and/or monitoring due to COVID-19.
- The sponsor or designee is responsible for the data management of this study including quality checking of the data. Detailed information about study data collection and management process can be found in the Data Validation Manual.
- The sponsor assumes accountability for actions delegated to other individuals (e.g., contract research organizations).
- Study monitors will perform ongoing source data verification to confirm that data entered into the eCRF by authorized site personnel are accurate, complete, and verifiable from source documents; that the safety and rights of participants are being protected; and that the study is being conducted in accordance with the currently approved protocol and any other study agreements, ICH GCP, and all applicable regulatory requirements. In addition, refer to Appendix 5 for details regarding allowed revisions to study conduct and/or monitoring due to COVID-19.
- Records and documents, including signed ICF, pertaining to the conduct of this study must be retained by the investigator for 25 years from the issue of the final clinical study report/ equivalent summary unless local regulations or institutional policies require a longer retention period. No records may be destroyed during the retention period without the written approval of the sponsor. No records may be transferred to another location or party without written notification to the sponsor.

#### 10.3.8. **Source Documents**

Source documents provide evidence for the existence of the participant and substantiate the integrity of the data collected. Source documents are filed at the investigator's site.

- Data reported on the CRF or entered in the eCRF that are transcribed from source documents must be consistent with the source documents or the discrepancies must be explained. The investigator may need to request previous medical records or transfer records, depending on the study. Also, current medical records must be available.
- Definition of what constitutes source data can be found in the Study Reference Manual.

### 10.3.9. Study and Site Start and Closure

GSK or its designee reserves the right to close the study site or terminate the study at any time for any reason at the sole discretion of GSK. Study sites will be closed upon study completion. A study site is considered closed when all required documents and study supplies have been collected and a study-site closure visit has been performed.

The investigator may initiate study-site closure at any time, provided there is reasonable cause and sufficient notice is given in advance of the intended termination.

Reasons for the early closure of a study site by the sponsor or investigator may include but are not limited to:

- Failure of the investigator to comply with the protocol, the requirements of the IRB/IEC or local health authorities, the sponsor's procedures, or GCP guidelines
- Inadequate recruitment of participants by the investigator
- Discontinuation of further study treatment development

If the study is prematurely terminated or suspended, the sponsor shall promptly inform the investigators, the IECs/IRBs, the regulatory authorities, and any contract research organization(s) used in the study of the reason for termination or suspension, as specified by the applicable regulatory requirements. The investigator shall promptly inform the participant and should assure appropriate participant therapy and/or follow-up.

## 10.3.10. Publication Policy

- The results of this study may be published or presented at scientific meetings. If this is foreseen, the investigator agrees to submit all manuscripts or abstracts to the sponsor before submission. This allows the sponsor to protect proprietary information and to provide comments.
- The sponsor will comply with the requirements for publication of study results.
   In accordance with standard editorial and ethical practice, the sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement.
- Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

## 10.4. Appendix 4: Algorithm for Determining Qualifying Uropathogens

In addition to other criteria indicated in Section 9.3, to be included in the micro-ITT Population, participants must have a qualifying bacterial uropathogen (defined in Figure 2) at Baseline from a quantitative bacteriology culture of a pretreatment clean-catch midstream urine specimen. For inclusion into the micro-ITT NTF-S Population, all baseline qualifying uropathogen(s) must also be susceptible to nitrofurantoin. Qualifying uropathogen susceptibilities will be monitored instream to ensure sufficient and balanced enrollment of participants with uropathogens resistant to specific microbiological classes. Please refer to the RAP for specific details.

The algorithm for determining qualifying uropathogens based on microbiology laboratory quantitative culture results is provided in Figure 2, with additional algorithm details provided in the RAP.

Figure 2 Baseline Algorithm for Determining Qualifying Uropathogens



CFU=colony-forming units.

Note: Only the following uropathogen species/groups will be considered for inclusion in the micro-ITT and other microbiological populations: Gram-negative bacilli (e.g., *E. coli, K. pneumoniae*, *P. mirabilis*), *S. saprophyticus*, and *Enterococcus* spp. Analysis details for the other uropathogens and uropathogen groups will be described in the RAP, as applicable.

#### References

McCarter YS, Burd EM, Hall GS, Zervos M. Cumitech 2C, Laboratory diagnosis of urinary tract infections. Coordinating ed., Sharp SE. Washington, DC; ASM Press; 2009.1-26.

Chan WW. Chapter 3.12: Urine cultures. In: Leber AL, editor. Clinical microbiology procedures handbook, 4<sup>th</sup> ed. Vol 1-3. Washington, DC; ASM Press; 2016.

## 10.5. Appendix 5: COVID-19 Protocol Information

#### 10.5.1. Overall Rationale for this Appendix

The COVID-19 pandemic may impact the conduct of clinical studies. Challenges may arise from quarantines, site closures, travel limitations, interruptions to the supply chain for the investigational product or other considerations if site personnel or study participants become infected with COVID-19. These challenges may lead to difficulties in meeting protocol-specified procedures.

This appendix outlines measures that may be applicable for any study site impacted by the COVID-19 pandemic. The purpose of the appendix is to provide information on the measures to be taken to protect participants' safety, welfare and rights, and promote data integrity. These measures are expected to be temporary and study sites will be notified of any change to these allowances as the COVID-19 pandemic evolves.

## 10.5.2. Study Procedures During the COVID-19 Pandemic

During the special circumstances caused by the current COVID-19 pandemic, sites should consider specific public health guidance, the impact of any travel restrictions implemented by local/regional health authorities and local institutions, and individual benefit/risk when making enrollment and treatment decisions for study participants.

Every effort should be made to adhere to protocol-specified assessments for participants on study treatment, including follow-up assessments; however, when not possible, for the duration of these special circumstances, the following measures may be implemented:

- Only where applicable country and local regulations and infrastructure allow, home healthcare (home visits and telemedicine visits) may be performed at the discretion of the investigator and following the participant signing of an informed consent/assent form specific for home healthcare. Specific details will be described in the Study Reference Manual. The participant should be informed of the home healthcare plan and any potential risks associated with home visits and telemedicine. The participant must sign an informed consent form specific to home healthcare.
- For all study visits, to minimize the amount of time that participants spend at the clinic, eConsent may be utilized and remote collection of study-related data may be obtained as described in the Study Reference Manual. Thus, some visit data may be collected through a combination of telemedicine and on-site visits. Collection of information via telemedicine will be performed only where local regulations permit.
- Clinical investigators should document in site/participant/source files how
  restrictions related to COVID-19 led to changes in study conduct, the duration of
  those changes, and indicate which trial participants were impacted and how those
  trial participants were impacted (as per the current local COVID-19 related
  regulatory guidance).
- Missing protocol-required data/visits due to COVID-19 should be noted in site/participant/source files and recorded as a COVID-19 protocol deviation.

#### CONFIDENTIAL

TMF-13817737

## Specifically for data management and monitoring the following will apply:

- If on-site monitoring is no longer permitted, GSK/PPD will consider remote Source Data Verification/Source Document Review (SDV/SDR) where permitted by the clinical site/institution. Remote SDV/SDR will be proposed to study sites to meet a participant and/or critical quality need, e.g., to assess participant safety or to ensure data integrity. In case of remote SDV/SDR, GSK/PPD will work with the site to ensure participant privacy.
- eCRF/CRF Final or Interim Sign-Off Process: The principal investigator is responsible for ensuring that the data within the eCRF casebook and any other data sources utilized during the study for each study participant is complete and consistent with source documents throughout the study (ICH GCP 4.9.1 4.9.2). The principal investigator may sign/re-sign the eCRF from any computer/location by accessing the validated system using his/her unique eCRF log-in credentials. The principal investigator may delegate this activity to another medically qualified and trained subinvestigator and this must be documented on the Delegation of Responsibilities Log. It is recommended that the principal investigator identifies a subinvestigator as a back-up for eCRF signatures and that appropriate training on the protocol and eCRF requirements is provided and documented.
- Essential Document Sign-Off Process: If an investigator is unable to print and sign essential documents such as Protocol/Amendment signature page then e-mail approval can be accepted by replying to the relevant e-mail that is sent by GSK/PPD.

# 10.6. Appendix 6: Clinical Signs and Symptoms Score for Acute Cystitis

212390

Clinical signs and symptoms of acute cystitis will be recorded as follows:

| | None | Mild | Moderate | Severe |
|---|---|---|---|---|
| Clinical Signs | | Symptom is easily tolerated, causing minimal discomfort and not interfering with everyday activities | Symptom is<br>sufficiently<br>discomforting to<br>interfere with<br>normal everyday<br>activities | Symptom prevents normal everyday activities |
| and Symptoms | SCORE 0 | SCORE 1 | SCORE 2 | SCORE 3 |
| Dysuria | | | | |
| Frequency | | | | |
| Urgency | | | | |
| Lower abdominal or suprapubic pain | | | | |







TMF-13817737 212390

#### 10.8. **Appendix 8: Clinical Laboratory Tests**

- The tests detailed in Table 15 will be performed by the central laboratory.
- Local laboratory results are only required in the event that the central laboratory results are not available in time for a response evaluation. If a local sample is required, it is important that the sample for central analysis is obtained at the same time.
- Protocol-specific requirements for inclusion or exclusion of participants are detailed in Section 5 of the protocol.
- Additional tests may be performed at any time during the study as determined necessary by the investigator or required by local regulations.

## **Pregnancy Testing**

- Refer to Section 5.1 Inclusion Criteria for screening pregnancy criteria.
- Women of childbearing potential (WOCBP) should only be included after a confirmed menstrual period and a negative urine pregnancy test.
- Pregnancy testing will be performed at Baseline (Day 1) before study treatment administration. The urine pregnancy test at Baseline will determine study contraception and abstinence requirements as follows:
  - Pregnancy testing at Baseline (Day 1) should be performed using the urine test kit provided to the study site (FIRST RESPONSE Early Result Pregnancy Test with a high sensitivity of ≤6.3 mIU/mL). Participants with a negative urine pregnancy test result from this test kit may be included in the study with no pretreatment contraception or abstinence requirements. Women of childbearing protentional are not required to be using contraception or to have practiced abstinence within 14 days prior to study entry if the high sensitivity urine pregnancy test results are negative at Baseline (Day 1).

**Note:** ONLY if the study-specific pregnancy kit provided to the study site is unavailable, a standard urine pregnancy test with a sensitivity of 25 mIU/mL may be used as an exception. A participant with a negative urine pregnancy test result from the standard test may be included in the study only if the participant has used a highly effective contraception method as described in Section 10.2.2 or has practiced abstinence from penile/vaginal intercourse for at least 14 days before receiving study treatment.

After Dose 4 and before Dose 8, an additional pregnancy test using the urine test kit provided to the study site (FIRST RESPONSE Early Result Pregnancy Test with a sensitivity of ≤6.3 mIU/mL) is required to be performed for WOCBP who have not used a highly effective contraception method (in Section 10.2.2) or have not practiced abstinence from penile/vaginal intercourse for at least 14 days prior to the first dose of study treatment. It is preferable for this pregnancy test to be performed at the study site; however, for participants for whom this is not possible, the urine

## TMF-13817737 CONFIDENTIAL

pregnancy kit will be provided to the participant to perform as an outpatient during the defined window. For any participant with a positive pregnancy test result, study treatment must be immediately discontinued.

212390

- A pregnancy test will also be performed at the Test-of-Cure (Day 10 to 13) Visit, 5 to 8 days after the last dose of study treatment.
- Pregnancy testing will be performed whenever a menstrual cycle is missed or when pregnancy is otherwise suspected.
- Additional serum or urine pregnancy tests may be performed, as determined necessary by the investigator or required by local regulation, to establish the absence of pregnancy at any time during the subject's participation in the study.

Table 15 Protocol-Required Safety Laboratory Assessments

| Laboratory<br>Assessments | Parameters | | | | | |
|---|---|---|---|---|---|---|
| Hematology | Platelet count RBC count Hemoglobin Hematocrit | | RBC Indices:<br>MCV<br>MCH | | WBC Count With Differential: Neutrophils Lymphocytes Monocytes Eosinophils Basophils | |
| Clinical<br>Chemistry <sup>a</sup> | Blood urea nitrogen | | ssium | AST/SGOT | | Total and direct bilirubin |
| | Creatinine Glucose nonfasting Chloride | Sodium Calcium Magnesium | | ALT/SGPT Alkaline phosphatase Phosphorus | ! | Total protein Albumin |
| Routine<br>Urinalysis | <ul> <li>Specific gravity</li> <li>pH, glucose, protein, blood, ketones, nitrite, and leukocyte esterase by dipstick</li> <li>Microscopic examination (if blood or protein is abnormal)</li> </ul> | | | | | |
| Other<br>Screening<br>Tests | Serum or urine alcohol and drug screen (to include at minimum: amphetamines, barbiturates, cocaine, opiates, cannabinoids, and benzodiazepines) | | | | | ninimum: |
| | Urine hCG pregnancy test (as needed for women of childbearing potential) <sup>b</sup> Note: See text earlier in this section for pregnancy test sensitivity requirements and additional pregnancy testing details. | | | | | |
| | Serology (HBsAg, hepatitis C virus antibody, and HIV). If serology testing was performed within 3 months prior to the first dose of study treatment and results were positive, testing at Baseline is not required. If testing was performed within 3 months and any result was negative, testing at Baseline is required. **Transferance: AST-percentate aministransferance: HBsAg-hepatitis B surface antigen: hCG-humperstansferance: AST-percentate aministransferance: HBsAg-hepatitis B surface antigen: hCG-humperstansferance: hC | | | | | study treatment<br>uired. If testing<br>ative, testing at |

ALT=alanine aminotransferase; AST=aspartate aminotransferase; HBsAg=hepatitis B surface antigen; hCG=human chorionic gonadotropin; HIV=human immunodeficiency virus; MCH=mean corpuscular hemoglobin; MCV=mean corpuscular volume; RBC=red blood cell; SGOT=serum glutamic-oxaloacetic transaminase; SGPT=serum glutamic-pyruvic transaminase; WBC=while blood cell.

- a. Details of liver chemistry stopping criteria and required actions and follow-up assessments after liver stopping or monitoring event are given in Section 7.1 and Appendix 10. All events of ALT ≥3 × upper limit of normal (ULN) and bilirubin ≥2 × ULN (>35% direct bilirubin) or ALT ≥3 × ULN and international normalized ratio (INR) >1.5, if INR measured, which may indicate severe liver injury (possible Hy's Law), must be reported as a serious adverse event.
- b. Local urine testing will be standard for the protocol unless serum testing is required by local regulation or the Institutional Review Board/Independent Ethics Committee.

Laboratory results that could unblind the study will not be reported to study sites or other blinded personnel until the study has been unblinded.

# 10.9. Appendix 9: Additional Guidance on Permitted and Prohibited Medications and Crediblemeds.org

For quick reference, a list of some common concomitant medications that are permitted for participants to take during the study for nausea, vomiting, pain, diarrhea, etc. per investigator discretion is provided below. A list of some of the commonly used medications that are prohibited is also provided in this appendix. Lastly, a topline overview of how to use crediblemeds.org is also provided.

A further detailed list of medications will be provided in the Study Reference Manual.

#### **List of Concomitant Medications Permitted During the Study:**

| Generic Name <sup>a</sup> | Common Therapeutic Use(s) |
|---|---|
| Acetylsalicylic acid | Only allowed for the prevention of cardiovascular disease events at a low dose of ≤100 mg/day |
| Dolasetron | Nausea, vomiting |
| Granisetron | Nausea, vomiting |
| Metoclopramide | Nausea, vomiting |
| Palonosetron | Nausea, vomiting |
| Promethazine | Nausea, vomiting |
| Acetaminophen or paracetamol | Pain, fever |
| Tramadol | Pain |
| Hydrocodone ER | Pain, severe |
| Loperamide | Diarrhea |
| Cetirizine | Antihistamine (H <sub>1</sub> ) |
| Ebastine | Antihistamine (H <sub>1</sub> ) |
| Fexofenadine | Antihistamine (H <sub>1</sub> ) |
| Loratadine | Antihistamine (H <sub>1</sub> ) |
| Clindamycin | Antibiotic – topical, nonsystemic only |
| Neomycin | Antibiotic – topical, nonsystemic only |
| Polymyxin | Antibiotic – topical, nonsystemic only |
| Clotrimazole | Antifungal – topical, nonsystemic only |
| Tolnaftate | Antifungal – topical, nonsystemic only |
| Ketoconazole | Antifungal – topical, nonsystemic only |

ER=extended release.

Note: See also Section 6.5.1 for other permitted medications.

a. Check within each local country to assess if other generic names apply.

## **List of Prohibited Concomitant Medications:**

| Generic Name or Category <sup>a</sup> | Common Therapeutic Use(s) |
|---|---|
| Ondansetron | Nausea, vomiting |
| Acetylsalicylic acid (doses >100 mg/day) | Pain, other |
| Celecoxib | Pain |
| Diclofenac | Pain |
| Diflunisal | Pain |
| Etodolac | Pain |
| Ibuprofen | Pain, fever |
| Indomethacin | Pain |
| Ketoprofen | Pain |
| Ketorolac | Pain |
| Nabumetone | Pain |
| Naproxen | Pain |
| Oxaprozin | Pain |
| Phenazopyridine | Pain (urinary tract) |
| Piroxicam | Pain |
| Rofecoxib | Pain |
| Salsalate | Pain |
| Sulindac | Pain |
| Tolmetin | Pain |
| Valdecoxib | Pain |
| Other investigational products | Various |
| Systemic antibiotics (e.g., ciprofloxacin, amoxicillin/clavulanate, cephalexin, doxycycline) | Antibiotic – all systemic |
| Systemic antifungals (e.g., itraconazole, fluconazole, terbinafine) | Antifungal – <i>all systemic</i> |
| Prednisolone or equivalent (refer to Section 6.5.2 for details) | Immunosuppressive therapy |
| Strong CYP3A4 inhibitors and strong CYP3A4 inducers | See Study Reference Manual |
| St John's wort | Herbal, various |
| Uva ursi | Herbal, various |
| D-mannose | Nutritional supplement, various |
| Cranberry supplements | Nutritional supplement, various |
| Probenecid | Uric acid reducer |
| Sulfinpyrazone | Uric acid reducer |
| Magnesium trisilicate | Antacid (common ingredient) |
| Succinylcholine and other nondepolarizing paralytic agents | Muscle relaxation, muscle paralysis |

CYP3A4=cytochrome P450 enzyme 3A4; NSAIDS=nonsteroidal anti-inflammatory medications.

Note: See also Section 6.5.2 for other prohibited medications and details for the when these medications are prohibited. All NSAIDS are prohibited; this list may not be an exhaustive list of all NSAIDS available globally.

a. Check within each local country to assess if other generic names apply.

#### **Crediblemeds.org Instructions**

Instructions for accessing www.crediblemeds.org and searching for an exclusionary drug due to its "Known Risk of Torsades de Pointes (TdP)" category are summarized below.

To access www.crediblemeds.org, copy and paste this link into the internet search bar: https://www.crediblemeds.org/

On the main home page, there are 2 search options available. Choose the first option to search for 1 drug at a time, which does not require registration.



Choosing that option brings you to a screen that allows for you to enter a generic or brand drug name and choose Search. If it has a Known Risk of TdP (i.e., is a prohibited exclusionary medication), it will show a red triangle with an exclamation point as shown here:



Always check the www.crediblemeds.org website for the most up-to-date information on drugs with a Known Risk of TdP for participant safety.

## 10.10. Appendix 10: Liver Safety: Required Actions and Follow-up Assessments

Phase III liver chemistry stopping and increased monitoring criteria have been designed to assure participant safety and evaluate liver event etiology.

Phase III liver chemistry stopping criteria and required follow-up assessments

| Liver Chemistry Stopping Criteria | | | | |
|---|---|---|---|---|
| ALT-absolute | ALT ≥8xULN | | | |
| ALT Increase | ALT ≥5xULN but <8 x ULN persists for ≥2 weeks | | | |
| | ALT ≥3xULN but <5 x ULN persists for ≥4 weeks | | | |
| Bilirubin <sup>a,b</sup> | ALT ≥3xULN and bilirubin ≥2 x ULN (>35% direct bilirubin) | | | |
| INRb | ALT ≥3xULN and INR>1.5 | | | |
| Cannot<br>Monitor | ALT $\geq$ 5xULN but <8 x ULN <b>and</b> cannot be monitored weekly for $\geq$ 2 weeks ALT $\geq$ 3xULN but <5 x ULN <b>and</b> cannot be monitored weekly for $\geq$ 4 weeks | | | |
| Symptomatic <sup>c</sup> | ALT ≥3 x ULN associated with symptoms (new or worsening) believed to be related to liver injury or hypersensitivity | | | |
| | Required Actions and Follow-up Assessments | | | |
| Actions | | Follow-up Assessments | | |
| <ul> <li>Immediately</li> </ul> | discontinue study treatment | Viral hepatitis serology <sup>d</sup> | | |
| <ul> <li>Report the event to GSK/PPD within 24 hours</li> <li>Complete the liver event eCRF and complete an SAE data collection tool if the event also meets the criteria for an SAE<sup>b</sup></li> </ul> | | Only in those with underlying chronic Hepatitis B at study entry (identified by positive hepatitis B surface antigen) and quantitative hepatitis B DNA | | |
| <ul> <li>Perform liver event follow-up assessments</li> <li>Monitor the participant until liver chemistries resolve, stabilize, or return to within baseline (see MONITORING below)</li> </ul> | | <ul> <li>Obtain INR and recheck with each liver<br/>chemistry assessment until the<br/>transaminases values show downward<br/>trend</li> <li>Obtain blood sample for pharmacokinetic</li> </ul> | | |
| | | | Do not restart/rechallenge participant with study treatment | (PK) analysis, within 24 hours after last dose |
| If restart/rechallenge not allowed or not granted, permanently discontinue study treatment and continue participant in the | | Serum creatine phosphokinase and lactate dehydrogenase | | |

study for any protocol-specified follow-up assessments

#### MONITORING:

#### For bilirubin or INR criteria:

- Repeat liver chemistries (include ALT, AST, alkaline phosphatase, bilirubin, and INR) and perform liver event follow-up assessments within 24 hours
- Monitor participant twice weekly until liver chemistries resolve, stabilize, or return to within baseline
- A specialist or hepatology consultation is recommended

#### For All other criteria:

- Repeat liver chemistries (include ALT, AST, alkaline phosphatase, bilirubin, and INR) and perform liver event follow-up assessments within 24 to 72 hours
- Monitor participant weekly until liver chemistries resolve, stabilize, or return to within baseline

- Fractionate bilirubin, if total bilirubin
   ≥2 x ULN
- Obtain complete blood count with differential to assess eosinophilia
- Record the appearance or worsening of clinical symptoms of liver injury, or hypersensitivity, on the AE report form
- Record use of concomitant medications on the concomitant medications report form including acetaminophen, herbal remedies, other over-the-counter medications.
- Record alcohol use on the liver event alcohol intake eCRF page

#### For bilirubin or INR criteria:

- Antinuclear antibody, antismooth muscle antibody, type 1 antiliver kidney microsomal antibodies, and quantitative total IgG or gamma globulins.
- Serum acetaminophen adduct HPLC assay (quantifies potential acetaminophen contribution to liver injury in participants with definite or likely acetaminophen use in the preceding week [James, 2009]). NOTE: not required in China
- Liver imaging (ultrasound, magnetic resonance, or computed tomography) and/or liver biopsy to evaluate liver disease; complete liver imaging and/or liver biopsy eCRFs.

AE=adverse event; ALT=alanine aminotransferase; AST=aspartate aminotransferase; eCRF=electronic case report form; GSK=GlaxoSmithKline; HPLC=high-performance liquid chromatography; IgG=immunoglobulin G; IgM=immunoglobulin M; INR=international normalized ratio; PCR=polymerase chain reaction; PK=pharmacokinetic; SAE=serious adverse event; ULN=upper limit of normal.

- a. Serum bilirubin fractionation should be performed if testing is available. If serum bilirubin fractionation is not immediately available, discontinue study treatment for that participant if ALT ≥3 x ULN and bilirubin ≥2 x ULN. Additionally, if serum bilirubin fractionation testing is unavailable, record presence of detectable urinary bilirubin on dipstick, indicating direct bilirubin elevations and suggesting liver injury.
- b. All events of ALT ≥3 x ULN and bilirubin ≥2 x ULN (>35% direct bilirubin) or ALT ≥3 x ULN and INR >1.5 which may indicate severe liver injury (possible 'Hy's Law'), must be reported as an SAE (excluding studies of hepatic impairment or cirrhosis); the INR threshold value stated will not apply to participants receiving anticoagulants.
- c. New or worsening symptoms believed to be related to liver injury (such as fatigue, nausea, vomiting, right upper quadrant pain or tenderness, or jaundice) or believed to be related to hypersensitivity (such as fever, rash or eosinophilia).
- d. Includes: hepatitis A IgM antibody; hepatitis B surface antigen and hepatitis B core antibody; hepatitis C RNA; cytomegalovirus IgM antibody; Epstein-Barr viral capsid antigen IgM antibody (or if unavailable, heterophile antibody or monospot testing); and hepatitis E IgM antibody. In those with underlying chronic hepatitis B at study entry (identified by positive hepatitis B surface antigen) quantitative hepatitis B DNA and hepatitis delta antibody. If hepatitis delta antibody assay cannot be performed, it can be replaced with a PCR of hepatitis D RNA virus (where needed) [Le Gal, 2005].
- e. PK sample may not be required for participants known to be receiving placebo or noncomparator treatments. Record the date/time of the PK blood sample draw and the date/time of the last dose of study treatment prior to the PK blood sample draw in the eCRF. If the date or time of the last dose is unclear, provide the participant's best approximation. If the date/time of the last dose cannot be approximated OR a PK sample cannot be collected in the time period indicated above, do not obtain a PK sample. Instructions for sample handling and shipping are in the Study Reference Manual.

#### Phase III liver chemistry increased monitoring criteria with continued therapy

#### Liver Chemistry Increased Monitoring Criteria – Liver Monitoring Event Criteria Actions Notify the GSK/PPD medical monitor within **24 hours** of learning of the abnormality to discuss ALT $\geq$ 5 x ULN and <8 x ULN and participant safety. bilirubin <2 x ULN without symptoms believed to be related to liver injury or Participant can continue study treatment. hypersensitivity, and who can be Participant must return weekly for repeat liver monitored weekly for 2 weeks. chemistries (ALT, AST, alkaline phosphatase, OR bilirubin) until they resolve, stabilize or return to within baseline. ALT $\geq$ 3 x ULN and <5 x ULN and bilirubin <2 x ULN without symptoms If at any time participant meets the liver chemistry believed to be related to liver injury or stopping criteria, proceed as described above. hypersensitivity, and who can be If ALT decreases from ALT ≥5 x ULN and monitored weekly for 4 weeks. $<8 \times ULN$ to $\geq 3 \times ULN$ but $<5 \times ULN$ , continue to monitor liver chemistries weekly. If, after 4 weeks of monitoring, ALT <3 x ULN and bilirubin <2 x ULN, monitor participants twice monthly until liver chemistries normalize or return to within baseline.

ALT=alanine aminotransferase; AST=aspartate aminotransferase; GSK=GlaxoSmithKline; ULN=upper limit of normal.

#### References

James LP, Letzig L, Simpson PM, Capparelli E, Roberts DW, Hinson JA, et al. Pharmacokinetics of acetaminophen-adduct in adults with acetaminophen overdose and acute liver failure. Drug Metab Dispos 2009; 37:1779-1784.

Le Gal F, Gordien E, Affolabi D, Hanslik T, Alloui C, Dény P, et al. Quantification of hepatitis delta virus RNA in serum by consensus real-time PCR indicates different

## TMF-13817737 **CONFIDENTIAL** 212390

patterns of virological response to interferon therapy in chronically infected patients. J Clin Microbiol. 2005;43(5):2363-2369.

## 10.11. Appendix 11: Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting

#### 10.11.1. Definition of Adverse Event

#### **Adverse Event Definition**

- An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment.
- NOTE: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment.

#### **Events Meeting the AE Definition**

- Any abnormal laboratory test results (hematology, clinical chemistry, or urinalysis) or other safety assessments (e.g., electrocardiograms, radiological scans, vital signs measurements), including those that worsen from baseline, considered clinically significant in the medical and scientific judgment of the investigator (i.e., not related to progression of underlying disease).
- Exacerbation of a chronic or intermittent pre-existing condition including either an increase in frequency and/or intensity of the condition.
- New conditions detected or diagnosed after study treatment administration even though it may have been present before the start of the study.
- Signs, symptoms, or the clinical sequelae of a suspected drug-drug interaction.
- Signs, symptoms, or the clinical sequelae of a suspected overdose of either study treatment or a concomitant medication. Overdose per se will not be reported as an AE/serious AE (SAE) unless it is an intentional overdose taken with possible suicidal/self-harming intent. Such overdoses should be reported regardless of sequelae.
- "Lack of efficacy" or "failure of expected pharmacological action" per se will not be reported as an AE or SAE. Such instances will be captured in the efficacy assessments. However, the signs, symptoms, and/or clinical sequelae resulting from lack of efficacy will be reported as AE or SAE if they fulfill the definition of an AE or SAE.

#### **Events NOT Meeting the AE Definition**

- Any clinically significant abnormal laboratory findings or other abnormal safety
  assessments which are associated with the underlying disease, unless judged by
  the investigator to be more severe than expected for the participant's condition.
- The disease/disorder being studied or expected progression, signs, or symptoms of the disease/disorder being studied, unless more severe than expected for the participant's condition.
- Medical or surgical procedure (e.g., endoscopy, appendectomy): the condition that leads to the procedure is the AE.
- Situations in which an untoward medical occurrence did not occur (social and/or convenience admission to a hospital).
- Anticipated day-to-day fluctuations of pre-existing disease(s) or condition(s) present or detected at the start of the study that do not worsen.

#### 10.11.2. Definition of SAE

If an event is not an AE per definition above, then it cannot be an SAE even if serious conditions are met (e.g., hospitalization for signs/symptoms of the disease under study, death due to progression of disease).

#### An SAE is defined as any untoward medical occurrence that, at any dose:

- Results in death.
- o Is life-threatening

The term "life-threatening" in the definition of "serious" refers to an event in which the participant was at risk of death at the time of the event. It does not refer to an event, which hypothetically might have caused death, if it were more severe.

#### Requires inpatient hospitalization or prolongation of existing hospitalization

- In general, hospitalization signifies that the participant has been detained (usually involving at least an overnight stay) at the hospital or emergency ward for observation and/or treatment that would not have been appropriate in the physician's office or outpatient setting. Complications that occur during hospitalization are AE. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred or was necessary, the AE should be considered serious.
- Hospitalization for elective treatment of a pre-existing condition that did not worsen from baseline is not considered an AE.

#### Results in persistent or significant disability/incapacity

- The term disability means a substantial disruption of a person's ability to conduct normal life functions.
- This definition is not intended to include experiences of relatively minor medical significance such as uncomplicated headache, nausea, vomiting, diarrhea, influenza, and accidental trauma (e.g., sprained ankle) which may interfere with or prevent everyday life functions but do not constitute a substantial disruption.

#### Is a congenital anomaly/birth defect

#### Other situations:

- Medical or scientific judgment should be exercised in deciding whether SAE reporting is appropriate in other situations such as important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical treatment to prevent one of the other outcomes listed in the above definition. These events should usually be considered serious.
- Examples of such events include invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization, or development of drug dependency or drug abuse.

## 10.11.3. Cardiovascular Adverse Events of Special Interest and Cases of Clostridium Difficile

Investigators will be required to fill out the specific event page of the electronic case report form (eCRF) for the following cardiovascular AEs and SAEs, and for cases of *Clostridium difficile*:

#### **Cardiovascular Events:**

- Myocardial infarction/unstable angina
- Congestive heart failure
- Arrhythmias
- Valvulopathy
- Pulmonary hypertension
- Cerebrovascular events/stroke and transient ischemic attack
- Peripheral arterial thromboembolism
- Deep venous thrombosis/pulmonary embolism
- Revascularization

#### 10.11.4. Recording and Follow-Up of AE and SAE

#### AE and SAE Recording

- When an AE/SAE occurs, it is the responsibility of the investigator to review all documentation (e.g., hospital progress notes, laboratory, and diagnostics reports) related to the event.
- The investigator will then record all relevant AE/SAE information in the eCRF.
- It is **not** acceptable for the investigator to send photocopies of the participant's medical records to GlaxoSmithKline (GSK)/PPD in lieu of completion of the GSK/PPD AE/SAE eCRF page.
- There may be instances when copies of medical records for certain cases are requested by GSK. In this case, all participant identifiers, with the exception of the participant number, will be redacted on the copies of the medical records before submission to GSK.
- The investigator will attempt to establish a diagnosis of the event based on signs, symptoms, and/or other clinical information. Whenever possible, the diagnosis (not the individual signs/symptoms) will be documented as the AE/SAE.

#### **Assessment of Intensity**

• The severity of AEs and SAEs will be determined by the investigator according to the US National Institute of Allergy and Infectious Diseases Division of Microbiology and Infectious Diseases criteria for adult toxicity assessment [DMID, 2007a], with the exception of serum creatinine adolescent laboratory data, which be assessed using pediatric toxicity criteria [DMID, 2007b] (Appendix 13).

An event is defined as "serious" when it meets at least 1 of the predefined outcomes as described in the definition of an SAE, NOT when it is rated as severe.

#### Assessment of Causality

- The investigator is obligated to assess the relationship between study treatment and each occurrence of each AE/SAE.
- A "reasonable possibility" of a relationship conveys that there are facts, evidence, and/or arguments to suggest a causal relationship, rather than a relationship cannot be ruled out.
- The investigator will use clinical judgment to determine the relationship.
- Alternative causes, such as underlying disease(s), concomitant therapy, and other risk factors, as well as the temporal relationship of the event to study treatment administration will be considered and investigated.
- The investigator will also consult the investigator's brochure and/or product information, for marketed products, in his/her assessment.
- For each AE/SAE, the investigator <u>must</u> document in the medical notes that he/she has reviewed the AE/SAE and has provided an assessment of causality.

- There may be situations in which an SAE has occurred, and the investigator has minimal information to include in the initial report to GSK/PPD. However, it is very important that the investigator always make an assessment of causality for every event before the initial transmission of the SAE data to GSK/PPD.
- The investigator may change his/her opinion of causality in light of follow-up information and send an SAE follow-up report with the updated causality assessment.
- The causality assessment is one of the criteria used when determining regulatory reporting requirements.

#### Follow-up of AE and SAE

- The investigator is obligated to perform or arrange for the conduct of supplemental measurements and/or evaluations as medically indicated or as requested by GSK to elucidate the nature and/or causality of the AE or SAE as fully as possible. This may include additional laboratory tests or investigations, histopathological examinations, or consultation with other health care professionals.
- If a participant dies during participation in the study or during a recognized follow-up period, the investigator will provide GSK with a copy of any postmortem findings including histopathology.
- New or updated information will be recorded in the originally completed eCRF.
- The investigator will submit any updated SAE data to GSK/PPD within 24 hours of receipt of the information.

#### 10.11.5. Reporting of SAE to GSK/PPD

#### SAE Reporting to GSK/PPD via Electronic Data Collection Tool

- The primary mechanism for reporting SAE to GSK/PPD will be the electronic data collection tool.
- The site will enter the SAE data into the electronic system as soon as it becomes available.
- The investigator or medically qualified subinvestigator must show evidence within the eCRF (e.g., check review box, signature, etc.) of review and verification of the relationship of each SAE to study treatment/study participation (causality) within 72 hours of SAE entry into the eCRF.
- After the study is completed at a given study site, the electronic data collection tool will be taken off-line to prevent the entry of new data or changes to existing data.
- If a study site receives a report of a new SAE from a study participant or receives updated data on a previously reported SAE after the electronic data collection tool has been taken off-line, then the site can report this information to the medical monitor or SAE coordinator by telephone.

• Contacts for SAE reporting can be found in the Study Reference Manual.

#### 10.12. **Appendix 12: Genetics**

#### USE/ANALYSIS OF DNA

- Genetic variation may impact a participant's response to study treatment, susceptibility, severity and progression of disease. Variable response to study treatment may be due to genetic determinants that impact drug absorption, distribution, metabolism, and excretion; mechanism of action of the drug; disease etiology; and/or molecular subtype of the disease being treated. Therefore, where local regulations and institutional review board/independent ethics committee allow, a blood sample will be collected for DNA analysis.
- DNA samples will be used for research related to gepotidacin or uncomplicated urinary tract infections and related diseases. They may also be used to develop tests/assays (including diagnostic tests) related to gepotidacin and uncomplicated urinary tract infections. Genetic research may consist of the analysis of one or more candidate genes or the analysis of genetic markers throughout the genome [or analysis of the entire genome] (as appropriate).
- Additional analyses of DNA samples may be conducted if it is hypothesized that this may help further understand the clinical data.
- The samples may be analyzed as part of a multi-study assessment of genetic factors involved in the response to gepotidacin or study treatments of this class. The results of genetic analyses may be reported in the clinical study report or in a separate study summary.
- The sponsor will store the DNA samples in a secure storage space with adequate measures to protect confidentiality.
- The samples will be retained while research on gepotidacin (or study treatments of this class) or uncomplicated urinary tract infections continues but no longer than 15 years after the last participant last visit or other period as per local requirements.

# 10.13. Appendix 13: Division of Microbiology and Infectious Diseases Adult Toxicity Tables for Adverse Event Assessment

**ESTIMATING SEVERITY GRADE:** For abnormalities NOT found elsewhere in the Toxicity Tables, use the scale below to estimate grade of severity:

| GRADE 1 | Mild | Transient or mild discomfort (<48 hours); no medical intervention/therapy required |
|---|---|---|
| GRADE 2 | Moderate | Mild to moderate limitation in activity – some assistance may be needed; no or minimal medical intervention/therapy required |
| GRADE 3 | Severe | Marked limitation in activity, some assistance usually required; medical intervention/therapy required, hospitalizations possible |
| GRADE 4 | Life-threatening | Extreme limitation in activity, significant assistance required; significant medical intervention/therapy required, hospitalization or hospice care probable |

**SERIOUS OR LIFE-THREATENING AEs:** ANY clinical event deemed by the investigator to be serious or life-threatening should be considered a Grade 4 event. Clinical events considered to be serious or life-threatening include, but are not limited to: seizures, coma, tetany, diabetic ketoacidosis, disseminated intravascular coagulation, diffuse petechiae, paralysis, acute psychosis, and severe depression.

#### **COMMENTS REGARDING THE USE OF THESE TABLES**

- Standardized and commonly used toxicity tables (Division of AIDS, National Cancer Institute's Common Toxicity Criteria, and World Health Organization) have been adapted for use by the Division of Microbiology and Infectious Diseases (DAIDS) and modified to better meet the needs of participants in Division of Microbiology and Infectious Diseases (DMID) trials.
- For parameters not included in the following Toxicity Tables, study sites should refer to the "Guide for Estimating Severity Grade" located above.
- Criteria are generally grouped by body system.

Some protocols may have additional protocol-specific grading criteria, which will supersede the use of these tables for specified criteria.

**Note**: Adult DMID toxicity criteria will be applied for all laboratory parameters, with the exception of serum creatinine adolescent laboratory data, which will be assessed using pediatric DMID toxicity criteria. The DMID pediatric toxicity table may be accessed at https://www.niaid.nih.gov/sites/default/files/dmidpedtox.pdf.

| HEMATOLOGY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hemoglobin | 9.5 to 10.5 gm/dL | 8.0 to 9.4 gm/dL | 6.5 to 7.9 gm/dL | <6.5 gm/dL |
| Absolute Neutrophil Count | 1000 to 1500 /mm <sup>3</sup> | 750 to 999 /mm <sup>3</sup> | 500 to 749 /mm <sup>3</sup> | <500 /mm <sup>3</sup> |
| Platelets | 75,000 to 99,999 /mm <sup>3</sup> | 50,000 to 74,999 /mm <sup>3</sup> | 20,000 to 49,999 /mm <sup>3</sup> | <20,000 /mm <sup>3</sup> |
| White Blood Cells | 11,000 to 13,000 /mm <sup>3</sup> | 13,000 to 15,000 /mm <sup>3</sup> | 15,000 to 30,000 /mm <sup>3</sup> | >30,000 or <1000 /mm <sup>3</sup> |
| % Polymorphonuclear Leukocytes + Band Cells | >80% | 90 to 95% | >95% | N/A |
| Abnormal Fibrinogen | Low: 100 to 200 mg/dL<br>High: 400 to 600 mg/dL | Low: <100 mg/dL<br>High: >600 mg/dL | Low: <50 mg/dL<br>High: N/A | Fibrinogen associated with gross bleeding or with disseminated coagulation |
| Fibrin Split Product | 20 to 40 mcg/mL | 41 to 50 mcg/mL | 51 to 60 mcg/dL | >60 mcg/dL |
| Prothrombin Time (PT) | 1.01 to 1.25 × ULN | 1.26 to 1.5 × ULN | 1.51 to 3.0 × ULN | >3 × ULN |
| Activated Partial Thromboplastin (APTT) | 1.01 to 1.66 × ULN | 1.67 to 2.33 × ULN | 2.34 to 3 × ULN | >3 × ULN |
| Methemoglobin | 5.0 to 9.9% | 10.0 to 14.9% | 15.0 to 19.9% | >20% |

N/A=not applicable; ULN=upper limit of normal.

| CHEMISTRIES | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hyponatremia | 130 to 135 mEq/L | 123 to 129 mEq/L | 116 to 122 mEq/L | <116 mEq/L or abnormal sodium with mental status changes or seizures |
| Hypernatremia | 146 to 150 mEq/L | 151 to 157 mEq/L | 158 to 165 mEq/L | >165 mEq/L or abnormal sodium with mental status changes or seizures |
| Hypokalemia | 3.0 to 3.4 mEq/L | 2.5 to 2.9 mEq/L | 2.0 to 2.4 mEq/L or intensive replacement therapy of hospitalization required | <2.0 mEq/L or abnormal potassium with paresis, ileus, or life-threatening arrhythmia |
| Hyperkalemia | 5.6 to 6.0 mEq/L | 6.1 to 6.5 mEq/L | 6.6 to 7.0 mEq/L | >7.0 mEq/L or abnormal potassium with life-threatening arrhythmia |
| Hypoglycemia | 55 to 64 mg/dL | 40 to 54 mg/dL | 30 to 39 mg/dL | <30 mg/dL or abnormal glucose with mental status changes or coma |
| Hyperglycemia<br>(nonfasting and no prior<br>diabetes) | 116 to 160 mg/dL | 161 to 250 mg/dL | 251 to 500 mg/dL | >500 mg/dL or abnormal glucose with ketoacidosis or seizures |
| Hypocalcemia (corrected for albumin) | 8.4 to 7.8 mg/dL | 7.7 to 7.0 mg/dL | 6.9 to 6.1 mg/dL | <6.1 mg/dL or abnormal calcium with life-threatening arrhythmia or tetany |
| Hypercalcemia (corrected for albumin) | 10.6 to 11.5 mg/dL | 11.6 to 12.5 mg/dL | 12.6 to 13.5 mg/dL | >13.5 mg/dL or abnormal calcium <i>with</i> life-threatening arrhythmia |
| Hypomagnesemia | 1.4 to 1.2 mEq/L | 1.1 to 0.9 mEq/L | 0.8 to 0.6 mEq/L | <0.6 mEq/L or abnormal magnesium with life-threatening arrhythmia |
| Hypophosphatemia | 2.0 to 2.4 mg/dL | 1.5 to 1.9 mg/dL or replacement Rx required | 1.0 to 1.4 mg/dL intensive therapy or hospitalization required | <1.0 mg/dL or abnormal phosphate with life-threatening arrhythmia |
| Hyperbilirubinemia (when accompanied by any increase in other liver function test) | 1.1 to <1.25 × ULN | 1.25 to <1.5 × ULN | 1.5 to 1.75 × ULN | >1.75 × ULN |
| Hyperbilirubinemia (when other liver function tests are in the normal range) | 1.1 to <1.5 × ULN | 1.5 to <2.0 × ULN | 2.0 to 3.0 × ULN | >3.0 × ULN |
| Blood urea nitrogen | 1.25 to 2.5 × ULN | 2.6 to 5 × ULN | 5.1 to 10 × ULN | >10 × ULN |
| Hyperuricemia (uric acid) | 7.5 to 10.0 mg/dL | 10.1 to 12.0 mg/dL | 12.1 to 15.0 mg/dL | >15.0 mg/dL |
| Creatinine | 1.1 to 1.5 × ULN | 1.6 to 3.0 × ULN | 3.1 to 6.0 × ULN | >6 × ULN or dialysis required |

Rx=therapy; ULN=upper limit of normal.

| ENZYMES | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Aspartate aminotransferase (AST) | 1.1 to <2.0 × ULN | 2.0 to <3.0 × ULN | 3.0 to 8.0 × ULN | >8.0 × ULN |
| Alanine aminotransferase (ALT) | 1.1 to <2.0 × ULN | 2.0 to <3.0 × ULN | 3.0 to 8.0 × ULN | >8.0 × ULN |
| Gamma to glutamyl transferase (GGT) | 1.1 to <2.0 × ULN | 2.0 to <3.0 × ULN | 3.0 to 8.0 × ULN | >8.0 × ULN |
| Alkaline Phosphatase | 1.1 to <2.0 × ULN | 2.0 to <3.0 × ULN | 3.0 to 8.0 × ULN | >8.0 × ULN |
| Amylase | 1.1 to 1.5 × ULN | 1.6 to 2.0 × ULN | 2.1 to 5.0 × ULN | >5.1 × ULN |
| Lipase | 1.1 to 1.5 × ULN | 1.6 to 2.0 × ULN | 2.1 to 5.0 × ULN | >5.1 × ULN |

212390

ULN=upper limit of normal.

| URINALYSIS | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Drotoinurio | 1+ or | 2 to 3+ or | 4+ or | Nephrotic syndrome or |
| Proteinuria | 200 mg to 1 gm loss/day | 1 to 2 gm loss/day | 2 to 3.5 gm loss/day | >3.5 gm loss/day |
| I la ma atronia | Microscopic only | Gross, no clots | Gross, with or without clots, | Obstructive or |
| Hematuria | <10 RBC/HPF | >10 RBC/HPF | or red blood cells casts | required transfusion |

HPF=high-power field; RBC=red blood cells.

| CARDIOVASCULAR | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Cardiac rhythm | N/A | Asymptomatic, transient signs, no Rx required | Recurrent/persistent; symptomatic Rx required | Unstable dysrhythmia;<br>hospitalization and treatment<br>required |
| Hypertension | Transient increase >20 mm/Hg; no treatment | Recurrent, chronic increase >20 mm/Hg; treatment required | Acute treatment required; outpatient treatment or hospitalization possible | End organ damage or hospitalization required |
| Hypotension | Transient orthostatic hypotension with heart rate increased by <20 beat/min or decreased by <10 mmHg systolic BP. No treatment required | Symptoms due to orthostatic<br>hypotension or BP decreased by<br><20 mmHg systolic; correctable<br>with oral fluid treatment | Requires IV fluids;<br>no hospitalization required | Mean arterial pressure <60 mmHg<br>or end organ damage or shock;<br>requires hospitalization and<br>vasopressor treatment |
| Pericarditis | Minimal effusion | Mild/moderate asymptomatic effusion, no treatment | Symptomatic effusion; pain; EKG changes | Tamponade; pericardiocentesis or surgery required |
| Hemorrhage, Blood Loss | Microscopic/occult | Mild, no transfusion | Gross blood loss;<br>1 to 2 units transfused | Massive blood loss; >3 units transfused |

BP=blood pressure; IV=intravenous; EKG=electrocardiogram; N/A=not applicable; Rx=therapy.

| RESPIRATORY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Cough | Transient; no treatment | Persistent cough; treatment responsive | Paroxysmal cough; uncontrolled with treatment | N/A |
| Bronchospasm, Acute | Transient; no treatment; FEV <sub>1</sub> 70 to 80% of peak flow | Requires treatment; normalizes with bronchodilator; FEV <sub>1</sub> 50 to 70% of peak flow | No normalization with bronchodilator; FEV <sub>1</sub> 25 to 50% of peak flow; or retractions present | Cyanosis: FEV <sub>1</sub> <25% of peak flow; or intubation necessary |
| Dyspnea | Dyspnea on exertion | Dyspnea with normal activity | Dyspnea at rest | Dyspnea requiring oxygen therapy |

FEV<sub>1</sub>=forced expiratory volume in 1 second; N/A=not applicable.

| GASTROINTESTINAL | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Nausea | Mild or transient; maintains reasonable intake | Moderate discomfort; intake decreased significantly; some activity limited | No significant intake; requires IV fluids | Hospitalization required |
| Vomiting | 1 episode in 24 hours | 2 to 5 episodes in 24 hours | >6 episodes in 24 hours or needing IV fluids | Physiologic consequences requiring hospitalization or requiring parenteral nutrition |
| Constipation | Requiring stool softener or dietary modification | Requiring laxatives | Obstipation requiring manual evacuation or enema | Obstruction or toxic megacolon |
| Diarrhea | Mild or transient; 3 to<br>4 loose stools/day or mild<br>diarrhea lasting <1 week | Moderate or persistent; 5 to 7 loose stools/day or diarrhea lasting >1 week | >7 loose stools/day or bloody diarrhea;<br>or orthostatic hypotension or electrolyte<br>imbalance or >2L IV fluids required | Hypotensive shock or physiologic consequences requiring hospitalization |
| Oral discomfort/<br>Dysphagia | Mild discomfort; no difficulty swallowing | Some limits on eating/drinking | Eating/talking very limited; unable to swallow solid foods | Unable to drink fluids; requires IV fluids |

IV=intravenous.

| NEUROLOGICAL | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Neuro-Cerebellar | Slight incoordination dysdiadochokinesis | Intention tremor, dysmetria, slurred speech; nystagmus | Locomotor ataxia | Incapacitated |
| Psychiatric | Mild anxiety or depression | Moderate anxiety or depression;<br>therapy required; change in<br>normal routine | Severe mood changes requiring therapy; or suicidal ideation; or aggressive ideation | Acute psychosis requiring hospitalization; or suicidal gesture/attempt or hallucinations |
| Muscle strength | Subjective weakness; no objective symptoms/signs | Mild objective signs/symptoms; no decrease in function | Objective weakness; function limited | Paralysis |
| Paresthesia (burning, tingling, etc.) | Mild discomfort; no treatment required | Moderate discomfort; non-narcotic analgesia required | Severe discomfort; or narcotic analgesia required with symptomatic improvement | Incapacitating; or not responsive to narcotic analgesia |
| Neurosensory | Mild impairment in sensation (decreased sensation, e.g., vibratory, pinprick, hot/cold in great toes) in focal area or symmetrical distribution; or change in taste, smell, vision, and/or hearing | Moderate impairment (moderately decreased sensation, e.g., vibratory, pinprick, hot/cold to ankles) and/or joint position or mild impairment that is not symmetrical | Severe impairment (decreased or loss of sensation to knees or wrists) or loss of sensation of at least moderate degree in multiple different body areas (i.e., upper and lower extremities) | Sensory loss involves limbs and trunk; paralysis; or seizures |

| MUSCULOSKELETAL | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Arthralgia<br>(joint pain) | Mild pain not interfering with function | Moderate pain, analgesics and/or pain interfering with function but not with ADL | Severe paid; pain and/or analgesics interfering with ADL | Disabling pain |
| Arthritis | Mild pain with inflammation, erythema or joint swelling, but not interfering with function | Moderate pain with inflammation, erythema or joint swelling; interfering with function but not with ADL | Severe pain with inflammation,<br>erythema or joint swelling, and<br>interfering with ADL | Permanent and/or disabling joint destruction |
| Myalgia | Myalgia with no limitation of activity | Muscle tenderness (at other than injection site) or with moderate impairment of activity | Severe muscle tenderness with marked impairment of activity | Frank myonecrosis |

212390

ADL=activities of daily living.

| SKIN | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Mucocutaneous | Erythema; pruritus | Diffuse, maculo papular rash, dry desquamation | Vesiculation or moist desquamation or ulceration | Exfoliative dermatitis, mucous membrane involvement or erythema, multiforme or suspected Stevens-Johnson or necrosis requiring surgery |
| Induration | <15 mm | 15 to 30 mm | >30 mm | N/A |
| Erythema | <15 mm | 15 to 30 mm | >30 mm | N/A |
| Edema | <15 mm | 15 to 30 mm | >30 mm | N/A |
| Rash at injection site | <15 mm | 15 to 30 mm | >30 mm | N/A |
| Pruritus | Slight itching at injection site | Moderate itching at injection extremity | Itching over entire body | N/A |

N/A=not applicable.

| SYSTEMIC | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Allergic reaction | Pruritus without rash | Localized urticarial | Generalized urticarial; angioedema | Anaphylaxis |
| Headache | Mild, no treatment required | Transient, moderate; treatment required | Severe; responds to initial narcotic therapy | Intractable; requires repeated narcotic therapy |
| Fever: oral | 37.7 to 38.5°C or 100.0 to 101.5°F | 38.6 to 39.5°C or 101.6 to 102.9°F | 39.6 to 40.5°C or 103 to 105°F | >40°C or >105°F |
| Fatigue | Normal activity reduced <48 hours | Normal activity decreased 25 to 50%; >48 hours | Normal activity decreased >50%; cannot work | Unable to care for self |

212390

## 10.14. Appendix 14: Abbreviations and Trademarks

| ABSSSI | acute bacterial skin and skin structure infection |
|----------|----------------------------------------------------------|
| AE | adverse event |
| CCI | |
| ALT | alanine aminotransferase |
| AUC12h | area under the drug concentration-time curve over 12 |
| | hours |
| AUC24h | area under the drug concentration-time curve over 24 |
| | hours |
| BID | twice daily |
| CDC | Centers for Disease Control and Prevention |
| CE | Clinically Evaluable |
| CFU | colony-forming units |
| CI | confidence interval |
| CONSORT | Consolidated Standards of Reporting Trials |
| COVID-19 | coronavirus disease |
| CRF | case report form |
| CV | cardiovascular |
| CYP3A4 | cytochrome P450 enzyme 3A4 |
| DMID | Division of Microbiology and Infectious Diseases |
| EAGLE | Efficacy of Antibacterial Gepotidacin Evaluated |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| EMA | European Medicines Agency |
| ESBL | extended-spectrum β-lactamase |
| F | Fahrenheit |
| fAUC/MIC | ratio of the area under the free-drug concentration-time |
| | curve to minimum inhibitory concentration over 24 hours |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| GSK | GlaxoSmithKline |
| HPF | high-power field |
| HRT | hormonal replacement therapy |
| IA | interim analysis |
| IB | investigator's brochure |
| ICE | intercurrent event |
| ICF | informed consent form |
| ICH | International Council on Harmonisation |
| IDMC | Independent Data Monitoring Committee |
| IEC | independent ethics committee |
| IRB | institutional review board |
| IRT | interactive response technology |
| ITT | Intent-to-Treat |
| IV | intravenous |
| kg | kilogram |

| m | meter |
|-----------|------------------------------------------------------------|
| MDR | multidrug-resistant |
| ME | Microbiologically Evaluable |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | milligram |
| MIC | minimum inhibitory concentration |
| micro-ITT | Microbiological Intent-to-Treat |
| min | minute |
| mL | milliliter |
| mm | millimeter |
| msec | millisecond |
| NTF | nitrofurantoin |
| NTF-NS | not susceptible to NTF |
| NTF-S | susceptible to NTF |
| PD | pharmacodynamic |
| PK | pharmacokinetic |
| QTc | corrected QT interval |
| QTcB | QT interval corrected for heart rate according to Bazett's |
| QTCD | formula |
| QTcF | QT interval corrected for heart rate according to |
| QTCI | Fridericia's formula |
| RAP | reporting and analysis plan |
| SAE | serious adverse event |
| SDAC | Statistical Data Analysis Center |
| SoA | Schedule of Activities |
| SRM | Study Reference Manual |
| SRT | Safety Review Team |
| ST | sequence type |
| TdP | torsades de pointes |
| TOC | Test-of-Cure |
| TMP-SXT | trimethoprim-sulfamethoxazole |
| μg | microgram |
| ULN | upper limit of normal |
| UTI | urinary tract infection |
| WHO | World Health Organization |
| WOCBP | woman of childbearing potential |
| T. | "olimi of childocaring potential |

#### **Trademark Information**

| Trademarks of the GlaxoSmithKline group of companies |
|------------------------------------------------------|
| None |

| Trademarks not owned by the GlaxoSmithKline group of companies |
|----------------------------------------------------------------|
| FIRST RESPONSE |
| MedDRA |

### 10.15. Appendix 15: Protocol Amendment History

The Protocol Amendment Summary of Changes Table for the current amendment (i.e., Protocol Amendment 3) is located directly before the Table of Contents.

212390

#### Amendment 2 14-APR-2021

This global amendment was considered to be substantial.

Overall Rationale for the Amendment:

| indicated study operational allowances with regard to COVID-19; |
|---|
| incorporated past administrative letters to the sites; clarified estimand text; provided |
| minor statistical clarifications to the analysis populations, response and outcomes tables, |
| and accounted for supplementary analysis, which will be detailed in the RAP; increased |
| the planned total enrollment population; clarified On-therapy Visit electrocardiograms |
| will be collected in the first approximately 1200 participants; incorporated updates per |
| the most recent IB version 07; and globally replaced "intervention" with "treatment." The |
| amendment also includes additional minor administrative and wording edits. |

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| Synopsis 3 Objectives and Estimands/Endpoints Table 1 Estimand for the Secondary Endpoints 9.4.1 General Considerations 9.4.2 Efficacy Analysis | Separated estimand text from the endpoint text, revised the estimand language to include the 5 components per recent ICH guidelines on estimands, added estimand descriptions for the secondary endpoints | To provide expanded details on the primary and secondary estimands |
| Synopsis 3 Objectives and Estimands/Endpoints | For the secondary (updated only in the Synopsis) and exploratory objectives, an additional objective and endpoint were added to each section to examine the clinical response in female participants with acute cystitis with qualifying bacterial uropathogens(s) at Baseline that all are susceptible to nitrofurantoin | Consistency with the primary objective population |

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| Synopsis 9.2.1 Justification of Sample Size | Increased the total enrollment sample size to up to 2500 participants | To reflect the expected number of participants for full enrollment to support the required number of evaluable participants for the primary analysis |
| 1.2 Schema | Revised On-therapy Visit to state Days 2 to 4 | Protocol consistency |
| 2.3.1 Risk<br>Assessment<br>5.2 Exclusion Criteria<br>#5 | Added acute porphyria as an example of a risk for the nitrofurantoin comparator and excluded the medical condition for participant enrollment | Incorporation of the letter to sites dated 17-DEC-2019 |
| Section 2.3.1 Risk<br>Assessment | Removed exclusion for strong P-glycoprotein inhibitors | Consistency with the most current Version 07 of the investigator's |
| 5.2 Exclusion Criteria<br>#21 | | brochure |
| 6.5.2 Prohibited Medications and Nondrug Therapies | | |
| Section 10.9<br>Appendix 9 | | |
| 5.2 Exclusion Criteria<br>#10 | Expanded text to include, "or preclude complete resolution of acute cystitis symptoms" | Clarification purposes |
| 6.5 Concomitant<br>Therapy | Clarified that any antibiotic use within 6 months of the Baseline Visit should be recorded | To support the study analysis |
| 6.5.1 Permitted<br>Medications and<br>Nondrug Therapies | Clarified that low-dose acetylsalicylic acid is permitted as a concomitant medication if taken | To support study conduct and enrollment for a medication used in a manner that should not have |
| 6.5.2 Prohibited Medications and Nondrug Therapies | to prevent cardiovascular disease events | an impact on the efficacy evaluations |
| Section 10.9<br>Appendix 9 | | |

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| 6.5.2 Prohibited Medications and Nondrug Therapies | Added strong CYP3A4 inducers to the prohibited medications | Alignment with preliminary results from a recently completed Phase I study |
| Section 10.9<br>Appendix 9 | | |
| Schedule of Activities | Clarified that the physical examination at the Test-of-Cure | Incorporation of Protocol Administration Letter 2 |
| 8.2.1 Physical Examinations | Visit may be symptom directed and was only required if indicated for a specific participant | Administration Letter 2 |
| Schedule of Activities 8.2.3 Electrocardiograms | Clarified the collection of electrocardiograms at the On-therapy Visit would be collected for the first approximately 1200 participants enrolled | Consistency with the maximum planned sample size in protocol amendment 1 |
| 8.2.3<br>Electrocardiograms | Clarified text for the collection of electrocardiograms, including the order of collection, repeated electrocardiograms, and the window for collection during the On-therapy Visit | To support study conduct |
| 8.1.2.1<br>Microbiological<br>Outcome and<br>Response | Minor text clarifications were added to the outcome and response tables, and a new table (Table 5) was added to define participant-level microbiological outcomes and responses | To provide clarification to support the planned statistical analyses and programming details |
| 8.1.3 Clinical<br>Evaluation | Subsections were added for the different clinical evaluations planned for primary and exploratory objectives, minor text clarifications were added to the outcome and response tables | To provide clarification to support the planned statistical analyses and programming details |

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| Synopsis Schedule of Activities 8.1.3.3 Urinary Tract Infection Activity Impairment Assessment | Indicated this assessment should<br>be performed at the end of the<br>study visits and by a different<br>study staff member than the<br>person conducting the clinical<br>symptoms assessment and<br>scoring | To prioritize collection of the primary efficacy clinical measurements with separation from the exploratory clinical measurements |
| Schedule of Activities 8.1.3.1 Clinical Signs and Symptoms Scores, Clinical Outcomes, and Clinical Response Throughout Appendix 6 Clinical Signs and Symptoms Score for Acute Cystitis | Clarified that the clinical signs and symptoms scores should be performed by a physician or otherwise appropriately medically trained staff, and that the same scorer should perform the assessment at all time points whenever possible, and clarified additional instructions for the collection of data verbally to support the assessment | Incorporation of Protocol<br>Administrative Letter 2, which will<br>support consistent data collection |
| CCI | | |
| Schedule of Activities Throughout Appendix 5 | Added text to allow for eConsent, telemedicine study-related data collection, collection of visit data as a combination of telemedicine and on-site visits, remote source data verification, and eCRF signoff flexibility for investigators | To support ongoing study conduct from safety and operational perspectives during the COVID-19 pandemic |
| 9.3 Populations for<br>Analyses | Minor clarifications to the description of populations, including updates to analyze per randomized study treatment, where applicable | Consistency with the planned statistical analysis and required outputs |

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| 9.4.1 General<br>Considerations | Added text regarding supplemental analysis and additional analysis that may be needed per COVID-19 impact on the study | Consistency with the planned statistical analysis and required outputs |
| 9.4.2 Efficacy<br>Analyses<br>9.4.3 Safety Analyses | Minor clarifications to the plans for analysis | Consistency with the planned statistical analysis and required outputs |
| 2.3.1 Risk<br>Assessment<br>Throughout | Updates to protocol text, including risk/benefit and dose justification rationale text (i.e., added topline PK and safety results from a study in healthy adult and adolescent participants) per the most current investigator's brochure; no new safety signals were identified or added | Consistency with the most current Version 07 of the investigator's brochure |
| Appendix 4 Algorithm for Determining Qualifying Uropathogens | Minor clarifications per the current plans for analysis | Consistency with regulatory authority feedback and statistical analysis plans |
| Throughout | Where applicable, globally replaced "intervention" with "treatment" | Consistency with the planned statistical analysis and required outputs |
| Throughout | Revised the in-text definitions of microbiological and clinical success to remove "specific to the disease under study" regarding the use of other systemic antimicrobials | Corrected text to align with the original definitions of success in the endpoint definition tables |
| Throughout | Updated text to state <i>Clostridium</i> difficile and acetylcholinesterase inhibition events are considered adverse events of special interest | To support the planned safety analysis |
| Throughout | Minor editorial and document formatting revisions | Minor, therefore, have not been summarized |

#### Amendment 1 14-NOV-2019

Overall Rationale for the Amendment: This global amendment provided clarification on Inclusion Criteria 3 and 4, including no requirement for contraception use or abstinence within 14 days of study entry in women of childbearing potential (WOCBP) with a negative high sensitivity urine pregnancy test result at Baseline (Day 1), expanded the On-therapy Visit window, allowed flexible options for pregnancy testing and dose administration for the On-therapy Visit, and further defined the optimum window for pregnancy testing while participants were receiving study treatment. The amendment also included additional minor administrative edits.

212390

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| 5.1 Inclusion Criteria Schedule of Activities | Criterion 3, edited terminology to<br>"large" for the presence of<br>3+ leukocyte esterase | To correct terminology for laboratory results |
| 5.1 Inclusion Criteria Schedule of Activities Appendix 6 | Criterion 4, edited female entry criterion for clarity, including that no current or prior contraception use or abstinence is needed in WOCBP with a negative high sensitivity urine pregnancy test result at Baseline (Day 1) | To provide clarification on female participant requirements at study entry |
| Synopsis Schedule of Activities 4.1 Overall Design 8 Study Assessments and Procedures | Revised the study day range for<br>the On-therapy Visit from "Day 2<br>to 3" to "Day 2 to 4" and noted that<br>each treatment day will be<br>assessed over 24 hours based on<br>the time of the first dose of study<br>treatment | To support study conduct |
| Schedule of Activities<br>8 Study Assessments<br>and Procedures | Updated the definition of the On-therapy Visit to be "1 to 3 days" postrandomization | Protocol consistency |
| Schedule of Activities 6.1 Study Treatments Administered 8 Study Assessments and Procedures | Indicated that, based on the opinion of the investigator, flexible options are allowed for pregnancy testing and dose administration for the On-therapy Visit | To support study conduct |
| Schedule of Activities<br>8 Study Assessments<br>and Procedures | Revised the pregnancy test for WOCBP during study treatment to be performed "after Dose 4 and before Dose 8" | To ensure the pregnancy test is performed within an optimum safety window and to support |

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| Appendix 6 | | testing to preferably occur at the study site |
| 9.4.2 Efficacy<br>Analyses | Moved the microbiological outcome for new qualifying uropathogens from secondary to exploratory | Correction to the planned data analyses |
| Throughout | Expanded the definitions of microbiological and clinical success to include "specific to the disease under study" regarding the use of other systemic antimicrobials | To further clarify which antimicrobials will affect success or failure in the analysis |
| Throughout | Minor editorial and document formatting revisions | Minor, therefore, have not been summarized |

#### 11. REFERENCES

Abreu AG, Marques SG, Monteiro-Neto V, Gonçalves AG. Extended-spectrum β-lactamase-producing enterobacteriaceae in community-acquired urinary tract infections in Sãn Luís, Brazil. Braz J Microbiol. 2013;44(2):469-71.

Centers for Disease Control and Prevention (CDC). Antibiotic resistance threats in the United States, 2019. https://www.cdc.gov/drugresistance/pdf/threats-report/2019-arthreats-report-508.pdf. Accessed 20-Mar-2021.

European Association of Urology (EAU). EAU guidelines. Edn. presented at the EAU Annual Congress Barcelona 2019. ISBN 978-94-92671-04-2. https://uroweb.org/guideline/urological-infections/. Accessed 26-Jul-2019.

European Medicines Agency (EMA). Addendum to the guideline on the evaluation of medicinal products indicated for treatment of bacterial infections. CPMP/EWP/558/95 rev 2. 24-Oct-2013.

Fihn SD. Clinical practice. Acute uncomplicated urinary tract infection in women. N Engl J Med. 2003;349(3):259-66.

Flamm RK, Sader HS, Farell DJ, Jones RN. Ceftazidime-avibactam and comparator agents tested against urinary tract isolates from a global surveillance program (2011). Diagn Microbiol Infect Dis. 2014;80(3):233-8.

Foxman B, Barlow R, D'Arcy H, Gillespie B, Sobel JD. Urinary tract infection: self-reported incidence and associated costs. Ann Epidemiol. 2000;10(8):509-15.

Foxman B. Epidemiology of urinary tract infections: incidence, morbidity, and economic costs. Am J Med. 2002;113(Suppl 1A):5S-13S.

Foxman B. The epidemiology of urinary tract infection. Nat Rev Urol. 2010;7(12):653-60.

Gupta K, Hooton TM, Miller L; Uncomplicated UTI IDSA Guideline Committee. Managing uncomplicated urinary tract infection—making sense out of resistance data. Clin Infect Dis. 2011a;53(10):1041-2.

Gupta K, Hooton TM, Naber KG, Wullt B, Colgan R, Miller LG, et al. International clinical practice guidelines for the treatment of acute uncomplicated cystitis and pyelonephritis in women: a 2010 update by the Infectious Diseases Society of America and the European Society for Microbiology and Infectious Diseases. Clin Infect Dis. 2011b;52(5):e103-20.

Gupta K, Hooton TM, Roberts PL, Stamm WE. Short-course nitrofurantoin for the treatment of acute uncomplicated cystitis in women. Arch Intern Med. 2007;167(20):2207-12.

Ho PL, Poon WW, Loke SL, Leung MS, Chow KH, Wong RC, et al; COMBAT study group. Community emergence of CTX-M type extended-spectrum β-lactamases among urinary *Escherichia coli* from women. J Antimicrob Chemother. 2007;60(1):140-4.

Hooton TM. Clinical practice. Uncomplicated urinary tract infection. N Engl J Med. 2012;366(11):1028-37.

Johnson JR, Nicolas-Chanoine MH, DebRoy C, Castanheira M, Robicsek A, Hansen G, et al. Comparison of *Escherichia coli* ST131 pulsotypes, by epidemiologic traits, 1967-2009. Emerg Infect Dis. 2012;18(4):598-607.

Lan KK, DeMets D. Discrete sequential boundaries for clinical trials. Biometrika. 1983; 70:659-63.

Lob SH, Nicolle LE. Hoban DJ, Kazmierczak KM, Badal RE, Sahm DF. Susceptibility patterns and ESBL rates of *Escherichia coli* from urinary tract infections in Canada and the United States, SMART 2010-2014. Diagn Microbiol Infect Dis. 2016;85(4):459-65.

Miettinen O, Nurminen M. Comparative analysis of two rates. Stat Med. 1985;4(2):213-26.

National Institute for Health Care Excellence (NICE). Public Health England. Summary of antimicrobial prescribing guidance – managing common infections. Feb 2019. https://www.nice.org.uk/Media/Default/About/what-we-do/NICE-guidance/antimicrobial%20guidance/summary-antimicrobial-prescribing-guidance.pdf?UNLID=3157626232019111861. Accessed 19-Jun-2019.

Nicolas-Chanoine MH, Bertrand X, Madec JY. *Escherichia coli* ST131, an intriguing clonal group. Clin Microbiol Rev. 2014;27(3):543-74.

Oteo J, Bautista V, Lara N, Cuevas O, Arroyo M, Fernández S, et al; Spanish ESBL-EARS-Net Study Group. Parallel increase in community use of fosfomycin and resistance to fosfomycin in extended-spectrum beta-lactamase (ESBL)-producing *Escherichia coli*. J Antimicrob Chemother. 2010;65(11):2459-63.

Peirano G, Richardson D, Nigrin J, McGreer A, Loo V, Toye B, et al. High prevalence of ST131 isolates producing CTX-M-15 and CTX-M-14 among extended-spectrum-beta-lactamase-producing *Escherichia coli* isolates from Canada. Antimicrob Agents Chemother. 2010;54(3):1327-30.

Sanchez GV, Babiker A, Master RN, Luu T, Mathur A, Bordon J. Antibiotic resistance among urinary isolates from female outpatients in the United States in 2003 and 2012. Antimicrob Agents Chemother. 2016;60(5):2680-3.

Sanchez GV, Master RN, Karlowsky JA, Bordon JM. In vitro antimicrobial resistance of urinary *Escherichia coli* isolates among US outpatients from 2000 to 2010. Antimicrob Agents Chemother. 2012;56(4):2181-3.

Schito GC, Naber KG, Botto H, Palou J, Mazzei T, Gualco L, et al. The ARESC study: an international survey on the antimicrobial resistance of pathogens involved in uncomplicated urinary tract infections. Int J Antimicrob Agents. 2009;34(5):407-13.

212390

Stamm WE, Hooton TM. Management of urinary tract infections in adults. N Engl J Med. 1993;329(18):1328-34.

Talan DA, Stamm WE, Hooton TM, Moran GJ, Burke T, Iravani A, et al. Comparison of ciprofloxacin (7 days) and trimethoprim-sulfamethoxazole (14 days) for acute uncomplicated pyelonephritis in women: a randomized trial. JAMA. 2000;283(12):1583-90.

US Department of Health and Human Services, DHHS, Food and Drug Administration, Center for Drug Evaluation and Research, Clinical/Antimicrobial. Draft guidance for industry. Uncomplicated urinary tract infections: developing drugs for treatment. https://www.fda.gov/media/129531/download. Last updated August 2019. Accessed 29-Jul-2021.

US Department of Health and Human Services, DHHS, Food and Drug Administration, Center for Drug Evaluation and Research, Clinical/Antimicrobial. Guidance for industry. Complicated urinary tract infections: developing drugs for treatment. https://www.fda.gov/media/71313/download. Last updated June 2018. Accessed 29-Jul-2021.

US National Institute for Allergy and Infectious Disease Division of Microbiology and Infectious Diseases. Division of Microbiology and Infectious Diseases (DMID) Pediatric Toxicity Table. Draft. https://www.niaid.nih.gov/sites/default/files/dmidpedtox.pdf. Last updated November 2007b. Accessed 29-Jul-2019.

US National Institute for Allergy and Infectious Diseases, Division of Microbiology and Infectious Diseases. Division of Microbiology and Infectious Diseases (DMID) Adult Toxicity Table. Draft. https://www.niaid.nih.gov/sites/default/files/dmidadulttox.pdf. Last updated November 2007a. Accessed 29-Jul-2019.



World Health Organization (WHO). Antimicrobial resistance global report on surveillance, 2014.

http://apps.who.int/iris/bitstream/10665/112642/1/9789241564748\_eng.pdf. Accessed 19-Jun-2019.

World Health Organization (WHO). Global priority list of antibiotic-resistant bacteria to guide research, discovery, and development of new antibiotics. 2017. http://www.who.int/medicines/publications/WHO-PPL-Short\_Summary\_25Feb-ET\_NM\_WHO.pdf?ua=1. Accessed 19-Jun-2019.